

#### **PROTOCOL TITLE:**

POW-R Health: Power to Redefine your Health (Internal Title: A Pragmatic Dietary Intervention to Improve Bladder Cancer Survivorship)

#### **PROTOCOL NUMBER:**

I 661820

#### PRINCIPAL INVESTIGATOR:

Karen Yeary, PhD Roswell Park Comprehensive Cancer Center Elm and Carlton Street Buffalo, New York 14263 716-845-6231 karen.yeary@roswellpark.org@roswellpark.org

## **VERSION NUMBER:**

17

**DATE:** 

10/31/2022

SPONSOR: Roswell Park Comprehensive Cancer Center

**FUNDING: NIH & NCI** 

#### **Confidentiality Statement**

Any and all information presented in this document shall be treated as confidential and shall remain the exclusive property of the party (ies) mentioned above (Roswell Park Cancer Institute Corporation d/b/a Roswell Park Comprehensive Cancer Center). The use of such confidential information must be restricted to the recipient for the agreed purpose and must not be disclosed, published, or otherwise communicated to any unauthorized persons, for any reason, in any form whatsoever without the prior written consent of the party(ies) above.

10/31/2022 

## **Table of Contents**

| 1. | Objectives | 3 |
|-----|-----------------------------------------------------------------|----|
| 2. | Background | 4 |
| 3. | Inclusion and Exclusion Criteria | 6 |
| 4. | Local and Study-Wide Number of Subjects | 7 |
| 5. | Local and Study-Wide Recruitment Methods | 8 |
| 6. | Multi-Site Research | 9 |
| 7. | Study Timelines | 10 |
| 8. | Study Endpoints | 10 |
| 9. | Design | 11 |
| 10. | Treatment | 12 |
| 11. | Procedures Involved | 12 |
| 12. | Withdrawal of Subjects | 16 |
| 13. | Risks to Subjects | 16 |
| 14. | Potential Benefits to Subjects | 16 |
| 15. | Data and Specimen Banking | |
| 16. | Measurement of Effect | 17 |
| 17. | Safety Evaluation | |
| 18. | Data Management and Confidentiality | 18 |
| 19. | Statistical Plan | 19 |
| 20. | Provisions to Monitor the Data to Ensure the Safety of Subjects | 21 |
| 21. | Vulnerable Populations | 21 |
| 22. | Community-Based Participatory Research | |
| 23. | Sharing of Results with Subjects | 21 |
| 24. | Setting | |
| 25. | Provisions to Protect the Privacy Interests of Subjects | 23 |
| 26. | Resources Available | |
| 27. | Prior Approvals | |
| 28. | Compensation for Research-Related Injury | 24 |
| 29. | Economic Burden to Subjects | 24 |
| 30. | Consent Process | 25 |
| 31. | Process to Document Consent in Writing | 26 |
| 32. | Drugs or Devices | 26 |
| 33. | References | 27 |
| 34. | Appendices/ Supplements | 31 |

#### 1. OBJECTIVES

We hypothesize that a behavioral dietary intervention designed to modestly increase cruciferous vegetable intake in patients with Non-Muscle Invasive Bladder Cancer (NMIBC) will significantly reduce recurrence and progression. Findings from our *in vitro*, *in vivo*, and epidemiologic studies <sup>1-10</sup> have shown that dietary isothiocyanates (ITCs) exert potent anti-cancer activities against bladder cancer. ITCs are a group of phytochemicals primarily derived from cruciferous vegetables and oral consumption of dietary ITCs can be rapidly metabolized, delivered to the bladder, and concentrated in the urine—rendering the abnormal bladder epithelium the best target. In our retrospective study<sup>1</sup>, higher consumption of raw cruciferous vegetables was associated with reduced bladder cancer-specific and overall mortality.

We will use the ORBIT Model<sup>11</sup> to translate our strong preclinical findings into a novel, dietary behavioral intervention to reduce bladder cancer recurrence and progression in diverse patients with NMIBC. We will partner with the New York State Cancer Registry (NYSCR) to recruit and enroll eligible patients and their clinical care providers in our catchment area, which is characterized by a disproportionally high risk of and mortality rate for bladder cancer. The dietary intervention will be based on Social Cognitive Theory<sup>12</sup> and developed in collaboration with our Community Advisory Board consisting of bladder cancer care providers and patients to ensure optimal uptake by survivors. To facilitate the rapid translation of research into evidence-based practice, implementation support strategies will be identified at the clinic level as an incremental step towards integrating the dietary behavioral intervention into current healthcare systems serving patients with bladder cancer. The study's specific aims are:

**Specific Aim 1:** Develop an evidence-based behavioral intervention to increase cruciferous vegetable intake, with the goal of attaining desirable urinary ITC levels effective for anti-cancer activities. We will work with our Community Advisory Board to adapt materials and methods from current evidence-based fruit and vegetable interventions and leverage our findings on ITC yield from cruciferous vegetables to develop our dietary intervention, using a systematic process consisting of information gathering, discussion groups, and mock intervention delivery.

**Specific Aim 2:** Conduct a feasibility pilot of our dietary behavioral intervention through a hybrid I implementation randomized controlled design in 80 NMIBC survivors, where the treatment group (n=40) will receive an evidence-based telephone intervention to increase cruciferous vegetable intake and the control group (n=40) will receive a general fruit and vegetable intake intervention based on NCI guidelines. The primary outcomes will be cruciferous vegetable intake and urinary ITC levels, and the secondary outcome will be gene expression changes in urinary exfoliated epithelial cells as a surrogate for intermediate efficacy.

**Exploratory Aim:** Engage the clinical care providers of patients enrolled in our intervention to ascertain the barriers and facilitators of intervention implementation within clinical practice through conducting 20 semi-structured interviews. The goal is to gain feedback and refine the intervention for "real-world' implementation.

#### **Primary Objective(s)**

 Develop an evidence-based behavioral intervention to increase cruciferous vegetable intake, with the goal of attaining desirable urinary ITC levels effective for anti-cancer activities. We will work with our Community Advisory Board to adapt materials and methods from current evidence-based fruit and vegetable interventions and leverage

10/31/2022 

- our findings on ITC yield from cruciferous vegetables to develop our dietary intervention, using a systematic process consisting of information gathering, discussion groups, and mock intervention delivery.
- Conduct a feasibility pilot of our dietary behavioral intervention through a hybrid I implementation randomized controlled design in 80 NMIBC survivors, where the treatment group (n=40) will receive an evidence-based telephone intervention to increase cruciferous vegetable intake and the control group (n=40) will receive a general fruit and vegetable intake intervention based on NCI guidelines. The primary outcomes will be cruciferous vegetable intake and urinary ITC levels.

## **Secondary Objective(s)**

• The secondary outcome will be to ascertain the level of gene expression changes in urinary exfoliated epithelial cells (due to the intervention) as a surrogate for intermediate efficacy.

### **Exploratory Objective(s)**

• Engage the clinical care providers of patients enrolled in our intervention to ascertain the barriers and facilitators of intervention implementation within clinical practice through conducting 20 semi-structured interviews. The goal is to gain feedback and refine the intervention for "real-world' implementation.

#### 2. BACKGROUND

The problem of bladder cancer. Bladder cancer is the sixth most common cancer in the US, contributing to over 80,000 new cases and 17,000 deaths annually<sup>2</sup>. The majority of bladder cancer (70-80%) is diagnosed at an early stage with cancer confined to the epithelial and lamina propria layer of the bladder—also known as non-muscle invasive bladder cancer (NMIBC)<sup>4</sup>. The standard treatment for NMIBC is transurethral resection of bladder tumor, which is a routine clinic procedure without hospitalization. However, NMIBC typically recurs (50-80%) with some patients experiencing multiple recurrences at similar stages and others (20-30%) progressing to muscle-invasive disease, which is associated with cystectomy and poor survival<sup>3-5</sup>. Depending on pathological characteristics, approximately 15% of tumors are defined as high-risk and receive one or more doses of intravesical therapeutic agents<sup>6</sup>, of which Bacillus Calmette-Guerin (BCG) has been the gold standard for four decades<sup>7</sup>. Yet approximately 30% of these patients will be nonresponders to BCG, and high incidence of local side effects are concerns<sup>7</sup>. For the majority of NMIBC patients, no other treatment is available, although they are still at risk of recurrence and progression. Current clinical management requires life-long surveillance by cystoscopy for NMIBC patients, amounting to bladder cancer being the most expensive cancer to treat per patient<sup>8-10</sup>. An estimated 696,440 people are living with bladder cancer in the US<sup>23</sup>, the majority of which are off treatment and under surveillance. Novel, non-invasive, cost-effective strategies to control NMIBC recurrence and progression are urgently needed.

**Dietary isothiocyanates (ITCs) in bladder cancer chemoprevention.** Dietary ITCs are a group of phytochemicals primarily derived from cruciferous vegetables (cruciferae) with multi-faceted anti-cancer mechanisms. Our group has published 10 peer-reviewed papers<sup>11-20</sup> involving *in vitro*, *in vivo*, and epidemiologic studies demonstrating the important role of dietary ITCs and ITC-rich cruciferae in preventing bladder cancer recurrence and progression. The four most common dietary ITCs and their primary urinary metabolites potently inhibited the growth of a panel of human

10/31/2022 

bladder cancer cells including NMIBC cells with  $IC_{50}$  values around  $10\mu M$  averagely<sup>15, 17</sup>, which is realistically achievable in the urine with a single oral dose of ITC at  $10 \mu mol/kg$  weight in rats<sup>24</sup>. ITC at  $10 \mu mol/kg$  (approximately 1 mg/kg) is also readily achievable in humans, with some cruciferae yielding as much as 3.4 mg ITC per gram<sup>25</sup>. Daily oral administration of ITC at the same dose level for three weeks significantly inhibits orthotopic bladder cancer growth<sup>20</sup>. Importantly, we demonstrated that dietary ITCs not only inhibit bladder cancer development, but also prevent tumor progression into muscle-invasive disease<sup>18, 20</sup>. Our group also discovered that orally ingested ITCs are rapidly and almost exclusively delivered to the bladder and concentrated in urine, showing 2-3 orders of magnitude higher concentration of ITCs and metabolites in the urine than in the plasma within 3 hours of dosing<sup>18,20</sup>. Storage of the urine in the bladder further enhances exposure of malignant cells to ITCs. Therefore, this unique metabolism and disposition pathway makes the bladder the best target for ITCs or ITC-rich cruciferae. In our retrospective study of 239 bladder cancer patients<sup>11, 12</sup>, raw cruciferae intake was inversely associated with bladder cancer risk, and importantly, associated with a significantly improved disease-specific survival (hazard ratio = 0.43, 95% confidence interval = 0.25-0.74).

**Low cruciferae intake in bladder cancer survivors (BCS).** Although the potential beneficial effect of dietary ITCs in bladder cancer is compelling, the consumption of the primary dietary resource of ITCs—cruciferae—is generally low among BCS. An average of 0.45 serving per day was observed in our retrospective study<sup>12</sup>, similar to the report of the daily consumption of 0.44 servings in a pilot study of 48 BCS<sup>26</sup>. Preliminary analysis of food frequency questionnaire (FFQ) data from over 1,400 newly diagnosed NMIBC patients from our Be-Well study (R01CA172855)<sup>27</sup> reported that daily intake of cruciferae was about 52.7 gram, or approximately 0.7 servings; while urinary ITC level was around 4.4 μM, which is below the averagely 10 μM of ITCs observed to stop or kill at least 50% of bladder cancer cells in *in vitro* models<sup>15, 17</sup>. Based on our recent findings on the diverse range of ITC yield from cruciferae and the various impact of cooking methods on the ITC yield<sup>28, 29</sup>, we believe that *at least one serving* (~1 cup raw or ½ cup cooked) of cruciferae per day, with guidance on the choice of vegetables and cooking conditions, will increase urinary ITC levels to the desirable doses needed to exert anti-cancer activities in the bladder.

Lack of interventions to increase cruciferae intake. Systematic reviews<sup>30-34</sup> and metaanalyses<sup>35</sup> have documented the effectiveness of behavioral dietary interventions to increase vegetable intake in adults, including older and male participants, who comprise the majority of BCS<sup>4</sup>. Only one study tested an intervention designed to increase vegetable intake in BCS<sup>26</sup>. Compared to control participants, intervention participants significantly increased their daily vegetable intake (2.4 to 3.9 servings) from baseline to 6-months, but not cruciferae intake. The intervention also failed to deliver the corresponding increase in urinary ITC concentrations, showing comparable ITC levels between intervention and control groups at 6-month follow-up. We will use our prior work to maximize ITC exposure in the following ways: 1) ITC yield varies as much as 300-fold from raw cruciferae<sup>28</sup>, thus we will recommend proper vegetables (e.g. arugula, cabbage) in our intervention; 2) heavily cooking largely reduces ITC yield, while lightly cooking substantially increases ITC yield from cruciferae<sup>28</sup>. Thus, we will recommend proper cooking conditions (e.g. stir-frying, microwaving) in our intervention; 3) peak urinary concentration is achieved within 3 hours of dosing and more than 50% of the dose is excreted and accumulated in urine within 8 hours of dosing<sup>20, 36</sup>. Thus, we will recommend consumption at dinner time to avoid ITCs being quickly excreted out of body from frequent urination during the day.

10/31/2022 

Scientific premise. Bladder cancer will recur in the majority (50-80%) of NMIBC patients, yet current management is close monitoring with additions of intravesical therapies for a small portion of patients (15%) only<sup>4, 6</sup>. Effective interventions are needed to prevent disease recurrence and progression and improve cancer-specific survival for NMIBC survivors with minimum side effects, participant/provider burden, and cost. Robust preclinical and epidemiological data document the promising anti-cancer effects of cruciferae as a source of ITCs against bladder cancer. Numerous dietary interventions have effectively increased vegetable intake in diverse adults. Yet an effective intervention designed to improve bladder cancer prognosis through increasing cruciferae intake has not been developed. We propose to translate our basic science research findings in dietary ITCs and bladder cancer into an evidence-based behavioral intervention for NMIBC patients with potential for population-level impact. The proposed research will accelerate what we currently know into an intervention that could meaningfully impact cancer survivorship in a population at high risk of recurrence and progression that are currently under surveillance.

**Preliminary Studies.** Dr. Tang's work has documented the anti-cancer potential of dietary ITCs and ITC-rich cruciferae against bladder cancer<sup>11-20</sup>. Her recent findings on ITC composition data in food commonly consumed in the Western diet and the effects of cooking methods on ITC yield from cruciferae<sup>28</sup> informed the proposed intervention. Dr. Tang co-led the <u>Be-Well study</u> (R01CA172855), a prospective cohort of NMIBC survivors<sup>27</sup>, which provided data to support the need of a behavioral dietary intervention to increase cruciferae intake to boost urinary ITC levels. Dr. Yeary led <u>The WORD study</u> (2P20MD002329-06), a behavioral weight loss trial of 426 adults that included a dietary component to meet intake goals of at least 5-9 servings of fruits and vegetables a day<sup>38</sup>. The intervention significantly increased vegetable intake by 3.44 (1.51, 5.36) servings from baseline to 6 months. Components of this intervention will be used in our cruciferae intervention for BCS.

#### 3. INCLUSION AND EXCLUSION CRITERIA

#### **Inclusion Criteria**

**Cancer Patient:** 

To be included in this study, participants must meet the following criteria:

- 1. Age 18 years old or older (no upper limit).
- 2. English speaking.
- 3. Diagnosed with stage Tis, Ta, or T1 bladder cancer.
- 4. Resides in the Western New York catchment area.
- 5. Did not receive a partial or radical cystectomy.
- 6. Does not have a prior cancer diagnosis within 12 months of their bladder cancer diagnosis.
- 7. Does not have a subsequent more advanced bladder cancer diagnosis.
- 8. For Roswell Park Cancer Registry only: Bladder cancer diagnosed 2016-2018, 2019-current.
- 9. Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

10/31/2022 

#### Physician:

To be included in this study, physicians must meet the following criteria:

- 1. English speaking.
- 2. Physician in a clinic located in the catchment area.
- 3. Currently treats bladder cancer patients.

Refer to **Appendix A** for the Investigator Study Eligibility Verification Form: Inclusion Criteria.

#### **Exclusion Criteria**

Cancer Patient:

Participants Recruitment will be excluded from this study for the following:

- 1. Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
- 2. Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
- 3. Adults unable to consent.
- 4. Adults unable to complete study measures in English.
- 5. Individuals who are not yet adults (infants, children, teenagers).
- 6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
- 7. Unwilling or unable to follow protocol requirements.

#### Physician:

1. Unable to complete the study measures in English.

Refer to **Appendix B** for the Investigator Study Eligibility Verification Form: Exclusion Criteria.

## **Inclusion of Women and Minorities**

Both men and women and members of all races and ethnic groups are eligible for this study.

#### **Special Populations**

The following special populations ae excluded from this study:

- Cognitively impaired adults/adults with impaired decision-making capacity
- Individuals who are not yet adults (infants, children, teenagers)
- Pregnant women
- Prisoners

#### 4. LOCAL AND STUDY-WIDE NUMBER OF SUBJECTS

We will recruit 80 bladder cancer patients  $\geq$  18 years of age. We will recruit up to 20 physicians in the Western New York area. Recruitment for both patients and physicians will take place over the span of two years (study duration).

10/31/2022 

#### 5. LOCAL AND STUDY-WIDE RECRUITMENT METHODS

Patient Recruitment. Using ICD-O-3 codes provided, Dr. Kuliszewski of the NYSCR will lead her staff to identify qualifying patients from their database based on the study's eligibility requirements. The NYSCR has identified 199 cases that meet the study's eligibility criteria in 2018 and anticipate at least 400 eligible cases in total in 2018 and 2019. A total of 250 eligible patients will be contacted to enable researchers to recruit from a pool of at least 100 patients. In prior studies, 52.4% to 62.5% of patients contacted by the NYSCR agreed to be contacted by researchers for study consent. The NYSCR will send a letter to the physician of record for selected cases notifying that the patient was identified for the study, requesting that the NYSCR be notified if the patient is unable or ineligible to participate in the study, and requesting information about the case's primary care physician if different from the contacted physician. If no contraindication has been received from the physician or if the physician has not responded within 3 weeks, the NYSCR will send an informational packet to the patient. The packet will contain: 1) a letter with study information; 2) a participant information sheet; and 3) a release of information consent form. After two weeks without response, a reminder packet will be sent and followed with up to five phone calls. If the NYSCR can't reach the patient, the patient will be considered a refusal. The NYSCR's materials and procedures will be reviewed by the New York State Department of Health IRB. For patients who agree to be contacted about the study, the NYSCR will securely share the patient's name, contact information, and information about their diagnosis with the Roswell study team through a secure file transfer. We estimate that from the pool of at least 100 patients who consent to be contacted, we will be able to obtain informed consent from at least 80 patients (80%). Research staff will contact patients who have agreed to be contacted by phone, whereby they will provide a general study overview and conduct a screening interview to confirm eligibility. Staff will obtain informed consent to participate in the study by phone; the consent form along with a Participant Welcome Letter (Appendix O) will be mailed to participants for record. To assist with study retention, we will ask participants for contact information to be used in follow-up. Participants will also be given incentives for completing study assessments. The Roswell study team will share information with the NYSCR team on the patients who agree to participate in the study, as well as any information obtained from study participants that does not match the information provided from the NYSCR database (e.g., race, ethnicity).

Roswell Park Cancer Registry. Due to low enrollment from the NYS Cancer Registry, we will also recruit participants from the Roswell Park Cancer Registry that meet the study's eligibility criteria. To avoid overlap with NYS Cancer Registry patients, we will identify potential participants by focusing on patients diagnosed within last five years and exclude patients diagnosed within 2018-2019 (original parameters for the NYS Cancer Registry recruitment list). Study staff will consult with Roswell Park urologist to determine if the patient is unable or ineligible to participate in the study. The patients accessioned from the Roswell Park Cancer Registry will be contacted by letter (See Appendix T) asking them to participate in the study. Study staff will follow-up with potential participants to determine whether they received the letter and if they are interested in participating.

**Physician Recruitment.** We will ask intervention participants to nominate physicians to participate in a short 15-minute semi-structured interview. Research staff will mail an invitation letter to nominated physicians that will include an information sheet (Appendix J), opt-in/opt-card card, and stamped reply envelope. Within 2-weeks, physicians who do not respond will be contacted by phone, fax, or email with no more than 5 attempts. Participating physicians will

10/31/2022 

receive \$100. Physicians who verbally consent to participate will be asked to refer other physicians to the study. Community Advisory Board (CAB) members will also utilize their networks to nominate physicians for staff to contact. We will recruit up to 20 physicians to ensure data saturation<sup>61</sup>. Among clinicians involved in cancer treatment, enrollment rates between 46.3%-92% have been reported<sup>60, 62, 63</sup>, with one study reporting an enrollment rate of 48% among clinicians involved in bladder cancer treatment<sup>62</sup>. Out of the 80 participants enrolled in our intervention, we anticipate 40 to nominate their physicians and we expect to receive referrals for 5 additional physicians from enrolled physicians and 5 physicians nominated by our CAB. Given an anticipated enrollment rate of 48%, we anticipate recruitment of 20 physicians.

#### 6. MULTI-SITE RESEARCH

Since this is NIH funded study, Single IRB will be pursued for the NYS DOH (NYS CR) and Roswell Park will be serving as the IRB of Record.

10/31/2022 

## 7. STUDY TIMELINES

Figure 1

| Study Timeline | ! | | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| zoudy 11111011110 | | | | | | Ye | ar 1 | | | | | | | | | | Y | ear | 2 | | | | | |
| Specific Aim 1: | Dev | elon | an | ovel | dieta | | | vent | ion f | or b | ladd | er c | ance | r sui | rvivo | ors | | | | | | | | |
| Phase 1: | X | <i>3.</i> 0 ( | | | | | | 7.1. | | | | | | | | | | | | | | | | |
| Information | 11 | | | | | | | | | | | | | | | | | | | | | | | |
| gathering | | | | | | | | | | | | | | | | | | | | | | | | |
| Phase 2: | | X | X | | | | | | | | | | | | | | | | | | | | | |
| Review | | 2 % | 2 1 | | | | | | | | | | | | | | | | | | | | | |
| intervention | | | | | | | | | | | | | | | | | | | | | | | | |
| components | | | | | | | | | | | | | | | | | | | | | | | | |
| Phase 3: | | | | X | X | | | | | | | | | | | | | | | | | | | |
| Mock | | | | 2 % | 2 % | | | | | | | | | | | | | | | | | | | |
| intervention | | | | | | | | | | | | | | | | | | | | | | | | |
| delivery to | | | | | | | | | | | | | | | | | | | | | | | | |
| CAB | | | | | | | | | | | | | | | | | | | | | | | | |
| Phase 4: | | | | | | X | X | | | | | | | | | | | | | | | | | |
| Refine | | | | | | 2 % | 2 % | | | | | | | | | | | | | | | | | |
| intervention | | | | | | | | | | | | | | | | | | | | | | | | |
| Train staff to | | | | | | | | X | X | | | | | | | | | | | | | | | |
| deliver the | | | | | | | | 2 <b>L</b> | 2 % | | | | | | | | | | | | | | | |
| intervention | | | | | | | | | | | | | | | | | | | | | | | | |
| Specific Aim 2: | Hv | hrid | Tvr | e I I | leasi | hilit | v Tr | ial | | | | | | | | | | | | | | | | |
| NYSCR and | X | X | | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Roswell Park | 2 % | 2 % | 11 | 2 % | 2 % | 2 % | 21 | 21 | 2 % | 2 % | 2 % | 1 | 1 | 2. | 11 | 21 | 1 | 2 1 | 2 % | 2 % | 2 <b>L</b> | 2 1 | <b>7 L</b> | 2 1 |
| Cancer | | | | | | | | | | | | | | | | | | | | | | | | |
| Registry | | | | | | | | | | | | | | | | | | | | | | | | |
| recruitment | | | | | | | | | | | | | | | | | | | | | | | | |
| (patient agree | | | | | | | | | | | | | | | | | | | | | | | | |
| to contact) | | | | | | | | | | | | | | | | | | | | | | | | |
| Participant | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| recruitment | 2. | 1 | 11 | | 1 2 | 11 | 11 | 1. | 1 2 | - | - | 1. | - | 1. | 1. | - | - | | - | - | - | 1 1 | | _ |
| Participant | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| participation* | | | | | | | | | | | | | | | | | | | | | | | | |
| Data analysis | | | | | | | | | | | | | | | | | | | | | | X | X | X |
| and | | | | | | | | | | | | | | | | | | | | | | | | |
| dissemination | | | | | | | | | | | | | | | | | | | | | | | | |
| Exploratory Air | n: | Enga | ige n | rovi | ders | to a | scer | tain | imp | eme | ntat | ion s | strat | egie | S | | | | | | | | | |
| Recruit | | | 8 1 | | | | | | | | | | | 8 | | | X | X | X | X | | | | |
| providers | | | | | | | | | | | | | | | | | | <del>-</del> | I - | [ <u>- </u> | | | | |
| Conduct | | | | | | | | | | | | | | | | | | X | X | X | X | | | |
| semi- | | | | | | | | | | | | | | | | | | | 1 | - | - | | | |
| structured | | | | | | | | | | | | | | | | | | | | | | | | |
| interviews | | | | | | | | | | | | | | | | | | | | | | | | |
| Data analysis | | | | | | | | | | | | | | | | | | | | | | X | X | X |
| and | | | | | | | | | | | | | | | | | | | | | | <del></del> | - | <del>-</del> |
| dissemination | | | | | | | | | | | | | | | | | | | | | | | | |
| a | | | | | | | | | | | | | | l | I | 1 | l | L | 1 | l | l | l | | L |

<sup>\*</sup>Participant study participation is only for a total of 6 months after enrollment.

10/31/2022 

#### 8. STUDY ENDPOINTS

## **Primary Endpoint(s)**

• <u>Urinary ITC levels</u> will be measured using HPLC-based cyclocondensation assay<sup>14, 51</sup>, which measures ITCs and metabolites as low as a few picomoles and has been routinely performed in Dr. Tang's laboratory. The results will be adjusted by urinary creatinine level using creatinine assay kits (Caymen, Ann Arbor, MI). <u>Cruciferae intake</u> will be assessed using a questionnaire adapted from Thomson et al.<sup>52</sup> to capture both intake and cooking styles.

## **Secondary Endpoint(s)**

- Gene expression will be evaluated via RNA-seq as a surrogate for intermediate efficacy, conducted at Roswell Park's Genomics Shared Resource using NextSeq500 platform (Illumina Inc.). We have worked with the Genomics core to optimize the extraction of RNA samples from urine. With the addition of TRIzol<sup>TM</sup> right before the storage of the cell pellet samples, we were able to extract sufficient amounts of RNA and generate high quality RNA-seq data. <u>Dietary intake</u> will be evaluated by three non-consecutive 24-hour dietary recalls (two weekdays, one weekday) conducted by trained staff using the interview-administered Nutrition Data System for Research (NDSR)<sup>53</sup>.
- Additional urinary metabolites and potential biomarkers will be explored using proteomic and/or metabolomic approaches.

## **Exploratory Endpoint(s)**

• Our exploratory endpoint will be identification of barriers, facilitators, and other process-related measures relevant to informing the implementation of an evidence-based cruciferae intervention within clinical practice.

#### 9. DESIGN

We will use a Hybrid I implementation randomized-controlled design to simultaneously gather outcomes regarding the intervention's feasibility and process data to facilitate wide-spread implementation and dissemination of the intervention into clinical practice if the intervention is effective. A total of 80 patients will be recruited on a rolling basis. Forty will be randomized to intervention and 40 to control.

10/31/2022 

#### 10. TREATMENT

The planned evidence-based behavioral intervention using techniques associated with effective dietary change in older adults (Table 1): problem solving, plan social support, goal setting, follow-up prompts, and provide feedback. The 6-month intervention will likely consist of the following, although aspects of the intervention may change based on data from the adaptation process: 1) Mailed educational materials about the importance of consuming cruciferae, how to maximize

urinary ITC levels, serving size goals, the importance of selfmonitoring, and strategies to increase intake, along with booklets to record daily cruciferae intake; 2) One live phone call (~45-60 minutes) delivered two weeks after mailing materials to verify understanding of the educational information and help participants complete a personalized action plan where participants will identify barriers and facilitators (e.g. social support) to meet identified goals (problem solving); 3) Interactive Voice Response (IVR) phone messages that will begin by asking participants to input the servings of cruciferae consumed the previous week (follow-up prompt). Depending

| ٠. | | | | |
|---|---|---|---|---|
| | Table 1. Interv | vention Components | | |
| | Intervention | Intervention content/ | SCT Construct | CAB adaptation |
| ) | component | behavior technique | | |
| ı | Educational | <ul> <li>Relationships between</li> </ul> | <ul> <li>Knowledge</li> </ul> | <ul> <li>Barriers and</li> </ul> |
| , | Materials | cruciferae, ITC yield,<br>and bladder cancer | <ul> <li>Outcome<br/>expectations</li> </ul> | facilitators to meeting goals, |
| • | | <ul> <li>Type of vegetable,</li> </ul> | Behavioral skills | examples from BCS |
| ) | | cooking methods, and | <ul> <li>Barriers and</li> </ul> | day-to-day life, |
| 3 | | timing of intake for<br>maximum ITC exposure | opportunities | strategies to meet goals, visuals |
| 2 | | Program goal of 1 | Intentions | pleasing to BCS |
| า | | serving of cruciferae per | | |
| ì | | day/Goal setting | | |
| ֓֓֓֓֓֓֓֓֓֓֓֓֓֜֜֓֓֓֓֓֓֡֜֜֓֓֓֓֡֓֜֡֓֓֓֓֓֡֜֡֡֓֓֡֡ | | Keeping track of acryings exten per day | | |
| 1 | 1 Live | servings eaten per day | Manual adam | Detential much laws |
| 5 | phone call | Review materials Action plan to proof | Knowledge Debouierel skille | Potential problems and subsequent |
| l | priorie can | <ul> <li>Action plan to meet<br/>program goal/problem</li> </ul> | <ul><li>Behavioral skills</li><li>Barriers and</li></ul> | and subsequent solutions for BCS to |
| 3 | | solving | opportunities | meet goals |
| | | 3 | Self-efficacy | J |
| | 11 | Participants enter by | <ul> <li>Barriers and</li> </ul> | How to structure the |
| 1 | Interactive | phone servings of | opportunities | cruciferae intake |
| ı | Voice<br>Response | cruciferae eaten in prior | Reinforcement | form to make it easy for BCS to use |
| ) | (IVR) phone | week/follow-up prompt • Automated feedback | Self-efficacy | |
| • | calls | based on the extent | | Construct library of<br>IVR feedback |
| ٦ | Jano | | | |
| , | | goal/ feedback | | to BCS |
| 5 | calls | participants met program | | messages relevant |

on number of servings participants input, they will be routed to one of three paths: a) meeting goals, b) not meeting goals but has some progress, c) no progress. Participants on each path will receive a tailored phone message (provision of feedback) selected from a library of messages to enable participants to meet or maintain their cruciferae goal. A total of 11 IVR calls will be delivered weekly for the first three weeks and then bi-weekly for the remainder of the 6-month intervention.

#### 11. PROCEDURES INVOLVED

## Aim 1: Develop an evidence-based behavioral intervention to increase cruciferous vegetable intake

**Adaptation.** Working with our Community Advisor Board (CAB) consisting of a urologist, clinic staff, and BCS, we will refine current evidence-based vegetable interventions to develop a novel dietary intervention for BCS. We will use a systematic process consisting of information gathering, discussion groups, and mock intervention delivery. Dr. Yeary, who has extensive experience adapting evidence-based behavioral interventions for diverse groups, will lead the team through a four-stage adaptation process based on the Barrera and Castro framework<sup>42</sup> and PEN-3 model for cultural adaptation<sup>43</sup>. We will: 1) identify relevant factors to increase cruciferae intake in BCS; 2)

10/31/2022 

use the PEN-3 model to review each of the intervention's components (e.g. graphics, terminology, saliency of behavioral messages); 3) administer the revised intervention to the CAB for their feedback; and 4) refine the intervention based on Step 3. We will also present the program to the BCS group meeting at Roswell Park to ensure the intervention is salient to our target population by demographic characteristics. The final product will be a 6-month cruciferae intervention for BCS grounded in Social Cognitive Theory (SCT). CAB members will each be compensated \$100 per meeting (up to three meetings), each meeting lasting about 1.5 hours and will be conducted via phone or computer. CAB members (bladder cancer survivors) may be asked to complete a structured interview over the phone and complete some demographic questions about themselves. Structured interviews will last approximately 60 minutes and CAB members will be paid \$50 for completion of the structured interview. See Appendix K for Study Information Sheet for CAB members and Appendix L for CAB Interview Guide)

**Intervention Design.** Drawing from the large body of literature on evidence-based behavioral fruit and vegetable interventions, the intervention will likely include components used by Wolf et al. 44 and Djuric et al. 45 (i.e. educational materials, phone calls, written plans, self-monitoring), who significantly increased vegetable intake among participants whose demographic characteristics mirror the majority of our target population (i.e. age 65 and older, diverse, male). The following evidence-based behavioral techniques associated with effective dietary change in older adults<sup>46</sup> will also be incorporated (Table 1): problem solving, plan social support, goal setting, follow-up prompts, and provide feedback. The 6-month intervention will likely consist of the following, although aspects of the intervention may change based on data from the adaptation process: 1) Mailed educational materials about the importance of consuming cruciferae, how to maximize urinary ITC levels, serving size goals, the importance of self-monitoring, and strategies to increase intake, along with booklets to record daily cruciferae intake (See Appendix P); 2) One live phone call (~45-60 minutes) delivered two weeks after mailing materials to verify understanding of the educational information and help participants complete a personalized action plan where participants will identify barriers and facilitators (e.g. social support) to meet identified goals (problem solving) (See Appendix Q); 3) 11 Interactive Voice Response (IVR) phone messages that will begin by asking participants to input the servings of cruciferae consumed the previous week (follow-up prompt). Depending on number of servings participants input, they will be routed to one of three paths: a) meeting goals, b) not meeting goals but has some progress, c) no progress. Participants on each path will receive a tailored phone message (provision of feedback) selected from a library of messages to enable participants to meet or maintain their cruciferae goal. A total of 11 IVR calls will be delivered weekly for the first three weeks and then bi-weekly for the remainder of the 6-month intervention. The CAB will give specific feedback about visual material that would be the most appealing to BCS, specific barriers survivors may have to meet study goals, examples from survivors' day-to-day lives to incorporate in the materials, specific phrases and language to clearly convey the content, strategies to consume cruciferae with minimum effort, and tailored wording or terms that would optimize the participants' response to IVR feedback. We selected phone and mail modalities of intervention delivery because: 1) Phone-based dietary interventions are effective<sup>35</sup>; 2) phone-based interventions are more feasible to implement on a wide-scale compared to face-to-face interventions, which take more resources<sup>47</sup>; 3) IVR would be more cost-effective for a clinic to incorporate within its system vs. dedicating staff to provide frequent calls. Further, IVR is more feasible and accessible to the target population because BCS are typically older (average age at diagnosis is 73 years old); use of text messaging is lower among older groups, with less than half reporting email or text messaging for communication<sup>48</sup>.

10/31/2022 

**Control intervention.** Participants in the control arm will receive mailed materials about general fruit and vegetable intake intervention based on published NCI (https://cancercontrol.cancer.gov/ocs/). The control intervention will utilize the same delivery method (i.e. mailed educational materials, live phone call, IVR calls) and follow the same contact schedule as the treatment schedule (See Appendix P and Appendix Q). We intend to compare our tailored cruciferae program with general program on increase of fruit and vegetable intake. We anticipate minimal contamination between intervention and control because BCS will be recruited throughout our catchment area and our intervention will be delivered individually with each BCS.

**Personnel Training.** Dr. Yeary will utilize her extensive experience in training others in the delivery of behavioral interventions to train project staff to implement the intervention. A training-of-trainers model that incorporates didactic education, trainee practice, and written and verbal feedback will be used. Training will build knowledge about behavior change promotion, with a specific emphasis on delivering the live phone call with fidelity, utilizing participant booklets to program the IVR messages, and communicating effectively with participants about health. The training will conclude with project staff demonstrating mastery of concepts through mock phone sessions and live phone calls, and accurate programming based on booklet data received. Project staff will be asked to complete a checklist of topics to monitor intervention fidelity.

## Aim 2: Conduct a feasibility pilot of our evidence-based dietary behavioral intervention

**Study Design.** We will use a Hybrid I implementation randomized-controlled design to simultaneously gather outcomes regarding the intervention's feasibility and process data to facilitate wide-spread implementation and dissemination of the intervention into clinical practice if the intervention is effective. A total of 80 patients will be recruited on a rolling basis. Forty will be randomized to intervention and 40 to control.

Participant Recruitment. Eligibility criteria include: 1) English speaking; 2) diagnosed with stage Tis, Ta, or T1 bladder cancer; 3) resides in the Western New York (WNY) catchment area (Niagara, Orleans, Genesee, Erie, Wyoming, Chautauqua, Cattaraugus, and Allegany counties); 4) did not receive a partial or radical cystectomy; 5) does not have a prior cancer diagnosis within 12 months of their bladder cancer diagnosis 6) does not have a subsequent more advanced bladder cancer diagnosis; and 7) (for Roswell Park Cancer Registry only) diagnosed 2016-2018, 2019current. We chose not to include current cruciferae intake as an eligible criterion because prior studies have reported that BCS consumed an average of 0.44-0.45 servings per day<sup>12, 26</sup>, less than half our recommended amount. Using ICD-O-3 codes provided, Dr. Kuliszewski of the NYSCR will lead her staff to identify qualifying patients from their database based on the study's eligibility requirements. The NYSCR has identified 199 cases that meet the study's eligibility criteria in 2018 and anticipate at least 400 eligible cases in total in 2018 and 2019. A total of 250 eligible patients will be contacted to enable researchers to recruit from a pool of at least 100 patients. In prior studies, 52.4% to 62.5% of patients contacted by the NYSCR agreed to be contacted by researchers for study consent. The NYSCR will send a letter to the physician of record for selected cases notifying that the patient was identified for the study, requesting that the NYSCR be notified if the patient is unable or ineligible to participate in the study, and requesting information about the case's primary care physician if different from the contacted physician. If no contraindication has been received from the physician or if the physician has not responded within 3 weeks, the NYSCR will send an informational packet to the patient. The packet will contain: 1) a letter with study information; 2) a participant information sheet; and 3) a release of information consent form. After two weeks without response, a reminder packet will be sent and followed with up to five phone

10/31/2022 

calls. If the NYSCR can't reach the patient, the patient will be considered a refusal. The NYSCR's materials and procedures will be reviewed by the New York State Department of Health IRB. For patients who agree to be contacted about the study, the NYSCR will securely share the patient's name, contact information, and information about their diagnosis with the Roswell study team. For the Roswell Park Cancer Registry, study staff will consult with Roswell Park urologist to determine if the patient is unable or ineligible to participate in the study. The patients accessioned from the Roswell Park Cancer Registry will be contacted by letter (See Appendix T) asking them to participate in the study. Study staff will follow-up with potential participants to determine whether they received the letter and if they are interested in participating. We estimate that from the pool of at least 100 patients who consent to be contacted, we will be able to obtain informed consent from at least 80 patients (80%). The Roswell study team will share information with the NYSCR team on the patients who agree to participate in the study, as well as any information obtained from study participants that does not match the information provided from the NYSCR database (e.g., race, ethnicity).

Participant Data and Sample Collection Procedures. Research staff will contact patients who have agreed to be contacted by phone, whereby they will provide a general study overview and conduct a screening interview to confirm eligibility. The consent form will be mailed out to patients prior to the consenting discussion. We will ask the patient to mail back the consent form with the appropriate signatures. We will also provide an additional copy of the consent form for their records. We will include a paid postage pre-addressed envelope for the patient to mail back the signed consent form to study staff. Baseline Data Collection will be conducted within four weeks prior to intervention start. The Data Collector, masked to treatment assignment, will conduct telephone surveys with participants and directly enter participants' responses into pre-programmed data collection forms in REDCap<sup>49, 50</sup>. Surveys will cover sociodemographic variables, faith and spirituality beliefs, dietary, and cruciferae intake (Appendix F). Additionally, 24-hour dietary recalls will be conducted and instructions (Appendix M) and a reference guide (Appendix N) will be mailed out to participants prior to their scheduled recall interview. Participants will also be mailed out track books to help keep track of their fruit and/or vegetable intake during the intervention (Appendix R). Follow-up Assessment (Appendix G1) will be conducted at 6 months following the same protocol as the baseline assessment (Appendix F). Participants will receive \$100 for completing the baseline and 6-month follow-up assessments. In addition, we will ask participants' feedback on the intervention (Appendix G2) as part of the Follow-Up Assessment (Appendix G1). The feedback questions (Appendix G2) will be given to those in the cruciferous arm only. For cruciferous arm study participants that have completed the 6-month follow-up assessment as of the March 21, 2022 Protocol revision, the study participants will be called back to complete the feedback questions (Appendix G2). These study participants will first be sent an information sheet (Appendix W) regarding the additional feedback questions before being called. When they are called regarding the study feedback questions, they will provide verbal consent before proceeding with answering the feedback questions.

Urine Sample Collection will be conducted at baseline and 6-months. Participants will be instructed to collect first-void urine continuously for three days, which will provide a more reliable measurement than one-spot urine samples. A specially designed urine collection device consisting of a 10-mL container and sponge with a plastic holder will be used, which does not impact urinary ITC measurement and has been used in the Be-Well study with documented ease of collection and minimal shipment burden. Staff will mail urine collection kits and instructions (Appendix C) to participants. Given that recent behaviors may have a large impact on urinary ITC levels,

10/31/2022 

participants will be asked to complete a brief 2-page specimen collection survey (Appendix D) on medical and lifestyle status in the past two days. They will then return the survey and urine samples to Roswell Park in the provided shipping box with biohazard labels and ice packs via pre-paid overnight shipping service. Once received, the urine will be spun down from the sponge, aliquoted, and stored at -80°C at Dr. Li Tang's lab (x8247) at Roswell Park. The urine aliquots will be assayed at Dr. Tang's Lab for ITC analysis using HPLC-based cyclocondensation assay.<sup>64</sup> This method is able to accurately measure as low as a few picomoles of ITCs and their metabolites. Dr. Tang's lab has experience and expertise in running this assay.<sup>65</sup> and will process the urine samples and perform the measurements. The results will be adjusted by urinary creatinine level, which will also be performed in the laboratory, using a commercially available creatinine assay kit (Caymen, Ann Arbor, MI). The cell pellets from three urine samples per participant will be combined and delivered to Genomics Shared Resources at Roswell Park for RNA-seq analysis in a batch. Additional urinary metabolites and potential biomarkers will be explored using proteomic and/or metabolomic approaches. All assays will be conducted on the stored urine samples. Neither new urine sample collection nor patient contact will occur.

## Exploratory Aim: Engage providers to ascertain specific clinic-level implementation factors

We will ask intervention participants to nominate physicians to participate in a short 15-minute semi-structured interview. Research staff will mail an invitation letter to nominated physicians that will include an information sheet (Appendix J), opt-in/opt-card card, and stamped reply envelope. Within 2-weeks, physicians who do not respond will be contacted by phone, fax, or email with no more than 5 attempts. Participating physicians will receive \$100. Physicians who verbally consent to participate will be asked to refer other physicians to the study. CAB members will also utilize their networks to nominate physicians for staff to contact.

We will conduct brief 15-minute semi-structured interviews using an interview guide. The guide will give physicians a brief overview of our cruciferae intervention. Research staff will then ask questions regarding facilitators and barriers of intervention adoption within clinical practice<sup>37</sup>. Staff will ask physicians the needed implementation strategies to sustain the intervention post research funding, in addition to intervention modifications to maximize sustained clinic adoption<sup>37</sup>.

#### 12. WITHDRAWAL OF SUBJECTS

Participants can stop their participation at any time. Participants may refuse to answer any question and they may leave the study at any time.

#### 13. RISKS TO SUBJECTS

For the survey portion of the study, involvement in this study does not involve any physical risk. The possible risks might be feeling uncomfortable answering questions.

There are no known risks associated with providing a urine sample other than a potential loss of confidentiality.

#### 14. POTENTIAL BENEFITS TO SUBJECTS

Participants in the intervention and feasibility scale-up pilot may benefit from study participation by improving dietary habits and/or reducing bladder cancer recurrence. The information gained may also help other bladder cancer patients in the future. Participants will receive \$100 for completing each assessment—the study will ask participants to complete baseline (see Appendix

10/31/2022 

F) and 6-month follow-up assessments (See Appendix G1). Thus, participants will be able to receive up to \$200 total in assessments. Participating physicians will receive \$100 for the interview.

#### 15. DATA AND SPECIMEN BANKING

All questionnaire data will be stored in REDCap or in a locked file cabinet. REDCap is a secure application supported by Partners Research Computing, Enterprise Research Infrastructure & Services (ERIS). ERIS has all the necessary physical and operational securities in place to meet or exceed Federal and State security and privacy regulations for data transmission and storage using REDCap. Data will only be removed when coded, entered, or audited. The urine samples will be processed and stored at Dr. Tang's laboratory and a dataset will be created to track and record the results obtained from laboratory assays on urine samples. The dataset will only contain study IDs without any personal identifiable information. The file that contains the link between study ID and subject identifiable information will be maintained separately and can only be accessed by Drs. Yeary and Tang and will never be released to any laboratory staff.

#### 16. MEASUREMENT OF EFFECT

#### **Solid Tumors**

N/A

#### **Hematologic Tumors**

N/A

#### **Other Response Parameters**

We will assess the treatment intervention's effect on the consumption of cruciferae vegetables and ITC yield, as specified under the heading, "STUDY ENDPOINTS". We will also assess changes in gene expression via RNA-Seq, so as to identify a panel of genes that respond specifically to consumption of cruciferae vegetables as specified in the section of STUDY ENDPOINTS. It is well known that isothiocyanates in cruciferae vegetables alter multiple signaling pathways. Therefore, the identified panel of genes can be used as biological biomarkers to understand how individuals respond to the consumption of cruciferae vegetables, and more importantly, be used as biomarkers to monitor the effect of cruciferae vegetables.

#### 17. SAFETY EVALUATION

#### **Reporting Unanticipated Problems.**

Unanticipated problem reporting will begin at the time of participant consent. The Reportable New Information (RNI) Form will be submitted to the Roswell Park Clinical Research Service (CRS) Quality Assurance (QA) Office within 1 business day of becoming aware of the Unanticipated Problem. After review, CRS QA Office will submit the RNI to the IRB.

When becoming aware of new information about an Unanticipated Problem, the updated information will be submitted to the CRS QA Office with an updated RNI Form. The site Investigator or designated research personnel will report all unanticipated problems to the IRB in accordance with their local institutional guidelines.

10/31/2022 

#### 18. DATA MANAGEMENT AND CONFIDENTIALITY

Individual confidentiality concerning study data and measurements will be ensured through the following ways: Participant data will not be identified by name (using only an identification number for identification), all data and records in locked storage areas accessible only to project staff, and password protected computer data files. Participants will not be personally identified in any scientific reports generated by the study. All results will be presented in aggregate form. All project staff will undergo training and ongoing continuing education about methods to protect confidentiality. All project staff will complete Human Subject Training Requirements.

We have contracted with an outside company Above Ground Development (AGD) to conduct the 11 Interactive Voice Response (IVR) phone messages that participants receive as part of the intervention. The study staff will share the following information with AGD that includes participant's name, date of birth and contact phone number. This PHI information will be entered into the secure web portal (user interface) and ALL data will be stored with AGD on a secure HIPAA Compliant server.

Safety of subjects. Data safety and monitoring will be overseen by Drs. Yeary and Tang. The proposed study is considered extremely low risk. Adverse events will be monitored routinely during questionnaire and data collection and participants will be instructed to contact study personnel for any issues. Monthly meetings with Dr. Yeary, Dr. Tang, and the Project Coordinator (Ms. Harfouche) will also be held to evaluate the status of study subjects. Dr. Qiang Li, a Board Certified Bladder Cancer Surgeon, will provide guidance and supervision regarding all the reported side effects or potential symptoms possibly related to study participation. Adverse events will be labeled as to whether attributed to behavior intervention or not, classified as mild, moderate, severe, life threatening, or causing death, and reported to Roswell Park IRB and NIH under Institute guidelines. We will track reporting of adverse events in the REDCap study database. All clinical trials at Roswell undergo yearly review by an independent Data Safety Monitoring Board.

Collection of Data and Biospecimens. Project staff will collect questionnaire data from research subjects by telephone interview, as dictated by study protocol. Questionnaire data will be directly entered into REDCap, a secure web application for building and managing online surveys and databases. Only study identification number (Study ID) will be entered when the data are collected. All data collected by research assistants are considered part of the subject's confidential record. REDCap is a secure application supported by Partners Research Computing, Enterprise Research Infrastructure & Services (ERIS). ERIS has all the necessary physical and operational securities in place to meet or exceed Federal and State security and privacy regulations for data transmission and storage using REDCap. All data will remain confidential. A file will be separately maintained that associates the subject name with that subject's study ID. This file will remain in a locked file cabinet and will not be stored with the actual study data. The urine samples will be collected by the participants at home and directly shipped to Roswell Park using prepaid and addressed shipping labels. All urine samples will be labeled with assigned study IDs only and no personal information will be provided.

#### Storage of Collected Data and Biospecimens.

N/A

**Data Entry Requirement.** All data will be coded prior to entry. Any ambiguity in the response to a question will be brought to the attention of Ms. Harfouche for clarification. If Ms. Harfouche is

10/31/2022 

unsure how to code the response, the matter will be brought to the attention of Drs. Yeary, Tang, and consulted with the statistician (Dr. Yu). Ms. Harfouche will maintain a log, so that future occurrences of problems will be handled in the same manner.

The data entry system will require a login identification and password in order to gain access to the data. Where appropriate, validation and range rules will be applied to the actual entry fields. Only Dr. Yeary, Dr. Tang, Dr. Yu, and data entry personnel will be able to view the data in its raw state. All other authorized personnel will view data via forms and reports in aggregate form created by Dr. Yeary, Dr. Tang, and Dr. Yu.

Access to Cleaned Computer Data. Only Drs. Yeary, Tang, and Yu can give permission for the release of aggregated study data. No confidential information will be released without permission.

#### 19. STATISTICAL PLAN

**Patient.** We will use SAS for data analysis and R for RNA-seq data. We will generate descriptive statistics and assess group differences at baseline and examine treatment drop-out and missing data patterns' impact on treatment effects. We will calculate summary statistics and compare study endpoints and patient baseline characteristics by treatment group using independent sample t-tests and Fisher's exact tests. We will summarize changes between pre- and post-intervention for both arms and calculate point estimates and their corresponding 95% confidence intervals. We will analyze between-group differences in the change of outcome variables between baseline and postintervention using analysis of covariance (ANCOVA). The intervention group will be used as factors and the baseline variables used as covariates. Within-group difference between two timepoints will be compared by paired sample t-tests, while between-group differences at each timepoint will be compared by independent sample t-tests or Wilcoxon rank sum tests. RNA-seq data will be processed and quality-checked by the Bioinformatics Shared Resource at Roswell Park; sample relationships will be explored using sample clustering and principle component analysis. We will use DESeq258 to identify significantly differentially expressed (SDE) genes and conduct pathway analysis with GSEA59 using rank-based gene list from SDE analysis. All tests will be two-sided at the significance level of 0.05. We will use the Benjamini-Hochberg's method to calculate the false discovery rate for gene expression.

**Physician.** Interviews will be audio-recorded, transcribed verbatim, checked for accuracy and entered into a software program for the management of text data (e.g. NVivo 12). We will code transcripts using content analysis. Coding decisions and emergent findings will be discussed until an agreement is reached<sup>57</sup>.

#### **Sample Size Determination**

<u>Patient</u>: With n=40 for each group, the ANCOVA can achieve 80% power to detect a difference of 0.57 within-group standard deviations (SDs) between groups assuming the correlation of post-intervention and baseline outcome is R2=0.2. Data from the Be-Well study reports a within-group SD of 8.9  $\mu$ M for urinary ITCs and 62 g/day for cruciferae intake; thus, we can detect a difference equivalent to 5.1  $\mu$ M in urinary ITC and 35.3 g/day of cruciferae intake between groups. The intervention's goal is to increase urinary ITC levels from the baseline of 4.4  $\mu$ M to the desirable biological dose of 10  $\mu$ M and cruciferae intake from the baseline of 52.7 gram (0.7 serving) to at least 75 gram (a typical serving size) at 6-month follow up. Given the generally lower cruciferae intake observed in other BCS studies (around 0.44-0.45 serving, equivalent to 33-34 gram per day)<sup>11, 26</sup>, the proposed study will have sufficient power to detect our projected differences.

10/31/2022 

<u>Physician</u>: We will recruit up to 20 physicians to ensure data saturation<sup>61</sup>. Among clinicians involved in cancer treatment, enrollment rates between 46.3%-92% have been reported<sup>60, 62, 63</sup>, with one study reporting an enrollment rate of 48% among clinicians involved in bladder cancer treatment<sup>62</sup>. Out of the 80 participants enrolled in our intervention, we anticipate 40 to nominate their physicians and expect to receive referrals for 5 additional physicians from enrolled physicians and 5 physicians nominated by our CAB. Given an anticipated enrollment rate of 48%, we anticipate recruitment of 20 physicians.

## Randomization

Subjects will be randomized in a 1:1 fashion to the control arm and interventional arm using permutated block randomization. We will employ random block sizes of 4 and 2. Randomization will be carried out by the Department of Biostatistics and Bioinformatics.

#### **Demographics and Baseline Characteristics.**

Descriptive statistics (as appropriate: n, percent, mean, median, min and max) will be used to summarize demographic and baseline characteristics. The patient characteristics will also be summarized by treatment group. The baseline characteristics between groups will be compared by independent sample t-tests and Fisher's exact tests as appropriate.

## Primary Analysis.

For primary analysis, the aim is to investigate the between-group differences in the change of urinary ITC levels and cruciferae intake between baseline and post-intervention. The comparison of change from baseline will be made utilizing analysis of covariance (ANCOVA) and F-tests ( $\alpha$ =0.05). The intervention group will be used as factors and the baseline variables used as covariates. A coefficient for interventional group that is significantly greater than 0 will indicate that the intervention increases the ITC levels or cruciferae intake. Within-group difference between two time-points will be compared by two-sided paired sample t-tests, while between-group difference at each time-point will be compared by two-sided independent sample t-tests ( $\alpha$ =0.05). Since this is a pilot feasibility study, no adjustment for multiple comparisons will be planned.

#### Secondary Analyses.

The aim of secondary analysis is to investigate the difference in gene expression patterns between two groups. Three urine samples per participant will be collected at baseline and month 6, and the cell pellets from three urine samples per participants will be combined and subject to RNA-seq. RNA-seq data will be processed and quality-checked by Bioinformatics Shared Resource at Roswell Park; sample relationships will be explored using sample clustering and principle component analysis. We will use DESeq to identify significantly differentially expressed (SDE) genes and conduct pathway analysis with GSEA using rank-based gene list from SDE analysis. All tests will be two-sided at significance level of 0.05. We will use the Benjamini-Hochberg's method to calculate the false discovery rate (FDR) for gene expression.

The additional metabolites and biomarkers will be analyzed using the same approach as in primary analysis. The univariate distributions of these variables will be examined, and appropriate transformations may be applied before analysis. Benjamini-Hochberg's method to control the FDR.

10/31/2022 

#### **Exploratory Analysis.**

Qualitative methodology using content analysis will be used to ascertain physician barriers and facilitators to the intervention's implementation within clinic settings.

## **Safety Analysis**

N/A

#### **Interim Analysis**

None

## 20. PROVISIONS TO MONITOR THE DATA TO ENSURE THE SAFETY OF SUBJECTS

N/A

#### 21. VULNERABLE POPULATIONS

N/A

#### 22. COMMUNITY-BASED PARTICIPATORY RESEARCH

The study does not use a "pure" community-based participatory research approach but does include community engagement, which will include engagement of a Community Advisory Board to develop the cruciferae intervention.

#### 23. SHARING OF RESULTS WITH SUBJECTS

Aggregate study results will be disseminated to the project's Community Advisory Board, the Bladder Cancer Survivorship Group at Roswell Park Comprehensive Cancer Center, the New York State Department of Health Cancer Registry, and to participating patients and health care providers who consented to be part of the research, written informed consent for participating patients and verbal consent for participating health care providers. Study participants will be mailed aggregate study results with no personal identifiers. Study results will also be disseminated to academic and practice audiences through scientific papers and conferences.

#### 24. SETTING

Participant Recruitment. NYSCR will send a letter to the physician of record for selected cases notifying him/her that the patient was identified for the study, requesting that NYSCR be notified if the patient is unable or ineligible to participate in the study, and requesting information about the case's primary care physician if different from the contacted physician. If no contraindication has been received from the physician or if the physician has not responded within 3 weeks, the NYSCR will send an informational packet to the patient. The packet will contain: 1) a letter with study information; 2) a participant information sheet; and 3) a release of information consent form. After two weeks without response, a reminder packet will be sent and followed with up to five phone calls. If NYSCR can't reach the patient, the patient will be considered a refusal. The NYSCR's materials and procedures will be reviewed by the New York State Department of Health IRB. For patients who agree to be contacted about the study, the NYSCR will securely share the patient's name, contact information, and information about their diagnosis with the Roswell study team. For the Roswell Park Cancer Registry: study staff will consult with Roswell Park urologist

10/31/2022 

to determine if the patient is unable or ineligible to participate in the study. The patients accessioned from the Roswell Park Cancer Registry will be contacted by letter (See Appendix T) asking them to participate in the study. Study staff will follow-up with potential participants to determine whether they received the letter and if they are interested in participating. We estimate that from the pool of at least 100 patients who consent to be contacted, we will be able to obtain informed consent from at least 80 patients (80%). Research staff will contact patients who have agreed to be contacted by phone, whereby they will provide a general study overview and conduct a screening interview to confirm eligibility. The consent form will be mailed out to patients prior to the consenting discussion. We will ask the patient to mail back the consent form with the appropriate signatures. We will also provide an additional copy of the consent form for their records. We will include a paid postage pre-addressed envelope for the patient to mail back the signed consent form to study staff. To assist with study retention, we will ask participants for contact information to be used in follow-up. The Roswell study team will share information with the NYSCR team on the patients who agree to participate in the study, as well as any information obtained from study participants that does not match the information provided from the NYSCR database (e.g., race, ethnicity).

The process for contacting the patient, including the number of contact attempts, the letter text and/or phone script, the consent form, the data to be collected, and information on any incentives for participation will be reviewed by the NYSCR, New York State Department of Health (NYSDOH), and the NYSDOH IRB prior to the initiation of any patient/proxy contact. In addition, the research team will follow all NYSDOH procedures in conducting their study, including the following procedures:

- 1. All written materials must include contact information for people who can answer questions about the research and participant rights.
- 2. Patient consent to participate must be obtained.
- 3. If a patient asks to be removed from current or future research studies, this information must be sent within two weeks to the NYSCR, so that the patient's record can be flagged and the patient added to a "Do Not Contact" list.
- 4. Researchers must immediately report any complaints about the study or the release of patient information to the Director of the NYSCR and to the Administrator of the NYSDOH IRB.

If changes are made to any recruitment materials or processes after NYSDOH departmental and IRB approval, an IRB amendment must be submitted and approved before the changed materials may be used.

Before receiving case-level Registry data, the Principal Investigator for a research study will be required to read and sign a Research Data Use Agreement. This contract describes limitations on the use of the data, as well as restrictions on the dissemination of findings, use of personal identifiers, and contact with patients identified through data provided by the NYSCR. All staff working with confidential data, or with possible access to confidential information from the data, are required to have current IRB training certification and to sign a Confidentiality Pledge. The Research Data Use Agreement and Confidentiality Pledge documents can be obtaining by emailing the NYSCR at nyscr@health.ny.gov.

10/31/2022 

Researchers must agree to maintain the confidentiality of identifiable data received from the NYSCR. Identifiable data include any information that would permit, directly or indirectly, the identification of any individual. When applying to use the data, researchers should indicate how the data will be stored as well as how and when they will dispose of the data after the study is completed. In addition, researchers must attest that: 1) no data will be published or released in any form where a particular individual or establishment is directly or indirectly identifiable; 2) identifiable data obtained from the NYSCR will be used only for the proposed study; 3) identifiable information obtained from the NYSCR will not be released to anyone or any institution without prior written approval by the NYSDOH; and 4) any publication or report produced using the data will acknowledge the source of the data. In the event of a breach of confidentiality, researchers must notify the Director of the NYSCR as soon as possible but no later than two business days after learning of the breach.

**Physician Recruitment.** Research staff will mail an invitation letter to nominated physicians that will include an information sheet (Appendix J), opt-in/opt-card card, and stamped reply envelope. Within 2-weeks, physicians who do not respond will be contacted by phone, fax, or email with no more than 5 attempts. Participating physicians will receive \$100. Physicians who verbally consent to participate will be asked to refer other physicians to the study. CAB members will also utilize their networks to nominate physicians for staff to contact.

#### 25. PROVISIONS TO PROTECT THE PRIVACY INTERESTS OF SUBJECTS

Only de-identified data will be accessed and recorded. Data files will be coded numerically and assigned to each participant. Information gathered from participants will remain anonymous and will be referred to only by general category. There will be no reference by name to any participant in any qualitative or quantitative data capture. No patient identity will be disclosed in the event of publication or sharing of data.

For physicians, the study will not collect any identifiers from the physician. The data collected from physician participation would be qualitative only. Therefore, for the physicians only, we are requesting a waiver of HIPPA Authorization.

The data collected from this study will be organized by a unique identification number assigned to the participant so that their identity will be available only to project staff and will remain completely confidential. The data manager, study staff, Co-Is and PI of the study will have access to the data records.

All study records will be kept electronically in Roswell Park maintained and secured equipment. The electronic data records will be saved and secured on the Roswell Park shared server. Survey data will be filed in a locked cabinet located in 311 Carlton House and will not be taken off Roswell Park premises. The data will be kept in a locked room where it will remain for approximately five years following the completion of the project.

#### 26. RESOURCES AVAILABLE

The project will be co-led by Drs. Yeary and Tang, who will serve as multiple PIs on the project. Drs. Yeary and Tang will make joint decisions regarding the project. They will collaborate with the New York State Department of Health Cancer Registry and the Community Advisory Board in making collaborative decisions regarding the project. Communication between the PIs will be done in person, through video conferencing (e.g. Zoom, Webex), phone, and email.

10/31/2022 

The project will be coordinated by the Ms. Harfouche (Roswell Park) and all project data will be collected by the data collector (Ms. Dauphin). All data will be entered and managed by the database manager (Ms. Harfouche). All quantitative data analyses will be done by Dr. Yu.

Drs. Yeary and Tang will lead the completion of the study's aims, with Dr. Yeary focused on the intervention aspects of the study, and Dr. Tang focused on the biological aspects of the study. Dr. Yeary and Dr. Tang will oversee collaboration with the Community Advisory Board (including Dr. Qiang Li) in developing the intervention. Dr. Yeary will oversee the intervention's implementation and evaluation. Dr. Yeary will oversee Ms. Harfouche, who will oversee the recruiter (Ms. Dauphin), data collector (Ms. Dauphin), and interventionist (Ms. Clark). Dr. Yeary will train the interventionist to deliver the intervention. Both Drs. Yeary and Tang will work closely with the New York State Department of Health Cancer Registry during the initial stage of recruitment. Dr. Tang will oversee the laboratory work and ensure that the biological specimens are adequately collected, processed, and analyzed. Non-dietary data analysis will be led by Dr. Yeary and Tang, in close collaboration with Dr. Yu. Dietary data analysis will be led by Dr. McCann. Specific Aim 3 will be led by Drs. Yeary and Tang, who will oversee staff to recruit providers and complete provider telephone interviews.

The NYSCR employs a staff of over 50 to collect, process, and analyze reports on about 110,000 diagnosed cases of cancer among New Yorkers each year. The staff includes a 10-member research unit, five of whom hold a doctoral degree. Areas of expertise within this unit include cancer epidemiology, biostatistics, geographic analysis, and information science. The NYSCR has a strong national reputation and provides data to many national and international cancer studies.

The PIs will work with the New York State Department of Health Cancer Registry and the Community Advisory Board to disseminate project results and decide next steps.

#### 27. PRIOR APPROVALS

The NYSCR study team will obtain approval of study materials by the NYSDOH Bureau, Division, Center, and the NYSDOH IRB.

#### 28. COMPENSATION FOR RESEARCH-RELATED INJURY

If the subject believes they have been injured as a direct result of their participation in this research study, they will be advised to notify the Roswell Park Patient Advocate at (716) 845-1365 or the Dr. Karen Yeary at (716) 845-6231 or Dr. Li Tang at (716) 845-8247.

Medical diagnosis and treatment for the injury will be offered, and a determination will be made regarding appropriate billing for the diagnosis and treatment of the injury. A financial counselor (716-845-3161) will be able to provide an explanation of coverage and to answer questions the subject may have regarding study related billing.

The subject is not prevented from seeking to collect compensation for injury related to malpractice, fault, or blame on the part of those involved in the research.

#### 29. ECONOMIC BURDEN TO SUBJECTS

There are no costs associated with participation in the surveys and/or urine collection.

10/31/2022 

#### 30. CONSENT PROCESS

Prior to administration of any assessment, participants are informed of the purpose of the study and told that their participation is voluntary. Participants are also informed that their responses to questions will be kept confidential. If the patient consents verbally, NYSCR or Roswell Park Cancer Registry staff will fill out the consent to be contacted form and document that consent to be contacted was obtained via phone (Appendix H). If the Registry is unable to contact the patient via telephone, and no written response has been received, no other contact will be attempted, and the patient will be considered a refusal. At the end of the two registries work, we estimate that there will be a pool of at least 100 patients that have consented to be contacted by research staff based on response rates from previous studies participated in by the NYSCR. Research staff will then contact patients who have agreed to be contacted by phone, whereby they will provide a general study overview and conduct a screening interview to confirm eligibility.

We are requesting a waiver of written consent documentation at the time of initial call, and prior to receipt of the signed written consent, for purposes of starting the baseline survey (Appendix F). The consent script will be a review of the consent document that is being obtained. The consent form will then be mailed out to patients. We will ask the patient to mail back the consent form with the appropriate signatures. We will also provide an additional copy of the consent form for their records. We will include a paid postage pre-addressed envelope for the patient to mail back the signed consent form to study staff. The consent form will indicate that a participant retains the right to withdraw at any time and that their health care will not be affected by their decision to participate or refuse to participate in the study. All investigators and project staff will satisfy the required IRB training and certification requirements. The IRB training will be completed during the early months of the project. For recruitment of health care providers, we will ask intervention participants to nominate physicians to participate in short 15-minute semi-structured interviews. Intervention participants will provide informed consent before providing their health care providers' contact information.

For cruciferous arm study participants that have completed the 6-month follow-up assessment as of the March 21, 2022 Protocol revision, the study participants will be called back to complete the feedback questions (Appendix G2). Therefore, these study participants will first be sent an information sheet (Appendix W) regarding the additional feedback questions before being called. When they are called regarding the study feedback questions, they will provide verbal consent before proceeding with answering the feedback questions.

Our Community Advisory Board members will also utilize their networks to nominate physicians for the research team to contact. Research staff will mail an invitation letter to nominated physicians that will include an information sheet (Appendix K), opt-in/opt-out card (Appendix U), and stamped reply envelop. Within 2-weeks, physicians who do not respond will be contacted by phone, fax, or email with at most five attempts. Follow-up contact will use the same invitation letter originally sent out or a phone script mirroring the information sheet (Appendix J). Physicians who decide to participate in the study will provide verbal consent. Physicians who verbally consent to participate will also be asked to refer other physicians to the study. We will recruit up to 20 physicians to ensure data saturation.

The key elements of the informed consent procedure which will be explained to the participants are: 1) the research status of the study- particularly the assessment; 2) the prospect of psychological risk and the provisions for it; 3) the lack of guarantee of benefit from participation in the

10/31/2022 

assessment, 4) the confidentiality of subjects responses to all study measures; 5) the voluntary nature of the study; 6) the receipt of the money for participating in the assessment, and 7) the freedom to withdraw from the study or to refuse to answer specific questions at any time.

Before the survey is conducted, research study staff members will explain: 1) the nature and purpose of the research endeavor, 2) that participation in the research component is completely voluntary, and 3) that data collected from participants will be confidential and assessed, evaluated and reported as aggregate data, as well as precautions taken in the storage of the data.

The Roswell Park Standard Operating Procedures (SOP): Informed Consent Process for Research (HRP-090) will be followed.

#### 31. PROCESS TO DOCUMENT CONSENT IN WRITING

The Roswell Park "SOP: Written Documentation of Consent (HRP-091)" will be followed:

The Investigator (or IRB specified designee) is responsible for obtaining written consent from each patient participant in accordance with GCP guidelines using the approved informed consent form, before any study specific procedures (including screening procedures) are performed. The informed consent form acknowledges all information that must be given to the participant according to applicable GCP guidelines, including the purpose and nature of the study, the expected efficacy and possible side effects of the treatment(s), and specifying that refusal to participate will not influence further options for therapy. Any additional information that is applicable to the study must also be included. Additional national or institutionally mandated requirements for informed consent must also be adhered to. The participant should also be made aware that by signing the consent form, processing of sensitive clinical trial data and transfer to other countries for further processing is allowed. For physician participants, we are requesting a waiver of written consent. We would not collect any identifiers from the physician. The data from physicians would be qualitative only. Physicians will provide verbal consent.

The Investigator or designee shall provide a copy of the signed consent form to the participant and the signed original shall be maintained in the Investigator File. A copy of the signed consent form must be filed in the participant file. At any stage, the participant may withdraw from the study and such a decision will not affect any further treatment options.

#### 32. DRUGS OR DEVICES

N/A

10/31/2022 

#### 33. REFERENCES

- 1. Al-Zalabani AH, Stewart KF, Wesselius A, Schols AM, Zeegers MP. Modifiable risk factors for the prevention of bladder cancer: a systematic review of meta-analyses. Eur J Epidemiol. 2016;31: 811-851.
- 2. Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019;69: 7-34.
- 3. Woldu SL, Sanli O, Lotan Y. Tackling non-muscle invasive bladder cancer in the clinic. Expert Rev Anticancer Ther. 2017;17: 467-480.
- 4. Kamat AM, Hahn NM, Efstathiou JA, et al. Bladder cancer. Lancet. 2016;388: 2796-2810.
- 5. Holmang S, Hedelin H, Anderstrom C, Johansson SL. The relationship among multiple recurrences, progression and prognosis of patients with stages Ta and T1 transitional cell cancer of the bladder followed for at least 20 years. J Urol. 1995;153: 1823-1826; discussion 1826-1827.
- 6. Schulster M. Bladder Cancer Academy 2019 Selected Summaries. Rev Urol. 2019;21: 23-28.
- 7. Kamat AM, Li R, O'Donnell MA, et al. Predicting Response to Intravesical Bacillus Calmette-Guerin Immunotherapy: Are We There Yet? A Systematic Review. Eur Urol. 2018;73: 738-748.
- 8. Barocas DA, Globe DR, Colayco DC, et al. Surveillance and treatment of non-muscle-invasive bladder cancer in the USA. Advances in urology. 2012;2012: 421709.
- 9. Avritscher EB, Cooksley CD, Grossman HB, et al. Clinical model of lifetime cost of treating bladder cancer and associated complications. Urology. 2006;68: 549-553.
- 10. Botteman MF, Pashos CL, Redaelli A, Laskin B, Hauser R. The health economics of bladder cancer: a comprehensive review of the published literature. Pharmacoeconomics. 2003;21: 1315-1330
- 11. Tang L, Zirpoli GR, Guru K, et al. Intake of cruciferous vegetables modifies bladder cancer survival. Cancer Epidemiol Biomarkers Prev. 2010;19: 1806-1811.
- 12. Tang L, Zirpoli GR, Guru K, et al. Consumption of raw cruciferous vegetables is inversely associated with bladder cancer risk. Cancer Epidemiol Biomarkers Prev. 2008;17: 938-944.
- 13. Tang L, Zhang Y, Jobson HE, et al. Potent activation of mitochondria-mediated apoptosis and arrest in S and M phases of cancer cells by a broccoli sprout extract. Mol Cancer Ther. 2006:5: 935-944.
- 14. Tang L, Zhang Y. Mitochondria are the primary target in isothiocyanate-induced apoptosis in human bladder cancer cells. Mol Cancer Ther. 2005;4: 1250-1259.
- 15. Tang L, Zhang Y. Dietary isothiocyanates inhibit the growth of human bladder carcinoma cells. J Nutr. 2004;134: 2004-2010.
- 16. Tang L, Zhang Y. Isothiocyanates in the chemoprevention of bladder cancer. Curr Drug Metab. 2004;5: 193-201.
- 17. Tang L, Li G, Song L, Zhang Y. The principal urinary metabolites of dietary isothiocyanates, N-acetylcysteine conjugates, elicit the same anti-proliferative response as their parent compounds in human bladder cancer cells. Anticancer Drugs. 2006;17: 297-305.
- 18. Munday R, Mhawech-Fauceglia P, Munday CM, et al. Inhibition of urinary bladder carcinogenesis by broccoli sprouts. Cancer Res. 2008;68: 1593-1600.
- 19. Geng F, Tang L, Li Y, et al. Allyl isothiocyanate arrests cancer cells in mitosis, and mitotic arrest in turn leads to apoptosis via Bcl-2 protein phosphorylation. J Biol Chem. 2011;286: 32259-32267.
- 20. Bhattacharya A, Tang L, Li Y, et al. Inhibition of bladder cancer development by allyl isothiocyanate. Carcinogenesis. 2010;31: 281-286.
- 21. Czajkowski SM, Powell LH, Adler N, et al. From ideas to efficacy: The ORBIT model for developing behavioral treatments for chronic diseases. Health Psychol. 2015;34: 971-982.

10/31/2022 

- 22. Baranowski T, Perry CL, Parcel GS. How Individuals, Environments, and Health Behavior Interact: Social Cognitive Theory. In: Glanz K, Rimer BK, Lewis FM, editors. Health Behavior and Health Education: Theory, Research, and Practice. San Francisco: Jossey-Bass., 2003.
- 23. Jung A, Nielsen ME, Crandell JL, et al. Quality of Life in Non-Muscle-Invasive Bladder Cancer Survivors: A Systematic Review. Cancer Nurs. 2019;42: E21-E33.
- 24. Bhattacharya A, Tang L, Li Y, et al. Inhibition of Bladder Cancer Development by Allyl Isothiocyanate. Carcinogenesis. 2009.
- 25. Sultana T, Savage GP, McNeil DL, Porter NG, Martin RJ, Deo B. Effects of fertilisation on the allyl isothiocyanate profile of above-ground tissues of New Zealand-grown wasabi. J. Sci. Food Agric. 2002;82: 1477-1482.
- 26. Parsons JK, Pierce JP, Natarajan L, et al. A randomized pilot trial of dietary modification for the chemoprevention of noninvasive bladder cancer: the dietary intervention in bladder cancer study. Cancer Prev Res (Phila). 2013;6: 971-978.
- 27. Kwan ML, Garren B, Nielsen ME, Tang L. Lifestyle and nutritional modifiable factors in the prevention and treatment of bladder cancer. Urol Oncol. 2019;37: 380-386.
- 28. Wang Z, Pratt R, Kwan ML, et al. Effects of cooking methods on total isothiocyanate yield from cruciferous vegetables. Under review. 2019.
- 29. Tang L, Paonessa JD, Zhang Y, Ambrosone CB, McCann SE. Total isothiocyanate yield from raw cruciferous vegetables commonly consumed in the United States. J Funct Foods. 2013;5: 1996-2001.
- 30. Thomson CA, Ravia J. A systematic review of behavioral interventions to promote intake of fruit and vegetables. J Am Diet Assoc. 2011;111: 1523-1535.
- 31. Pomerleau J, Lock K, Knai C, McKee M. Interventions designed to increase adult fruit and vegetable intake can be effective: a systematic review of the literature. J Nutr. 2005;135: 2486-2495.
- 32. Ammerman AS, Lindquist CH, Lohr KN, Hersey J. The efficacy of behavioral interventions to modify dietary fat and fruit and vegetable intake: a review of the evidence. Prev Med. 2002;35: 25-41.
- 33. Appleton KM, Hemingway A, Saulais L, et al. Increasing vegetable intakes: rationale and systematic review of published interventions. Eur J Nutr. 2016;55: 869-896.
- 34. Hazavehei SM, Afshari M. The role of nutritional interventions in increasing fruit and vegetable intake in the elderlies: a systematic review. Aging Clin Exp Res. 2016;28: 583-598.
- 35. Lara J, Hobbs N, Moynihan PJ, et al. Effectiveness of dietary interventions among adults of retirement age: a systematic review and meta-analysis of randomized controlled trials. BMC Med. 2014;12: 60.
- 36. Ye L, Dinkova-Kostova AT, Wade KL, Zhang Y, Shapiro TA, Talalay P. Quantitative determination of dithiocarbamates in human plasma, serum, erythrocytes and urine: pharmacokinetics of broccoli sprout isothiocyanates in humans. Clin Chim Acta. 2002;316: 43-53.
- 37. Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012;50: 217-226.
- 38. Yeary KH, Cornell CE, Prewitt E, et al. The WORD (Wholeness, Oneness, Righteousness, Deliverance): design of a randomized controlled trial testing the effectiveness of an evidence-based weight loss and maintenance intervention translated for a faith-based, rural, African American population using a community-based participatory approach. Contemp Clin Trials. 2015;40: 63-73.
- 39. Registry NC. <a href="https://www.health.ny.gov/statistics/cancer/registry/">https://www.health.ny.gov/statistics/cancer/registry/</a>. 2012-2016.

10/31/2022 

- 40. Health NYSDo. Behavioral Risk Factor Surveillance System (BRFSS) Health Indicators by County and Region. https://www.health.ny.gov/statistics/brfss/expanded/, 2016.
- 41. Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999;89: 1322-1327.
- 42. Barerra Jr. M, Castro FG. A Heuristic Framework for the Cultural Adaptaion of Interventions. Clinical Psychology and Practice. 2006;13: 311-316.
- 43. Evans SD, Sheffer CE, Bickel WK, et al. The Process of Adapting the Evidence-Based Treatment for Tobacco Dependence for Smokers of Lower Socioeconomic Status. J Addict Res Ther. 2015;6.
- 44. Wolf RL, Lepore SJ, Vandergrift JL, Basch CE, Yaroch AL. Tailored telephone education to promote awareness and adoption of fruit and vegetable recommendations among urban and mostly immigrant black men: a randomized controlled trial. Prev Med. 2009;48: 32-38.
- 45. Djuric Z, Ellsworth JS, Ren J, Sen A, Ruffin MTt. A randomized feasibility trial of brief telephone counseling to increase fruit and vegetable intakes. Prev Med. 2010;50: 265-271.
- 46. Lara J, Evans EH, O'Brien N, et al. Association of behaviour change techniques with effectiveness of dietary interventions among adults of retirement age: a systematic review and meta-analysis of randomised controlled trials. BMC Med. 2014;12: 177.
- 47. Cobiac LJ, Vos T, Veerman JL. Cost-effectiveness of interventions to promote fruit and vegetable consumption. PLoS One. 2010;5: e14148.
- 48. Gell NM, Rosenberg DE, Demiris G, LaCroix AZ, Patel KV. Patterns of technology use among older adults with and without disabilities. Gerontologist. 2015;55: 412-421.
- 49. Harris PA, Taylor R, Minor BL, et al. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019;95: 103208.
- 50. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009;42: 377-381.
- 51. Zhang Y, Cho CG, Posner GH, Talalay P. Spectroscopic quantitation of organic isothiocyanates by cyclocondensation with vicinal dithiols. Anal Biochem. 1992;205: 100-107.
- 52. Thomson CA, Newton TR, Graver EJ, et al. Cruciferous vegetable intake questionnaire improves cruciferous vegetable intake estimates. J Am Diet Assoc. 2007;107: 631-643.
- 53. Nutrition Data System for Research (NDSR)
- 54. Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017;12: 108.
- 55. Linnan L, Steckler A. Process Evaluation for Public Health Interventions and Research: An Overview. In: Steckler A, Linnan L, editors. Process Evaluation for Public Health Interventions and Research. San Francisco, CA: Jossey-Bass, 2002:1-23.
- 56. Estabrooks PA, Allen KC. Updating, employing, and adapting: a commentary on What does it mean to "employ" the RE-AIM model. Evaluation & the health professions. 2013;36: 67-72.
- 57. SAS Institute Incorporated S. SASv9.2 Documentation. Cary, NC.
- 58. Love MI, Huber W, Anders S. Moderated estimation of fold change and dispersion for RNA-seq data with DESeq2. Genome Biol. 2014;15: 550.
- 59. Luo W, Friedman MS, Shedden K, Hankenson KD, Woolf PJ. GAGE: generally applicable gene set enrichment for pathway analysis. BMC Bioinformatics. 2009;10: 161.
- 60. Signorelli C, Wakefield CE, Fardell JE, et al. Recruiting primary care physicians to qualitative research: Experiences and recommendations from a childhood cancer survivorship study. Pediatr Blood Cancer. 2018;65.
- 61. Moser A, Korstjens I. Series: Practical guidance to qualitative research. Part 3: Sampling, data collection and analysis. Eur J Gen Pract. 2018;24: 9-18.

10/31/2022 

- 62. Walker M, French SD, Doiron RC, et al. Bladder-sparing radiotherapy for muscle-invasive bladder cancer: A survey of providers to determine barriers and enablers. Radiother Oncol. 2017;125: 351-356.
- 63. Dong ST, Butow PN, Agar M, et al. Clinicians' Perspectives on Managing Symptom Clusters in Advanced Cancer: A Semistructured Interview Study. J Pain Symptom Manage. 2016;51: 706-717 e705.
- 64. Zhang, Y., et al., Spectroscopic quantitation of organic isothiocyanates by cyclocondensation with vicinal dithiols. Anal Biochem, 1992. 205(1): p. 100-7.
- 65. Tang, L. and Y. Zhang, Mitochondria are the primary target in isothiocyanate-induced apoptosis in human bladder cancer cells. Mol Cancer Ther, 2005. 4(8): p. 1250-9.

10/31/2022 

## **34. APPENDICES/ SUPPLEMENTS**

| Appendix A | Investigator Study Eligibility Verification Form Inclusion Criteria |
|---|---|
| Appendix B | Investigator Study Eligibility Verification Form Exclusion Criteria |
| Appendix C | Participant Urine Collection Instructions |
| Appendix D | Participant Urine Questionnaire |
| Appendix E | Participant Interview Phone Script |
| Appendix F | Participant Baseline Bladder Questionnaire |
| Appendix G | Participant Follow-up |
| Appendix H | New York State Cancer Registry Contact Materials and Procedures |
| Appendix I | Physician Interview Guide |
| Appendix J | Physician Research Study Information Sheet for Structured Interviews |
| Appendix K | Community Advisory Board (CAB) Research Study Information Sheet |
| Appendix L | Community Advisory Board (CAB) Interview Guide |
| Appendix M | Participant 24-hour Dietary Recall Instructions |
| Appendix N | Participant Food Amounts Booklet (FAB) |
| Appendix O | Participant Welcome Letter |
| Appendix P | Participant Health Magazines (Intervention and Control) |
| Appendix Q | Live Call Scripts (Intervention and Control) |
| Appendix R | Participant Track Books |
| Appendix S | Participant Thank You Letter |
| Appendix T | Recruitment Letter for Roswell Park Cancer Registry |
| Appendix U. | Invitation Letter for Physician Interview and Opt-In/Out Card |
| Appendix V | POW-R Sympathy Card |
| Appendix W | Participant Information Sheet for Cruciferous Arm Feedback Questions (For Participants that Completed the 6-Month Follow-up Assessment) |

10/31/2022 

## Appendix A INVESTIGATOR STUDY ELIGIBILITY VERIFICATION FORM INCLUSION CRITERIA

| | ı | | INCLUSION CRITERIA | |
|---|---|---|---|---|
| Yes | No | N/A | All answers must be "Yes" or "N/A" for participant enrollment. | Date |
| | | | Age 18 years old or older (no upper limit) | |
| | | | 2. English speaking | |
| | | | 3. Diagnosed with stage Tis, Ta, or T1 bladder cancer. | |
| | | | 4. Resides in the Western New York catchment area. | |
| | | | 5. Did not receive a partial or radical cystectomy. | |
| | | | 6. Does not have a prior cancer diagnosis within 12 months of their bladder cancer diagnosis. | |
| | | | 7. Does not have a subsequent more advanced bladder cancer diagnosis. | |
| | | | 8. For Roswell Park Cancer Registry only: Bladder cancer diagnosed 2016-2018, 2019-current. | |
| | | | 9. Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure. | |

10/31/2022 

## Appendix B INVESTIGATOR STUDY ELIGIBILITY VERIFICATION FORM EXCLUSION CRITERIA

| Partic | ipant | Name | e: | |
|---|---|---|---|---|
| Medio | al Rec | ord N | No: | |
| | | | alth: Power to Redefine your Health (Internal title: A Pragmatic Dietary<br>prove Bladder Cancer Survivorship) | Ý |
| | EXCLUSION CRITERIA | | | |
| Yes | No | N/A | All answers must be "No" or "N/A" for participant enrollment. | Date |
| | | | 1. Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. | |
| | | | 2. Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. | |
| | | | 3. Adults unable to consent. | |
| | | | 4. Adults unable to complete study measures in English. | |
| | | | 5. Individuals who are not yet adults (infants, children, teenagers). | |
| | | | 6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. | |
| | | | 7. Unwilling or unable to follow protocol requirements. | |
| | - | | s all entry criteria: | |
| | | | ature: Date: Investigator: | |
| TIHILE | u man | ne oi i | invesugator: | |

10/31/2022 

## **Appendix C** Participant Urine Collection Instructions

## **POW-R Health: Power to Redefine your Health**

# Program INSTRUCTIONS FOR URINE COLLECTION AND SHIPMENT

Thank you for being a part of this study. This sheet provides instructions for urine collection. The first morning urine (the time you typically get up and start daily routine) should be collected over three consecutive days (3 days in a row).

#### Materials in provided urine collection kit:

| 1. | Urine collection device (see below picture on the left) | 3 |
|----|--------------------------------------------------------------|---|
| 2. | Urine collection hat (see below picture on the right) | 3 |
| 3. | Biohazard bag with 2 absorbent pads | 1 |
| 4. | Ice packs* | 2 |
| 5. | Styrofoam shipping box with biohazard label and UN3373 label | 1 |
| 6. | FedEx shipping priority overnight label | 1 |
| 7. | Packing tape strips | 2 |
| 8. | Urine collection questionnaire | 1 |
| 9. | Plastic bag for urine collection guestionnaire | 1 |





\* **First**, <u>place the ice packs in your freezer</u> as soon as you get the kit so that they are frozen by the time the samples are ready to be shipped.

#### **URINE COLLECTION INSTRUCTIONS**

- 1. Collect the first void urine in the morning.
- 2. Urine can be collected in two ways:

<u>Using the urine collection device</u>: take out the sponge with holder from the container, directly urinate onto the sponge, and then insert sponge back into the container.

#### OR

<u>Using the urine collection hat</u>: place the urine collection hat on the toilet and urinate into it, then submerge the sponge into the urine, and insert the sponge

10/31/2022 

back into the container. Throw away the urine collection hat into a trash receptacle; do not ship the urine collection hat.

- 3. Write the date and time of the collection using a pen directly onto the label on the urine collection device.
- 4. Store the urine sample in its collection device, including both the sponge and container, in your refrigerator. The urine is absorbed into the sponge so it should not leak from the device.
- 5. Repeat the first morning urine collection for two more days in a row (Steps 1-4), storing the samples in the refrigerator until ready for shipment.

#### SCHEDULING A FEDEX PICKUP

After collecting the urine samples for three consecutive days, the samples can be shipped to Roswell Park Cancer Institute in Buffalo, NY for processing.

- \*\* NOTE: FedEx pickups should be scheduled for Monday through Thursday only, to ensure prompt delivery to the POW-R Health staff at Roswell Park Cancer Institute. Keep the urine samples and collection devices in the refrigerator until the scheduled shipping day. \*\*
  - 6. Call FedEx (1-800-GO-FEDEX; 1-800-463-3339) to schedule a pickup to ship the box to Roswell Park Cancer Institute. Do <u>not</u> take the package to a FedEx retail store for shipment or drop in a FedEx drop box.
    - a.) Once you have placed the call to FedEx, say "Schedule a Pickup"
    - b.) After the automated system has registered your request, dial 0, followed by the # sign to be directly transferred to a FedEx representative
    - c.) Let the representative know your samples will be delivered via **FedEx Express service** (priority overnight shipping)
    - d.) Provide the address from where you would like your samples to be retrieved

NOTE: If the FedEx representative asks for the account number, let them know you do not have it. The FedEx charge for your package has been pre-paid, and as long as the provided FedEx shipping priority overnight label is on the outside of your package, it will be picked up.

If you would prefer a FedEx pickup be scheduled on your behalf, please call the POW-R Health Study hotline at 1-716-845-8319.

#### PREPARING THE PACKAGE FOR SHIPMENT

7. Place all three urine samples and collection devices, including the containers and sponges, in the biohazard bag with absorbent pads. Seal the biohazard bag completely.

10/31/2022 

- 8. Remove the styrofoam lid of the shipping box, and place one pre-frozen ice pack on the bottom of the styrofoam shipping box.
- 9. Place the biohazard bag with the urine samples and collection devices on top of the ice pack in the shipping box.
- 10. Place the second pre-frozen ice pack on top of the biohazard bag, and replace the styrofoam lid on the shipping box.
- 11. Complete the urine collection questionnaire. Place the questionnaire in the provided plastic baggie and put it into the shipping box on top of the closed styrofoam container.
- 12. Seal the shipping box with the provided packing tape strips. As a reminder, the urine collection hats should be thrown away and not shipped back to us.
- 13. Remove the adhesive on the provided FedEx shipping priority overnight label and place the label on the top of the sealed shipping box.

| SHIPPING CHECKLIST |
|---|
| The following items should be included in your shipping box: |
| <ul> <li>□ 3 urine samples and collection devices in biohazard bag</li> <li>□ 2 frozen ice packs</li> <li>□ Urine collection questionnaire</li> <li>□ FedEx label on outside of shipping box</li> </ul> |

If you have any questions about collection or shipping, please contact:

Li Tang, Ph.D.
Roswell Park Comprehensive Cancer Center
Basic Science Building 708
Elm and Carlton Streets
Buffalo, NY 14263

Tel: 716-845-8247

10/31/2022 
**Urine Sample** 

☐ No

### Appendix D Participant Urine Questionnaire

## POW-R Health: Power to Redefine your Health Program Urine Collection Questionnaire

**Time of Collection** 

Please complete the following table with the date and time of collection for each urine sample:

**Date of Collection** 

| Sample #1 | | /<br>Month Day | | : | _ AM / PM<br>Circle one |
|---|---|---|---|---|---|
| Sample #2 | | /<br>Month Day | /<br>Year | : | _ AM / PM<br>Circle one |
| Sample #3 | | /<br>Month Day | /<br>Year | : | _ AM / PM<br>Circle one |
| the <u>day</u> | owing questi<br><u>before</u> your<br><u>before</u> your first | first urine | collection | on | |
| 1. Eat Broc | coli? | | | | |
| $\square$ Yes $\rightarrow$ Cooked | Please specify t | the type: 🗌 F | Raw □ Ligh | itly Cooked 🔲 T | horoughly |

10/31/2022 

Roswell Park Protocol No.: I 661820

2. Eat Broccoli Sprouts?

☐ Yes → Please specify the type: ☐ Raw ☐ Lightly Cooked ☐ Thoroughly Cooked
☐ No

3. Eat Cabbage?

☐ Yes → Please specify the type: ☐ Raw ☐ Lightly Cooked ☐ Thoroughly Cooked
☐ No

Continue to Next Page

10/31/2022 

Roswell Park Protocol No.: I 661820 4. Eat Carrots?  $\square$  Yes  $\rightarrow$ Please specify the type: Raw Lightly Cooked Thoroughly Cooked ☐ No 5. Eat Cauliflower?  $\square$  Yes  $\rightarrow$ Please specify the type: Raw Lightly Cooked Thoroughly Cooked □ No 6. Eat Brussels Sprouts? Please specify the type: Raw Lightly Cooked Thoroughly ☐ Yes → Cooked ☐ No 7. Eat Corn? Please specify the type: Raw Lightly Cooked Thoroughly  $\square$  Yes  $\rightarrow$ Cooked ☐ No 8. Eat Kale, Collard Greens, Mustard Greens, or Turnip Greens? Please specify the type: Raw Lightly Cooked Thoroughly  $\square$  Yes  $\rightarrow$ Cooked ☐ No 9. Eat Peas?

10/31/2022 

 $\square$  Yes  $\rightarrow$  Cooked

☐ No

Please specify the type: Raw Lightly Cooked Thoroughly

| 10. Eat Bok | Choy or Chinese cabbage? |
|---|---|
| $\square$ Yes $\rightarrow$ Cooked | Please specify the type: Raw Lightly Cooked Thoroughly |
| ☐ No | |
| 11. Eat Gard | den or Water Cress? |
| $\square$ Yes $\rightarrow$ Cooked | Please specify the type: Raw Lightly Cooked Thoroughly |
| □No | |
| 12. Eat Rad | ish or Turnip? |
| $\square$ Yes $\rightarrow$ Cooked | Please specify the type: Raw Lightly Cooked Thoroughly |
| □No | |
| 13. Eat Cele | ery? |
| $\square$ Yes $\rightarrow$ Cooked | Please specify the type: Raw Lightly Cooked Thoroughly |
| □No | |
| 14. Eat Sauc | erkraut? |
| ☐ Yes | |
| □No | |
| Continue to N | Next Page |

10/31/2022 

| Roswell Park Protocol No.: 1 661820 |
|---|
| 15. Eat Horseradish, Mustard, or Wasabi? |
| ☐ Yes<br>☐ No |
| 16. Take any antibiotic prescription medications (e.g., Cipro®, Septra®, penicillins, or other)? |
| ☐ Yes |
| □ No |
| 17. Smoke cigarettes? ☐ Yes → Please specify the total number of cigarettes: ☐ No |
| 18. Consume any alcoholic drink? |
| $\square$ Yes $\rightarrow$ Please specify the total number of drinks: |
| □ No |
| Date this questionnaire was completed _ / / Month Day Year |

Thank you very much for your time!

10/31/2022 

#### **Appendix E** Participant Interview Phone Script

# POW-R Health: Power to Redefine your Health Program PHONE SCREENING Paper Copy

| Today's Date | Time | |
|---|---|---|
| Leave the following message on the Cancer Institute) | A/M of potential participants (d | lo not say Roswell Park |
| Hi, this message is for POW-R Health: Power to Redefine younterest in our study. I would like to you. Please call me back between the reach me, please leave a message included to call. Thank you and I hope to speak | take a few minutes to explain the<br>e hours of 8:30am and 5 pm at _<br>luding your name, telephone nur | o on your call expressing<br>e study in more detail to<br>If you cannot |
| Speaking to participants: | | |
| "This is calling follow-up on your call expressing into Program being conducted here at Ross study in more detail to you. Is this a | swell Park. I would like to take a | titute. I'm calling to<br>yer to Redefine your Health<br>a few minutes to explain the |
| If NO: When would be the best day a | and time to call you back? | |
| If YES, or if first contact with resp | ondent: | |
| "We are conducting a study here at R reduce their risk of bladder cancer co specifically interested in testing whet who had bladder cancer. | ming back in those who had blac | dder cancer. We are |
| Your participation will last a total of | 6 months (about 24 weeks) and i | includes the following: |

We will ask you to complete two assessments. One before the study begins, and one after

the study ends. Each assessment will consist of:

- o A 45-60-minute survey over the phone
- O Telling us what you've eaten over the past 24-hours. This is called a dietary recall. This will be done on 3 randomly selected days. Each time it will take about 15-20 minutes over the phone.
- o Sending us urine samples through the mail.
- Being part of a 6-month program to improve your diet. The program will consist of:

10/31/2022 

- o Receiving educational materials about a healthy diet
- One 20-minute phone call with a Roswell staff member to talk to you about a healthy diet
- o 11 interactive voice response automated phone calls, where you will receive a phone call from a machine that will ask you how many vegetables you ate during a certain time period.

To thank you for your time and participation, you will be given a \$40 gift card to Tops Markets for completing the phone survey and sending the urine sample; and a \$20 gift card from Tops Markets for completing each dietary recall. So, for each assessment you will have the opportunity to receive a total of \$100 in gift cards to Tops Markets. Across both assessments you will have the opportunity to receive a total of \$200 in gift cards to Tops Markets.

Are you still interested in being a part of the study?

May we get your verbal consent to complete the baseline

**If NO:** Thank you for your time.

### **Demographics**

| New Applicant Introduc | tion Form | | | |
|---|---|---|---|---|
| only be shared wit<br>about our program<br>program that focu<br>recruiting adults v<br>information to det | th our rese<br>n. POW-R<br>uses on eati<br>who live in<br>termine yo | arch team. I v<br>Health: Powe<br>Ing more vege<br>Western New<br>ur eligibility t | vould like to ser to Redefine tables to impr<br>York. During | versation is confidential and will hare some information with you your Health is a healthy eating ove health. We are currently g this call I will gather in the program and whether the ake up to 15 minutes. Is that ok? |
| (circle one) Yes | S | No | | |
| If YES, continue. | | | | |
| If NO, read this so<br>me to call you back | | | | vould be a good day and time for |
| Let's begin with yo | ur name a | nd address. | | |
| 1. First: | | Middle: | | Last: |
| 2. Are you male or | female? | □Male | □Female | |

10/31/2022 

Roswell Park Protocol No.: I 661820 3. Are you Hispanic or Latino/a or Spanish in origin? □ Yes Are you (check all that apply): Mexican, Mexican American, Chicano/a Puerto Rican Cuban Another Hispanic, Latino/a, or Spanish origin □ No 4. Which one or more of the following would you say is your race? (Check all that apply) □ White ☐ Black or African American ☐ American Indian or Alaska Native ☐ Asian Indian ☐ Native Hawaiian □ Chinese ☐ Filipino ☐ Japanese ☐ Korean □ Vietnamese ☐ Other Asian ☐ Other Pacific Islander 5. What is your address? Street: City: Zip Code: 6. I would like to get your phone numbers:

| Daytime Phone: () | (circle one) l | home | work | cell |
|-----------------------------------|----------------|------|------|------|
| Evening Phone: () | (circle one) 1 | home | work | cell |
| Other: | (circle one) l | home | work | cell |
| 6a. Do you have an email address? | | | | |

7. What is your date of birth?:

| Month: | Day: | Year: |
|--------|------|-------|
| Note: | | |

If individual will turn 18 BEFORE the current round of recruitment closes, age ineligibility applies and this script is read:

10/31/2022 

| 1 P 1 T 1 100 |
|---|
| Applicant Turning 18 Soon |
| I'm sorry, you are not eligible to participate in the program. The program is |
| made for those aged 18 and older. |
| Would you like to continue with the questionnaire? Yes No |
| If answer is YES, continue to Question 8. |
| If answer is NO, thank applicant for his/her interest in the program and End Interview. |
| IF THE INDIVIDUAL PASSES THESE SET OF QUESTIONS CONTINUE TO THE NEXT SECTION. |
| Cancer |
| 8. Have you been diagnosed with stage Tis, Ta, or T1 bladder cancer? These are early stages of bladder cancer where the cancer lesion stays in the superficial layer of the bladder wall and does not invade the muscle layer. Sometimes they are called superficial bladder cancer or non-muscle invasive bladder cancer. |
| If YES, continue to Question 9. |
| If DON'T KNOW, continue to Question 9. |
| If NO, read this script: |
| I'm sorry,, you are not eligible to participate in the program. The program is designed for people who have been diagnosed with stage Tis, Ta, or T1 bladder cancer. Thank you for your interest, but we will not be able to enroll you. |
| 9. Have you received a partial or radical cystectomy? A cystectomy is surgery where a part or the entire bladder is removed. |
| If NO, continue to Question 10. |
| If YES, read this script: |
| I'm sorry,, you are not eligible to participate in the program. The program is designed for people who have NOT received a partial or radical cystectomy. Thank you for your interest, but we will not be able to enroll you. |

10. Have you had been diagnosed with another cancer (other than bladder cancer) during the past 12 months?

10/31/2022 

Roswell Park Protocol No.: I 661820 If NO, continue to Question 11. If YES, read this script: I'm sorry, , you are not eligible to participate in the program. The program is designed for people who have NOT been diagnosed with another cancer in the past 12 months of your being diagnosed with bladder cancer. Thank you for your interest, but we will not be able to enroll you. 11. Have you had chemotherapy or radiotherapy within the last 2 months? If NO, continue to Question 12. If YES, read this script: I'm sorry, , you are not eligible to participate in the program. The program would not be safe for those who have had chemotherapy or radiotherapy within the last 2 months. Thank you for your interest, but we will not be able to enroll you. Medications/Health 12. Have you been told by a doctor that you have any of the following health conditions? (circle one) a. Ongoing or active infection; b. Crohn's disease; c. Inflammatory Bowel Disease; d. Other (specify: symptomatic heart failure, unstable angina pectoris, cardiac arrhythmia) e. Psychiatric or social situations that would affect your participation No – Skip to the Consent Section Yes – Go to question 12a 12a. Please tell me more about your limitations? **12b. Record eligibility based on health condition** (circle one): Ineligible Questionable- refer to PI

10/31/2022 

Acceptable to continue

| If debilitating or such that the individual would have a hard time completing the program |
|---|
| then ineligibility applies and this script should be read: |

| I'm sorry, | you are not eligible to participate in the program. Thank you for |
|---|---|
| your interest, but | we will not be able to enroll you. |

#### If questionable and referring to PI, then this script should be read:

\_\_\_\_\_, based on the information you have given me, I can't tell for sure if you are eligible for the program. I need to talk with the Program Coordinator about whether you are eligible or not. Someone from our team will call you to see if you are eligible. If you are eligible, the remaining screening questions will be asked at that time.

The interview is STOPPED and the individual will be called back.

### **Consent**

Congratulations, Mr./ Ms Applicant. You are eligible to participate in POW-R Health: Power to Redefine your Health Program. Are you still interested in being a part of study?

If Yes, continue to the consent section.

If No, read this script:

| For below: Ok Mr./Ms | , Thank you for your interest in the Program. We |
|-----------------------|--------------------------------------------------|
| appreciate your time. | |

I would like to now go over the consent form for the study with you. (go over consent form).

I will mail you a copy for you to keep.

Before the program begins, you will need to complete the first assessment. Our team will call you to collect general information about your health. Our team will also call you on three different days to ask what you've eaten in the last 24 hours. So in total, you will receive 4 separate phone calls from our team to collect this information. We will also mail you a urine sample collecting kit for you to mail back to us. After we collect this information, you will receive your gifts cards for the first assessment. The POW-R Health: Power to Redefine your Health program materials will also be sent to you in the mail and one of our interventionists will call you.

If you would like to complete the first assessment now, can we get your verbal consent before we proceed? [Ask participant to indicate a Yes or No] Do you have any questions?

[If participant chooses to do the survey at another time, we will review the script at that time] Welcome to POW-R Health! Someone will be in touch with you soon.

10/31/2022 

#### Appendix F Participant Baseline Bladder Questionnaire

| Hi, my name is | . I'm calling because you kindly agreed to participate in the POW-R Health: Power |
|---|---|
| to Redefine your Health Pro | gram. If you recall, part of being in the study is completing a survey—once before |
| the study starts, and a final t | ime after the study ends. The survey information will be used to see if our dietary |
| intervention worked to impr | ove your health. This phone survey will take about 45-60 minutes to complete. Do |
| you have time to take the sur | evey now? |

**If no:** What would be a good day and time for me to call you? (please use Telephone Disposition Sheet)

**If yes:** Thank you! Please remember that everything you say here will be confidential. Your information won't be identified by name (proceed to questions below).

Let's start off with some information about you.

#### **DEMOGRAPHICS**

- 1. What is your marital status?
  - 1 Married
  - 2 Living as married
  - 3 Divorced
  - 4 Widowed
  - 5 Separated
  - 6 Single, never been married
- 2. What is the highest grade or level of schooling you completed?
  - 1 Less than 8 years
  - 2 8-11 years
  - 3 12 years or completed high school
  - 4 Post high school training other than college (vocational or technical)
  - 5 Some college
  - 6 College graduate
  - 7 Postgraduate
- 3. Thinking about members of your family living in this household, what is your combined annual income, meaning the total pre-tax income from all sources earned in the past year?
  - 1 \$0-\$9,000
  - 2 \$10,000-\$14,999
  - 3 \$15,000-\$19,999
  - 4 \$20,000-\$34,999
  - 5 \$35,000-\$49,999
  - 6 \$50,000-\$74,999
  - 7 \$75,000-\$99,999
  - 8 \$100,000-199,999
  - 9 \$200,000 or more

10/31/2022 

| 4. Wha | t is your occupational status? |
|---|---|
| | 1 Employed |
| | 2 Unemployed |
| | 3 Homemaker |
| | 4 Retired |
| | 5 Disabled |
| | 6 Other (Specify) |
| 5. How | many people currently live in your home (include yourself)? |
| | ou have any kind of health care coverage, including health insurance, prepaid plans such as Os or government plans such as Medicare, or Indian Health Service? 1 Yes (if yes, go to 6a) |
| | 2 No |
| 6a. V | What is the primary source of your health care coverage? |
| | A plan purchased through an employer or union (including plans purchased through another person's employer) |
| | . A plan that you or another family member buys on your own |
| 3 | . Medicaid (primarily for people over age 65) or other state program |
| 4 | . Medicare |
| 5 | . TRICARE (formerly CHAMPUS), VA, or Military |
| 6 | . Alaska Native, Indian Health Service, Tribal Health Service |
| 7 | . Some other source |
| 7. We would database. | l like to confirm your current address. Do you still live at? Read address from |
| ¹ ☐ Yes<br>□ ☐ No (ple | ease specify current address): |
| (Name of s | treet, city, state, zip) update if necessary |
| <b>BLADDER</b> | CANCER DIAGNOSIS |
| The next set | of questions is about your bladder cancer diagnosis. |
| | l like to confirm the date of your bladder cancer diagnosis. According to our records, you agnosed on Is that correct? |
| 1 Yes | |
| $0 \square \text{No} \rightarrow$ | 8a. What was the date? |
| 8 Don't K | |
| 9 Refused | <b>=</b> |
| | / = |

10/31/2022 

| 9. Did your doctor uresection. | ise a scope to remove the bladder tumor? This procedure is called a transurethral |
|---|---|
| $1 \square Yes \rightarrow$ | 9a. What was the date? |
| 0 No | 8 Don't Know |
| 8 Don't Know 9 Refused | 9 Refused |
| 10. Have you receiv | ed any additional treatment for bladder cancer since your diagnosis? |
| 1 Yes | |
| 0 No | |
| 8 Don't Know 9 Refused | |
| If No, Don't Know o | or Refused, go to Question 14. |
| 11. Did you receive | chemotherapy (e.g., mitomycin C, thiotepa, doxorubicin)? |
| Yes No Don't Know Refused | |
| 12. Did you receive | immunotherapy (e.g., bacillus Calmette-Guerin [BCG], interferon)? |
| Yes No Don't Know Refused | |
| 13. Did you receive | any other treatment? |
| 1 | 13a. Specify: |

10/31/2022 

### **CURRENT LIFESYLE**

The next section is about your current lifestyle. Again, this information is completely confidential.

| 14. What is your present height witho | ut shoes | <b>5?</b> | | | | | |
|---|---|---|---|---|---|---|---|
| _ <b>ft.</b> <b>inches</b><br>8 Don't Know<br>9 Refused | | | | | | | |
| 15. How much do you currently weigh | 1? | | | | | | |
| pounds | | | | | | | |
| 8 Don't Know 9 Refused | | | | | | | |
| | Excell<br>ent | Very<br>Good | Good | Fair | Poor | Don't<br>Know | Refuse<br>d |
| 16. In general, would you say your health is: | 5 | 4 | 3 | 2 | 1 | 8 | 9 |
| 17. In general, would you say your quality of life is: | 5 | 4 | 3 | 2 | 1 | 8 | 9 |
| 18. What is the primary source of drin | king wa | iter at y | our cur | rent resi | dence? | | |
| Private Well Community Supply (tap water, water) Bottled Water Other (specify): Don't Know Refused | r filtered | at home | e) | | | | |
| 19. Over the past 30 days, how many g | glasses o | f water ] | per day | do you | usually ( | drink? | |
| Less than 1 glass 1—2 glasses 3—3-4 glasses 4—5 or more glasses 8—Don't Know 9—Refused | | | | | | | |

10/31/2022 

| day? |
|---|
| More frequently than once an hour Once an hour Once every 2 hours Once every 3-5 hours Only once or twice a day Don't Know Refused |
| 21. Are you currently following any special diet? |
| 1 ☐ Yes 0 ☐ No 8 ☐ Don't Know 9 ☐ Refused |
| If No, Don't Know or Refused, go to Question 23. |
| 22. What type of special diet (check all that apply): |
| Vegetarian (with fish) Vegetarian (no fish) Vegan (no meat, chicken, fish, dairy, or eggs) Macrobiotic Paleo Gluten-free Low Carb Other (specify) Don't Know Refused |
| 23 Do you currently smoke? |
| 1 ☐ Yes, every day 2 ☐ Yes, some days → 23a. On how many of the past 30 days did you smoke a cigarette? ☐ Days 8 ☐ Don't Know |
| 9 Refused |

20. Over the past 30 days, how often did you typically feel the need to empty your bladder during the

10/31/2022 

| Roswell Park Protocol No.: I 661820 |
|---|
| <b>24.</b> On average, how many cigarettes do/did you smoke each day? (Note to interviewer: 1 pack=20 cigarettes) |
| _ Cigarettes per day |
| 8 Don't Know 9 Refused |
| 25. Over the last 30 days, how many days per week did you exercise for 20 minutes or more? |
| ☐ None ☐ 1-2 days ☐ 3-4 days ☐ 5 or more days |
| <b>26.</b> Compared to other people your age, how would you rate the level of your usual physical activity? (I currently ill, think about your activity during the past 30 days before your illness). |
| <ul> <li>☐ Much more active</li> <li>☐ More active</li> <li>☐ About the same</li> <li>☐ Less active</li> <li>☐ Much less active</li> </ul> |
| <u>DIETARY INTAKE</u> |
| These next questions are about the fruits and vegetables you ate or drank during the <u>past 30 days</u> . Please think about all forms of fruits and vegetables including cooked or raw, fresh, frozen or canned. Please think about all meals, snacks, and food consumed at home and away from home. |
| 27. During the past month, how many times per week did you drink 100% PURE fruit juices? Do no include fruit-flavored drinks with added sugar or fruit juice you made at home and added sugar to. Only include 100% juice. |
| times per week |
| 28. During the past month, not counting juice, how many times per week did you eat fruit? Count fresh, frozen, or canned fruit. |
| times per week |
| 29. During the past month, how many times per week did you eat cooked or canned beans, such as refried, baked, black, garbanzo beans, beans in soup, soybeans, edamame, tofu or lentils. Do NO include long green beans. |
| times per week |

10/31/2022 

| 30. | During the past month, how many times per week did you eat dark green vegetables for example broccoli or dark leafy greens including romaine, chard, collard greens or spinach? |
|---|---|
| | times per week |
| 31. | During the past month, how many times per week did you eat orange-colored vegetables such as sweet potatoes, pumpkin, winter squash, or carrots? (write number) |
| 32. | Not counting the vegetables mentioned, about how many times per week did you eat OTHER vegetables? Examples of other vegetables include tomatoes, tomato juice or V-8 juice, corn, eggplant, peas, lettuce, cabbage, and white potatoes that are not fried such as baked or mashed potatoes. (write number) |
| | <u>times per week</u> |

These next questions are about other vegetables you ate during the **past 30 days**. Please think about all meals, snacks, and food consumed at home and away from home.

(Go through table. Frame questions as, "How often did you eat raw arugula? Never, a few times per year, once per month, 2-3 times per month, once a week, twice per week, 3-4 times per week, 5-6 times per week, or every day." If they answer never, go to the next vegetable. If they ate any amount, ask, "About how much raw arugula did you eat each time? The medium serving size is one cup of the vegetable, about the size of a baseball. Lightly cooked generally includes stir fry, sauté, microwave, short-term, e.g. less than 10 minutes, steam or bake, and thoroughly cooked includes stew, biol, or long-term, e.g. more than 10 minutes, steam or bake.)

10/31/2022 

| Vegetables | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Never | A Few<br>Times<br>Per<br>Year | Once per month | 2-3<br>Times<br>per<br>month | Once<br>per<br>week | Twice<br>per<br>week | 3-4<br>Times<br>per<br>week | 5-6<br>Times<br>per<br>week | Every day | w mich tin |
| Arugula | raw | | | | | | | | | | |
| | lightly cooked<br>(e.g. stir fry) | | | | | | | | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | | | |
| Broccoli | raw | | | | | | | | | | |
| | lightly cooked<br>(e.g. stir fry) | | | | | | | | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | | | |
| Broccoli sprout | raw | | | | | | | | | | |
| | lightly cooked<br>(e.g. stir fry) | | | | | | | | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | | | |
| Broccolini | raw | | | | | | | | | | |
| | lightly cooked (e.g. stir fry) | | | П | | П | | | | П | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | | | |
| Corn | raw | | | | | | | | | | |
| | lightly cooked (e.g. stir fry) | | | | | | | | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | | | |

10/31/2022 

| Green cabbage | 11000001110100 |
|---|---|
| Green cabbage | raw (e.g.<br>coleslaw) |
| | lightly cooked<br>(e.g. stir fry)<br>thoroughly |
| | cooked (e.g. stew) |
| Red/<br>Purple cabbage | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Sauerkraut | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Carrots | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Cauliflower | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly cooked (e.g. |
| | stew) |

10/31/2022

| | 1: 1.1 1 1 | I | 1 |
|----------------|-------------------------------------|---|---|
| | lightly cooked (e.g. stir fry) | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | |
| Kale | raw | | |
| | lightly cooked (e.g. stir fry) | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | |
| Kohlrabi | raw | | |
| | lightly cooked (e.g. stir fry) | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | |
| Collard greens | lightly cooked<br>(e.g. stir fry) | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | |
| Peas | raw | | |
| | lightly cooked<br>(e.g. stir fry) | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | |
| Mustard greens | raw | | |
| | lightly cooked (e.g. stir fry) | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | |
| Turnip | lightly cooked (e.g. stir fry) | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | |

10/31/2022

| | Protocor No., 1 00 | 1020 | 1 | 1 | Г | Τ | 1 | 1 | , |
|---|---|---|---|---|---|---|---|---|---|
| Turnip greens | lightly cooked<br>(e.g. stir fry) | | | | | | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | |
| Bok/ Pak choy | raw | | | | | | | | |
| | lightly cooked (e.g. stir fry) | | | | | | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | |
| Chinese cabbage/<br>Napa | raw | | | | | | | | |
| | lightly cooked (e.g. stir fry) | | | | | | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | |
| Daikon root | raw | | | | | | | | |
| | lightly cooked (e.g. stir fry) | | | | | | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | |
| Celery | raw | | | | | | | | |
| | lightly cooked (e.g. stir fry) | | | | | | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | |
| Garden cress | raw | | | | | | | | |
| | lightly cooked (e.g. stir fry) | | | | | | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | |
| Water cress | raw | | | | | | | | |

10/31/2022

| | lightly cooked (e.g. stir fry) |
|-----------|-------------------------------------|
| | thoroughly<br>cooked (e.g.<br>stew) |
| Radicchio | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Radishes | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly cooked (e.g. |

We're going to finish the survey by asking some final questions about sauces and condiments you ate during the **past 30 days**. Please think about all meals, snacks, and food consumed at home and away from home.

(Go through table. Frame questions as, "How often did you eat mayonnaise? Never, a few times per year, once per month, 2-3 times per month, once a week, twice per week, 3-4 times per week, 5-6 times per week, or every day." If they answer never, go to the next food. If they ate any amount, ask, "About how much mayonnaise did you eat each time? The size of your thumb from knuckle to tip or less? About two thumbs worth? Or more than 2 thumbs worth?"

For *horseradish*, if they consume any amount, ask, "about how much horseradish did you eat each time? Smaller than an egg, about the size of egg, or more than the size of an egg?)

10/31/2022 

| SAUCES AND CONDIMENTS | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | A Few | | | Once | | 3-4 | | Ever | | | ng<br>: | |
| | Never | Times<br>Per<br>Year | per<br>month | Times per month | 1 | week | | s per | | Medium<br>Serving | | | |
| | | | | | | | | | | | S | M | L |
| Mayonnaise and mayonnaise-type spreads | | | | | | | | | | 2 Tbsp. | | | |
| Horseradish | | | | | | | | | | ¹⁄₄ cup | | | |
| Mustard | | | | | | | | | | 2 Tbsp. | | | |
| Wasabi | | | | | | | | | | 2 Tbsp. | | | |

### **Belief into Action Scale**

Circle a <u>single</u> number for each question below:

### 1. Please circle the highest priority in your life now? (most valued, prized)

- 1. My health and independence
- 2. My family
- 3. My friendships
- 4. Job, career or business
- 5. My education
- 6. Financial security
- 7. Relationship with God
- 8. Ability to travel & see the world
- 9. Listening to music and partying
- 10. Freedom to live as I choose

#### 2. How often do you attend religious services? (circle a number below)

| Never | Rarely | Couple<br>times/yr | Every few mos | About once/mo | Several<br>times/mo | About every wk | Every<br>week | More than once/wk | Daily |
|---|---|---|---|---|---|---|---|---|---|
| 1 | | | | | | | | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |

10/31/2022 

# 3. Other than religious services, how often do you get together with others for religious reasons (prayer, religious discussions, volunteer work, etc.)?

| Nev | ver | Rarely | Couple<br>times/yr | Every few mos | About once/mo | Several<br>times/mo | About<br>every wk | Every<br>week | More than once/wk | Daily |
|---|---|---|---|---|---|---|---|---|---|---|
| | 1 | | 2 | <u>'</u> | | | _ | 0 | - | 10 |
| | 1 | 2 | 3 | 4 | 5 | 6 | 1 | 8 | 9 | 10 |

#### 4. To what extent (on a 1 to 10 scale) have you decided to place your life under God's direction?



### 5. What percentage of your gross annual income do you give to your religious institution or to other religious causes each year?



# 6. On average, how much time each $\underline{day}$ (in 24 hrs) do you spend listening to religious music or radio, or watching religious TV?

| 0 (never) | 1–5 min | 6–10 min | 11–20 min | 21–30 min | 31–60<br>min | More than 1 hr, less than 2 hr | More than 2 hr, less than 3 hr | 3–4 hrs | 5 hrs or<br>more |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |

# 7. On average, how much time each <u>day</u> do you spend reading religious scriptures, books, or other religious literature?

| 0 (n | ever) | 1-5 | min 6 | -10 min | 11–20 m | in 21–30 mi | n 31–60<br>min | More than 1 hr,<br>less than 2 hr | More than 2 hr,<br>less than 3 hr | 3–4 hrs | 5 hrs or<br>more |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | <br>1 | ·<br>2 | | 3 | <br>4 | 5 | 6 | <br>7 | 8 | 9 | 10 |

#### 8. On average, how much time each day do you spend in private prayer or meditation?

| 0 (never) | 1–5 min | 6–10 min | 11–20 min | 21–30 min | 31–60<br>min | More than 1 hr, less than 2 hr | More than 2 hr, less than 3 hr | 3–4 hrs | 5 hrs or<br>more |
|---|---|---|---|---|---|---|---|---|---|
| 1 | <br>2 | 3 | 4 | <br>5 | <br>6 | <br>7 | <br>8 | <br>9 | <br>10 |

10/31/2022 

## 9. On average, how much time each <u>day</u> do you spend as a volunteer in your religious community or to help others for religious reasons?

| 0 (never) | 1–5 min | 6–10 min | 11–20 min | 21–30 min | 31–60<br>min | More than 1 hr,<br>less than 2 hr | More than 2 hr, less than 3 hr | 3–4 hrs | 5 hrs or<br>more |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |

### 10. To what extent (on a 1 to 10 scale) have you decided to conform your life to the teachings of your religious faith?



You have finished the survey! Thank you so much for your time. Do you have any questions?

Again, welcome to POW-R Health Program!

10/31/2022 

### **Appendix G Participant Follow-up**

### Appendix G1. Participant 6-month Follow-up Questionnaire

| Health: Power to Recompleting a survey-<br>survey information w | define your Health Program. If you recall, part of being in the study is—once before the study starts, and a final time after the study ends. The vill be used to see if our dietary intervention worked to improve your health. ill take about 45-60 minutes to complete. Do you have time to take the |
|---|---|
| If no: What would be Sheet) | e a good day and time for me to call you? (please use Telephone Disposition |
| - | lease remember that everything you say here will be confidential. Your eidentified by name (proceed to questions below). |
| BLADDER CANCE | ER FOLLOW-UP |
| S | rey with questions about your bladder cancer status. These questions riod since we last talked with you, which is approximately the past 6 |
| 1. In the last 6 bladder cand | months, have you had a clinical assessment, or cystoscopy, for your cer? |
| | → Skip to Question 2 (cystectomy) |
| 8 Don't Know | → Skip to Question 2 (cystectomy) |
| 9 Refused | → Skip to Question 2 (cystectomy) |
| 1a. What was the da | ate of your last assessment? |
| 2. In the last 6 | months, have you had a cystectomy (surgery to remove the bladder)? |
| o No | → Skip to Question 3 (recurrence) |
| 8 Don't Know | → Skip to Question 3 (recurrence) |
| 9 Refused | → Skip to Question 3 (recurrence) |
| 2a. What was the da | ate of the cystectomy? |

10/31/2022 

| your d | last 6 months, have you had a recurrence of your bladder cancer (i.e., did octor say that the original cancer came back or that you had a new |
|---|---|
| | mass/tumor)? |
| 1 Yes | Strip to Opportion 10 (other concern) |
| | → Skip to Question 10 (other cancer) |
| 8 Don't Kno | 1 , |
| 9 Refused | → Skip to Question 10 (other cancer) |
| 3.1 How many | y recurrences have you had? (Number) |
| [Note to Interv | viewer: If more than 1 recurrence, record the date of the most recent (last) |
| 3.1a. What wa | as the date of your recurrence? |
| 4. Did yo 1 Yes 0 No 8 Don't Kno 9 Refused | ur recurrent bladder cancer progress to muscle-invasive disease? |
| proced | ur doctor use a scope to remove the recurrent bladder tumor? This lure is called a transurethral resection. becify Date in 5a |
| 8 Don't Kno<br>9 Refused | ow |
| 5a. What was | s the date of transurethral resection (TURBT)? |
| - | u receive chemotherapy (e.g., mitomycin C, thiotepa, doxorubicin) for your er cancer recurrence/progression? |
| Yes No Don't Kno | ow. |
| 9 Refused | |
| • | u receive immunotherapy (e.g., bacillus Calmette-Guerin [BCG], interferon)<br>ir bladder cancer recurrence/progression? |
| 1 Yes | |
| 0 No | |
| 8 Don't Kno | 0W |
| 9 Refused | |

10/31/2022 

Roswell Park Protocol No.: I 661820 8. Did you receive radiation therapy for your bladder cancer recurrence/progression? 1 Yes  $_{0}$  No 8 Don't Know 9 Refused 9. Did you receive any other treatment for your bladder cancer recurrence/progression? Yes  $\rightarrow$  Specify treatment in 9a  $_{0}$  No 8 Don't Know 9 Refused 9a. Specify other treatment received: 10. In the last 6 months, have you been diagnosed with any other types of cancer since your original bladder cancer diagnosis? Yes 0 | No → Skip to Question 11 → Skip to Question 11 8 Don't Know → Skip to Question 11 9 Refused 10a. When did you receive this diagnosis? 10b. What was your diagnosis? 11. Overall, how would you rate your satisfaction with your current understanding of bladder cancer and its treatment? Excellent Very Good Good Fair 5 Poor Don't Know 9 Refused Now that we've gone over your bladder cancer status, we're now going to talk about your current lifestyle. **CURRENT LIFESYLE** 12. What is your present height without shoes? | ft. | | | inches Don't Know 9 Refused

10/31/2022 

| 13. How much do you currently weig | gh? | | | | | | |
|---|---|---|---|---|---|---|---|
| <b>pounds</b><br>8 Don't Know<br>9 Refused | | | | | | | |
| | Excell<br>ent | Very<br>Good | Good | Fair | Poor | Don't<br>Know | Refus<br>d |
| 14. In general, would you say your health is: | 5 | 4 | 3 | 2 | 1 | 8 | 9 |
| 15. In general, would you say your quality of life is: | 5 | 4 | 3 | 2 | 1 | 8 | 9 |
| 16. What is the primary source of dri | nking wa | ater at y | our cur | rent res | idence? | | |
| Private Well Community Supply (tap water or w Bottled Water Cother (specify): Don't Know Refused | ater filter | red at ho | me) | | | | |
| 17. Over the past 30 days, how many | glasses o | f water | per day | do you | usually | drink? | |
| Less than 1 glass 1—2 glasses 3—3-4 glasses 4—5 or more glasses 8—Don't Know 9—Refused | | | | | | | |
| 18. Over the past 30 days, how often during the day? | did you t | ypically | feel the | need to | empty | your bla | dder |
| More frequently than once an hour Once an hour Once every 2 hours Once every 3-5 hours Only once or twice a day Don't Know Refused | | | | | | | |

10/31/2022 

| any other special diet? | of the POW-R Health Program, are you currently following |
|---|---|
| Yes No Don't Know Refused | |
| If No, Don't Know or Refuse | ed, go to Question 21. |
| 20. What type of special die | t (check all that apply): |
| Vegetarian (with fish) Vegetarian (no fish) Vegan (no meat, chicker Macrobiotic Paleo Gluten-free Low Carb Other (specify) Don't Know Refused | n, fish, dairy, or eggs) |
| 21. Do you currently smoke | e? |
| <ul><li>Yes, every day</li><li>Yes, some days →</li></ul> | 21a. On how many of the past 30 days did you smoke a cigarette? |
| | Days Don't Know Refused |
| <b>22.</b> On average, how many pack=20 cigarettes) | cigarettes do/did you smoke each day? (Note to interviewer: 1 |
| _ Cigarettes per day | |
| 8 Don't Know 9 Refused | |
| 23. Over the last 30 days, h more? | ow many days per week did you exercise for 20 minutes or |
| 0 ☐ None<br>1 ☐ 1-2 days | |

10/31/2022 

10/31/2022 

#### **DIETARY INTAKE**

These next questions are about the fruits and vegetables you ate or drank during the <u>past 30</u> <u>days</u>. Please think about all forms of fruits and vegetables including cooked or raw, fresh, frozen or canned. Please think about all meals, snacks, and food consumed at home and away from home.

| juice | es? Do not include fruit-flavored drinks with added sugar or fruit juice you e at home and added sugar to. Only include 100% juice. |
|---|---|
| | times per week |
| | ing the past month, not counting juice, how many times per week did you eat? Count fresh, frozen, or canned fruit. |
| | times per week |
| bear | ing the past month, how many times per week did you eat cooked or canned as, such as refried, baked, black, garbanzo beans, beans in soup, soybeans, name, tofu or lentils. Do NOT include long green beans. |
| | times per week |
| for $\epsilon$ | ing the past month, how many times per week did you eat dark green vegetables example broccoli or dark leafy greens including romaine, chard, collard greens binach? <u>times per week</u> |
| | <del></del> |
| | ing the past month, how many times per week did you eat orange-colored tables such as sweet potatoes, pumpkin, winter squash, or carrots? (write ber) |
| OTI<br>V-8 | counting the vegetables mentioned, about how many times per week did you eat IER vegetables? Examples of other vegetables include tomatoes, tomato juice or juice, corn, eggplant, peas, lettuce, cabbage, and white potatoes that are not I such as baked or mashed potatoes. (write number) |
| | times per week |

10/31/2022 

These next questions are about other vegetables you ate during the **past 30 days**. Please think about all meals, snacks, and food consumed at home and away from home.

(Go through table. Frame questions as, "How often did you eat raw arugula? Never, a few times per year, once per month, 2-3 times per month, once a week, twice per week, 3-4 times per week, 5-6 times per week, or every day." If they answer never, go to the next vegetable. If they ate any amount, ask, "About how much raw arugula did you eat each time? The medium serving size is one cup of the vegetable, about the size of a baseball. Lightly cooked generally includes stir fry, sauté, microwave, short-term, e.g. less than 10 minutes, steam or bake, and thoroughly cooked includes stew, biol, or long-term, e.g. more than 10 minutes, steam or bake.)

10/31/2022 

| Vegetables | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Never | A<br>Few<br>Times<br>Per<br>Year | Once<br>per<br>month | 2-3<br>Times<br>per<br>month | week | Twice<br>per<br>week | 3-4<br>Times<br>per<br>week | 5-6<br>Times<br>per<br>week | Every day | n<br><u>e</u><br><u>ti</u> | How<br>nuch<br>each<br>me' | ո<br><u>ւ</u> |
| Arugula | raw | | | | | | | | | | | | |
| | lightly cooked<br>(e.g. stir fry)<br>thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | | | | | |
| Broccoli | raw | | | | | | | | | | | | |
| | lightly cooked<br>(e.g. stir fry)<br>thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | | | | | |
| Broccoli sprout | raw | | | | | | | | | | | | |
| | lightly cooked<br>(e.g. stir fry)<br>thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | | | | | |
| Broccolini | raw | | | | | | | | | | | | |
| | lightly cooked<br>(e.g. stir fry)<br>thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | | | | | |
| Corn | raw | | | | | | | | | | | | |
| | lightly cooked<br>(e.g. stir fry)<br>thoroughly<br>cooked (e.g.<br>stew) | | | | | | | | | | | | |

10/31/2022 

| Green cabbage | raw (e.g.<br>coleslaw) |
|---|---|
| | lightly cooked<br>(e.g. stir fry)<br>thoroughly |
| | cooked (e.g. stew) |
| Red/<br>Purple cabbage | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Sauerkraut | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Carrots | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Cauliflower | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Brussels sprouts | raw |

10/31/2022 
| | lightly cooked |
|----------------|-------------------------------------|
| | (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Kale | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Kohlrabi | raw |
| | lightly cooked<br>(e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Collard greens | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Peas | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Mustard greens | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Turnip | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |

10/31/2022 

| Turnip greens | lightly cooked | | | |
|---|---|---|---|---|
| | (e.g. stir fry) | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | |
| Bok/ Pak choy | raw | | | |
| | lightly cooked (e.g. stir fry) | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | |
| Chinese cabbage/ Napa | raw | | | |
| | lightly cooked (e.g. stir fry) | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | |
| Daikon root | raw | | | |
| | lightly cooked (e.g. stir fry) | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | |
| Celery | raw | | | |
| | lightly cooked (e.g. stir fry) | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | |
| Garden cress | raw | | | |
| | lightly cooked (e.g. stir fry) | | | |
| | thoroughly<br>cooked (e.g.<br>stew) | | | |
| Water cress | raw | | | |
| | 1 | l | j | l |

10/31/2022 

| | lightly cooked (e.g. stir fry) |
|-----------|-------------------------------------|
| | thoroughly<br>cooked (e.g.<br>stew) |
| Radicchio | lightly cooked (e.g. stir fry) |
| | thoroughly<br>cooked (e.g.<br>stew) |
| Radishes | raw |
| | lightly cooked (e.g. stir fry) |
| | thoroughly cooked (e.g. stew) |

I am now going to ask some questions about sauces and condiments you ate during the **past 30** days. Please think about all meals, snacks, and food consumed at home and away from home.

(Go through table. Frame questions as, "How often did you eat mayonnaise? Never, a few times per year, once per month, 2-3 times per month, once a week, twice per week, 3-4 times per week, 5-6 times per week, or every day." If they answer never, go to the next food. If they ate any amount, ask, "About how much mayonnaise did you eat each time? The size of your thumb from knuckle to tip or less? About two thumbs worth? Or more than 2 thumbs worth?"

For *horseradish*, if they consume any amount, ask, "about how much horseradish did you eat each time? Smaller than an egg, about the size of egg, or more than the size of an egg?)

10/31/2022 

| SAUCES AND CONDIMEN | ITS | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | A Few | | | Once | | 3-4 | | Ever | | | ervii<br>Size | |
| | Never | Times<br>Per<br>Year | per<br>month | Times per month | 1 | week | | s per | | Medium<br>Serving | | | |
| | | | | | | | | | | | S | M | L |
| Mayonnaise and mayonnaise-type spreads | | | | | | | | | | 2 Tbsp. | | | |
| Horseradish | | | | | | | | | | ¹⁄₄ cup | | | |
| Mustard | | | | | | | | | | 2 Tbsp. | | | |
| Wasabi | | | | | | | | | | 2 Tbsp. | | | |

#### **Belief into Action Scale**

Circle a <u>single</u> number for each question below:

#### 1. Please circle the highest priority in your life now? (most valued, prized)

- 1. My health and independence
- 2. My family
- 3. My friendships
- 4. Job, career or business
- 5. My education
- 6. Financial security
- 7. Relationship with God
- 8. Ability to travel & see the world
- 9. Listening to music and partying
- 10. Freedom to live as I choose

#### 2. How often do you attend religious services? (circle a number below)

| Never | Rarely | Couple times/yr | Every few mos | About once/mo | Several times/mo | About<br>every wk | Every<br>week | More than once/wk | Daily |
|---|---|---|---|---|---|---|---|---|---|
| l | | | | | | | | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | |
| 9 | 10 | | | | | | | | |

10/31/2022 

### 3. Other than religious services, how often do you get together with others for religious reasons

(prayer, religious discussions, volunteer work, etc.)?

| Never | Rarely | Couple times/yr | Every few mos | About once/mo | Several times/mo | About<br>every wk | Every<br>week | More than once/wk | Daily |
|---|---|---|---|---|---|---|---|---|---|
| <br>1 | <br>2 | 3 | 4 | 5 | 6 | 7 | 8 | | |
| 9 | 10 | 3 | т | 3 | O | , | O | | |

### 4. To what extent (on a 1 to 10 scale) have you decided to place your life under God's direction?

| | at all<br>ly haven't tho | ought about it) | | То а | ı moderate deg | ree | | Completely, totally |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | . | - |
| i | | | • | • | ' | • | | |
| ] | 1 2 | $\frac{1}{2}$ | 3 | 4 5 | 5 6 | · | 7 | 8 |
| Ģ | ) 1( | ) | | | | | | |

# 5. What percentage of your gross annual income do you give to your religious institution or to other religious causes each year?

| 0% | Less<br>than 1% | 1%—2% | 3%-4% | 5%-6% | 7%-8% | 9%-10% | 11%—12% | 13%—14% | 15% or more |
|---|---|---|---|---|---|---|---|---|---|
| 1 | | 2 | 4 | ~ | ( | 7 | 0 | | |
| 1 | 2 | 3 | 4 | 5 | 6 | / | 8 | | |
| 9 | 10 | | | | | | | | |

## 6. On average, how much time each $\underline{day}$ (in 24 hrs) do you spend listening to religious music or radio, or watching religious TV?

| 0 (never) | 1–5 min | 6–10 min | 11–20 min | 21–30 min | 31–60<br>min | More than 1 hr,<br>less than 2 hr | More than 2 hr,<br>less than 3 hr | 3–4 hrs | 5 hrs or<br>more |
|---|---|---|---|---|---|---|---|---|---|
| | · <br>· | | | | | | | | |
| 1 | $\stackrel{1}{2}$ | 3 | 4 | 5 | 6 | 7 | 8 | | |
| 9 | 10 | | | | | | | | |

10/31/2022 

### 7. On average, how much time each $\underline{day}$ do you spend reading religious scriptures, books, or other religious literature?

| 0 (never) | 1–5 min | 6–10 min | 11–20 min | 21–30 min | 31–60<br>min | More than 1 hr,<br>less than 2 hr | More than 2 hr, less than 3 hr | 3–4 hrs | 5 hrs or<br>more |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | |
| 9 | 10 | | | | | | | | |

#### 8. On average, how much time each day do you spend in private prayer or meditation?

| 0 (never) | 1–5 min | 6–10 min | 11–20 min | 21–30 min | 31–60<br>min | More than 1 hr,<br>less than 2 hr | More than 2 hr,<br>less than 3 hr | 3–4 hrs | 5 hrs or<br>more |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | |
| 9 | 10 | | | | | | | | |

### 9. On average, how much time each <u>day</u> do you spend as a volunteer in your religious community or to help others for religious reasons?

| 0 (never) | 1–5 min | 6–10 min | 11–20 min | 21–30 min | 31–60<br>min | More than 1 hr,<br>less than 2 hr | More than 2 hr, less than 3 hr | 3–4 hrs | 5 hrs or<br>more |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | |
| 9 | 10 | | | | | | | | |

## 10. To what extent (on a 1 to 10 scale) have you decided to conform your life to the teachings of your religious faith?

| Not at all (really haven't thought about it) | | | t) | To a moderate degree | | | | Completely, totally |
|---|---|---|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
| | 9 | 10 | | | | | | |

We're going to finish the survey by asking your opinion about the dietary program you got.

I'm going to read some statements about the dietary program you got. Please let me know whether you completely disagree with the statement, disagree with the statement, neither agree nor disagree with the statement, agree with the statement, or completely agree with the statement.

10/31/2022 

| | Completely disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Completely agree |
|---|---|---|---|---|---|
| 1. The diet program I received met my approval. | ① | 2 | 3 | 4 | (5) |
| 2. The diet program I received was appealing to me. | ① | 2 | 3 | 4 | (5) |
| 3. I liked the diet program I received. | ① | 2 | 3 | 4 | (5) |
| 4. I welcomed the diet program I received. | ① | 2 | 3 | 4 | (5) |

| | Completely disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Completely agree |
|---|---|---|---|---|---|
| 1. The diet program I received fit into my lifestyle. | 1 | 2 | 3 | 4 | (\$) |
| 2. The diet program I received was suitable to my lifestyle. | ① | 2 | 3 | 4 | (5) |
| 3. The diet program I received was applicable to my lifestyle. | ① | 2 | 3 | 4 | (5) |
| 4. The diet program I received was a good match with my lifestyle. | ① | 2 | 3 | 4 | (5) |

#### Feasibility of Intervention Measure (FIM)

| | Completely disagree | Disagree | Neither agree nor disagree | Agree | Completely agree |
|---|---|---|---|---|---|
| 1. The diet program I received was implementable in my life. | 1 | 2 | 3 | 4 | (5) |
| 2. The diet program I received was possible to do in my life. | ① | 2 | 3 | 4 | (\$) |
| 3. The diet program I received was doable. | 0 | 2 | 3 | 4 | (5) |
| 4. The diet program I received was easy to use. | 1 | 2 | 3 | 4 | (5) |

If you are a part of Group A, there are a few feedback questions we would like to ask you at this time, is this okay?

If you are a part of Group B, you have finished the survey! Thank you so much for your time. Do you have any questions? Again, thank you for your participation in POW-R Health!

10/31/2022 

#### Appendix G2. POW-R Participant Additional Questions to Follow-Up Questionnaire

These questions will be given to those in the cruciferous arm only.

Thank you so much for being a part of the POW-R study. The program you went through consisted of a mailed magazine, a phone call with one of our Roswell staff, and then 11 automated phone calls. We would like to ask the feedback questions regarding the study at this time.

#### 1. What did you think about the magazine?

- a. What did you like about it?
- b. What would you change?

#### 2. What did you think about the phone call with the Roswell staff person?

- a. What did you like about it?
- b. What would you change?

#### 3. What did you think of the 11 automated calls?

- a. What did you like about it?
- b. What would you change?

#### 4. What do you think having this program as a phone app?

You have finished the survey! Thank you so much for your time. Do you have any questions? Again, thank you for your participation in POW-R Health!

10/31/2022 

#### Appendix H New York State Cancer Registry Contact Materials and Procedures

# POW-R Health: Power to Redefine your Health Program NYS Cancer Registry Patient Contact and Data Handling Procedures

The procedures described in this document are standard procedures the New York State Cancer Registry (NYSCR) follows for patient contact studies.

#### I. Approval Process

- 1. Roswell Park Cancer Institute IRB approval
- 2. NY State Health Department Administrative approval

# II. NYSCR Patient Consenting Process (i.e., physician notification and patient consent to release name, contact information, and diagnostic information to Roswell Park Cancer Institute)

Using ICD-O-3 codes provided in the study protocol, the NYSCR will conduct a search of its database to identify eligible patients who were diagnosed with stage Tis, Ta, or T1 bladder cancer in 2018 or later, who resided in one of eight counties of interest at diagnosis (Niagara, Orleans, Genesee, Erie, Wyoming, Chautauqua, Cattaraugus, and Allegany), who are 18 years of age or older, who did not receive a cystectomy, who did not have a prior cancer diagnosis within 12 months of their bladder cancer diagnosis, who did not have a subsequent more advanced bladder cancer diagnosis, and who have not died or opted out of research studies. This search will be repeated if needed until the recruitment goal is reached. The NYSCR will contact reporting facilities to obtain the patients' physician information, if missing in the database.

The NYSCR will send a letter to the physician of record for selected cases notifying him/her that the patient was identified for the study, requesting that the NYSCR be notified if the patient is deceased, too ill or otherwise unable or ineligible to participate in the study, and requesting information about the case's primary care physician if different from the contacted physician. The physician will have three weeks to respond.

If no contraindication is received from the physician or if the physician has not responded within three weeks, the NYSCR will send an informational packet to the patient. The packet will contain: 1) a letter explaining the study and requesting permission to release their name, contact information, and diagnostic information to the study's principal investigator at Roswell Park Cancer Institute; 2) a participant information sheet; and 3) a release of information consent form. If the NYSCR has not received any response after two weeks a reminder packet of information will be sent. Again, if no response is forthcoming after two more weeks, five telephone calls will be attempted by the NYSCR (three during regular business hours, and two during non-business hours) to describe the study and receive a response (either consent or refusal). If the patient consents verbally, NYSCR staff will fill out the consent form and document that the consent was obtained via phone. If the Registry is unable to contact the patient via telephone, and no written response has been received, no other contact will be attempted, and the patient will be considered a refusal

10/31/2022 

Upon receipt of the consent form, the patient's name, contact information, and diagnostic information will be provided by the NYSCR to the study's principal investigator at Roswell Park Cancer Institute via Roswell's secure File Transfer Solution (sFTP). The NYSCR will receive a unique user name and password in separate emails to transfer the data via sFTP.

#### **III. Roswell Park Patient Contact Procedures**

Upon receipt of the patient information from the NYSCR, the Roswell Park research team will contact the patient by telephone. All members of the Roswell Park research team will have completed Collaborative Institutional Training Initiative (CITI training). If the patient is not reached during the first attempt, the research team will make additional attempts using the following algorithm: five additional attempts at varying dates and times, for a total of six attempts over three weeks. Each attempt will be documented in the call manager portion of the Electronic Data Capture system. After all phone attempts are exhausted, a traceable Hard to Reach Letter will be mailed to the patient's address listed in the patient profile. The patient will be asked to contact the Roswell Park research team if they are interested in learning more about the study.

Upon contact with the patient, the Roswell Park research team member will again explain the study, administer the screening interview, and obtain consent for the patient's participation. The Roswell Park research team will record the patient's real time responses in the corresponding Patient Phone Screening Interview Form in the Electronic Data Capture system. The patient will be mailed a consent form for them to keep. For respondents who do not wish to participate, the telephone contact will be terminated, and they will be ineligible for the study. Information on non-participants will be provided to the NYSCR, as well as any information for any individuals who indicate that they do not want to be contacted about any future research studies.

#### IV. Data Handling, Dissemination and Storage Procedures

After receipt of the patient information from the NYSCR, the data will be entered and stored in REDCap. REDCap is a secure application supported by Partners Research Computing, Enterprise Research Infrastructure & Services (ERIS). ERIS has all the necessary physical and operational securities in place to meet or exceed Federal and State security and privacy regulations for data transmission and storage using REDCap. The dataset containing patient contact information will be separated from the research dataset including survey data and urine sample tracking data. The data will only be accessed by key members of the Roswell Park research team who are in charging of contacting patients. All the data communications between NYSCR and Roswell Park will be transferred via Roswell's secure File Transfer Solution (sFTP). A unique username and password will be used for each data transfer and sent in separate emails.

10/31/2022 

#### Exhibit A

The following information will be provided to Roswell Park for each bladder cancer case identified for possible inclusion in the study:

- 1. Reporting source
- 2. Patient name
- 3. Patient address and telephone number
- 4. Physician name and contact information
- 5. Basic demographic information (race, ethnicity, date of birth, county of residence)
- 6. Primary site
- 7. Summary stage
- 8. Histology
- 9. Laterality
- 10. Date of diagnosis
- 11. Age at diagnosis
- 12. First course of treatment
- 13. Primary surgical procedure
- 14. Chemotherapy
- 15. Date of last contact

10/31/2022 

#### Materials used by the New York State Cancer Registry for the

POW-R Health: Power to Redefine your Health Program [Letter from NYS Cancer Registry to Physician]

Month, Day, Year

{Physician Name} {Physician Address} {Physician City, State Zip}

Dear Dr. "M.D.\_LAST NAME":

We are writing to inform you that the New York State Department of Health's Cancer Registry is collaborating with Roswell Park Comprehensive Cancer Center on a pilot study of a dietary intervention with a goal to reduce the risk of recurrence in individuals diagnosed with non-muscle invasive bladder cancer. Patients diagnosed with non-muscle invasive bladder cancer (including Tis, Ta, and T1 disease) who did not receive cystectomy and who live in the counties of Niagara, Orleans, Genesee, Erie, Wyoming, Chautauqua, Cattaraugus, and Allegany may be eligible for the study.

Our records show that one of your patients was recently diagnosed with bladder cancer and meets the study criteria. The patient's name and other identifying information reported to the Cancer Registry are on the enclosed form. We would like to contact your patient to assess their interest in participating in the study.

Patients will be sent an introductory letter describing the study and requesting their consent for their name, contact information, and some information about their diagnosis to be shared with Roswell Park Comprehensive Cancer Center. Patients who consent will be contacted by phone regarding participation in the study. Patient participation in the study includes participation in a 6-month phone-based dietary intervention that will consist of educational materials mailed to the patient's home, one 20-minute phone call with Roswell Park staff to go over the educational materials, and 11 automated telephone calls asking participants to report the number of vegetable servings they have consumed in the prior week, followed by tailored feedback based on the servings reported. Patients will also be asked to complete two assessments, one at the beginning of the study, and one at the end. These assessments will include a 45-60-minute phone survey, self-collection of a urine sample, and three 24-hour dietary recalls. All information that could identify the patient will be kept confidential. Names and other identifying information will not be used in any publication about the study.

If you do not object to our contacting your patient, you do not need to do anything further. However, there may be some reason why your patient cannot or should not be contacted about

10/31/2022 

participation in this study; therefore, we would like to hear from you within the next three weeks if you prefer that we do not contact your patient.

If you prefer that we do not contact your patient please complete the enclosed form and fax it to "Attn: bladder cancer study" at (518) 473-6789 or mail it back to us in the enclosed self-addressed, stamped envelope. If you have any questions about the study or the form, please contact Dr. Maggie Kuliszewski at the New York State Cancer Registry at (518) 474-2255. Thank you very much for your assistance.

Sincerely,

Maria J. Schymura, Ph.D. Director, New York State Cancer Registry

10/31/2022 

| New York State Cancer Registry<br>POW-R Health: Power to Redefine your Health Program | |
|---|---|
| Patient Information Sheet for Physician | |
| Name of Physician<br>Address<br>Address<br>Address<br>Telephone number | |
| If information below is incorrect please provide correct information. Patient Name | |
| Patient Address | |
| Telephone number | |
| Patient DOB Sex<br>Race | |
| Diagnosed with non-muscle invasive Tis, Ta, or T1 bladder cancer? Yes No If yes, date first diagnosed | |
| Any medical contraindications to patient contact for the study? Yes If yes, please explain | |
| Physician signature Date | |
| Please fax the completed form to "Attn: bladder cancer study" at (518) 4 form in the enclosed self-addressed, stamped envelope to: | 73-6789. Or mail the |
| POW-R Health: Power to Redefine your Health Program, New York Sta<br>NYS Department of Health, Suite 361, Riverview Center, 150 Broadway | |
| Thank you for your assistance. | |
| Date sent | |

10/31/2022 

| [Letter from NYS Cancer Registry to Patient | ] |
|---------------------------------------------|---|
| {Patient Name} | |
| {Patient Street Address} | |
| {Patient City, State, ZIP} | |
| Dear : | |

The New York State Department of Health's Cancer Registry is contacting patients who may be eligible for a research study. The study is being done in collaboration with researchers at Roswell Park Cancer Institute. The purpose of the study is to learn more about how diet may reduce the risk of recurrence in individuals with early-stage bladder cancer. Men and women who were recently diagnosed with early-stage bladder cancer and who live in the counties of Niagara, Orleans, Genesee, Erie, Wyoming, Chautauqua, Cattaraugus, and Allegany may be eligible for the study.

Under New York State Public Health Law, hospitals and doctors must report all cases of cancer that they find to the New York State Cancer Registry. This is how we learned about your diagnosis.

Please take the time to read the enclosed information about this study. We would like to send your name, contact information, and some information about your diagnosis to researchers at Roswell Park Cancer Institute, so that they can contact you to see if you are eligible for the study and interested in participating. However, we need your consent in order to release your name and contact information. Please fill out the enclosed consent form to let us know if we can share your information with Roswell Park Cancer Institute.

Please mail the completed consent form back to us in the enclosed self-addressed, stamped envelope. If we do not receive the form, someone from our office will call you to make sure you received this letter and to discuss the study with you.

If you have any questions about this study, please call Dr. Maggie Kuliszewski at the New York State Cancer Registry at (518) 474-2255.

If you have any questions about your rights as a participant in this study or think you have been harmed by the study, please contact Mr. Tony Watson, the Administrator of the Institutional Review Board at the New York State Department of Health at (518) 474-8539.

We greatly appreciate your help with this study.

Sincerely,

Dr. Maria Schymura, Director New York State Cancer Registry

10/31/2022 

**Enclosures** 

POW-R Health: Power to Redefine your Health Program New York State Department of Health Cancer Registry

**Participant Information Sheet** 

The New York State Department of Health's Cancer Registry and Roswell Park Cancer Institute are collaborating on a research study of individuals with bladder cancer in New York State. The purpose of the study is to better understand how diet may reduce the risk of recurrence in men and women diagnosed with early-stage bladder cancer.

Procedure: A researcher from Roswell Park Cancer Institute will contact you to see if you are eligible for the study and would like to participate. If you decide to participate, you will receive a 6-month dietary intervention that may improve your health. The intervention will include educational materials mailed to your home, a 20-minute phone call with Roswell Park staff to go over the educational materials, and 11 automated phone calls that will give you feedback on your diet based on how many vegetables you report eating during the past week. To see if our dietary intervention improves health, we will also ask you to complete two assessments, one at the beginning of the study, and one at the end of the study. The assessment will include a 45-60-minute survey, a self-collected urine sample, and three dietary recalls. Individuals who are eligible for and participate in the study will receive up to \$200 in gift cards at a local retail store as a token of appreciation for their participation.

Voluntary Participation: Taking part in this study is up to you. You may stop taking part at any time. You may refuse to answer any question. If you decide not to take part, you will not lose any benefits that you would normally receive.

Confidentiality: We will keep all of your answers and health information private, as required by law. If you decide to participate in the study, we will assign a code to you and use the code instead of your name. Any records that include your name and could link you to the coded information will be kept in electronic files accessible only to assigned study staff and will be password-protected on the computer. Access will be allowed only to the researchers involved in the study who have signed a confidentiality agreement. Your name and other identifying information will not appear in any reports of this study. Your address will not be used to send any additional promotional information whatsoever.

Benefits: You may or may not benefit from the study intervention. Information about your experience in the study may contribute to our understanding of factors that reduce the risk of recurrence of early-stage bladder cancer and may help other people in the future.

Risks: There are no known risks to being part of this study. Talking about your health and your bladder cancer diagnosis may cause you some stress. There is also the potential (but unlikely) loss of confidentiality regarding your responses to questions. We have many procedures in place to prevent this. Please see the above section on confidentiality.

10/31/2022 

Questions about the Study:

If you have any questions about this study, please call Dr. Maggie Kuliszewski at the New York State Cancer Registry at (518) 474-2255.

If you have any questions about your rights as a participant in this study or think you have been harmed by the study, please contact Mr. Tony Watson, the Administrator of the Institutional Review Board at the New York State Department of Health at (518) 474-8539.

10/31/2022 

#### [NYS CANCER REGISTRY PATIENT CONSENT FORM]

## INFORMED CONSENT FOR FURTHER CONTACT POW-R Health: Power to Redefine your Health Program

I understand that by checking the first statement and by signing this form below I am agreeing to allow the New York State Cancer Registry to release my name, contact information, and some information about my bladder cancer diagnosis to Roswell Park Cancer Institute.

| Please check one of the following statements. Please sign and return in the enclosed envelope. |
|---|
| 1. I consent to the release of my name, contact information, and some information about my bladder cancer diagnosis to Roswell Park Cancer Institute. I understand that a researcher from that organization will contact me to see if I am eligible for the study and would like to participate. |
| Name (please print) |
| Signature |
| Address |
| Telephone # |
| Date |
| 2. I do not consent to the release of my name, contact information, or information about my bladder cancer diagnosis to Roswell Park Cancer Institute. I do not want anyone from that organization to contact me. |
| (Name of patient pre-printed on the bottom – in case above is illegible) |

10/31/2022 

# STATEMENT TO BE READ REGARDING THE STUDY PURPOSE, PROCEDURES INVOLVED, RISKS AND BENEFITS INVOLVED, AND CONFIDENTIALITY NYS Cancer Registry Patient Contact — (if mailed response was not obtained)

| Hello | my name is | . May I please speak with | )7 |
|---------|-----------------|---------------------------|-----|
| riciio, | , illy maine is | Ividy I picuse speak with | , . |

I'm from the New York State Department of Health's Cancer Registry. We're collaborating with Roswell Park Cancer Institute on a research study of individuals with bladder cancer in New York State. The purpose of the study is to better understand how diet may reduce the risk of recurrence in men and women diagnosed with early-stage bladder cancer. Men and women who were recently diagnosed with early-stage bladder cancer and who live in the counties of Niagara, Orleans, Genesee, Erie, Wyoming, Chautauqua, Cattaraugus, and Allegany may be eligible for the study. Recently, we sent you a letter asking for your consent for us to share your name, contact information, and some information about your bladder cancer diagnosis with Roswell Park Cancer Institute. Did you receive the letter?

IF "YES", PROCEED WITH SCRIPT BELOW.

IF "NO", ASK IF THEY WOULD LIKE TO CONTINUE OR HAVE YOU SEND ANOTHER LETTER.

IF "ANOTHER LETTER", VERIFY ADDRESS.

IF "CONTINUE", PROCEED WITH SCRIPT BELOW.

As the letter explains, the purpose of the study is to better understand certain factors that may reduce the risk of recurrence in men and women diagnosed with early-stage bladder cancer. If you consent for us to share your name and contact information with Roswell Park Cancer Institute, a researcher will contact you to see if you are eligible for the study and would like to participate. If you decide to participate, you will receive a 6-month dietary intervention that may improve your health. The intervention will include educational materials mailed to your home, a 20-minute phone call with Roswell Park staff to go over the educational materials, and 11 automated phone calls that will give you feedback on your diet based on how many vegetables you report eating during the past week. To see if our dietary intervention improves health, we will also ask you to complete two assessments, one at the beginning of the study, and one at the end of the study. The assessment will include a 45-60-minute survey, a self-collected urine sample, and three dietary recalls.

Taking part in this study is up to you. You may stop taking part at any time. You may refuse to answer any question. If you decide not to take part, you will not lose any benefits that you would normally receive. Individuals who are eligible for and participate in the study will receive up to \$200 in gift cards at a local retail store as a token of appreciation for their participation.

All of your answers will be kept private as required by law. All records that include your name will be kept in locked file cabinets. All records on the computer will be password-protected. Access will be allowed only to the researchers involved in the study. Your name and other identifying information will not appear in any reports of this study.

10/31/2022 

You may or may not benefit from the study intervention. Information about your experience in the study may contribute to our understanding of factors that reduce the risk of recurrence of early-stage bladder cancer and may help other people in the future. There are no known risks from being a part of the study. Talking about your health and your bladder cancer diagnosis may cause you some stress. There is also the potential (but unlikely) loss of confidentiality regarding your responses to questions. We have many procedures in place to prevent this.

If you have any questions about this study, please call Dr. Maggie Kuliszewski at the New York State Cancer Registry at (518) 474-2255.

If you have any questions about your rights as a participant in this study or think you have been harmed by the study, please contact Mr. Tony Watson, the Administrator of the Institutional Review Board at the New York State Department of Health at (518) 474-8539.

Do you consent to the release of your information to Roswell Park Cancer Institute? If so, someone from that organization will contact you by phone.

CHECK THE APPROPRIATE RESPONSE BOX ON THE PATIENT CONSENT FORM. SIGN AND DATE THE FORM IN THE BLANK SPACE ABOVE THE PATIENT SIGNATURE LINE AND ADD "BY TELEPHONE" AFTER THE DATE.

10/31/2022 

#### **Appendix I** Physician Interview Guide

#### **Physician Semi-Structured Interview**

To be administered right after verbal consent.

Thank you for agreeing to be a part of this study.

Our dietary intervention consists of giving bladder cancer patients 3 things: 1) educational materials by mail, 2) One 20 minute phone call with a trained staff member to go over the educational materials, and 3) 11 automated phone calls that ask patients to report the servings of vegetables they ate in the previous week, with automated feedback based on the number of servings reported.

If our study shows that this intervention significantly reduces bladder cancer recurrence in bladder cancer patients:

- 1. To what extent would you welcome such an intervention? Probe: What would make you like this intervention more?
- 2. To what extent would you think the intervention would be a good match for your clinic? Probe: What would make this intervention fit better within your clinic?
- 3. To what extent do you think the intervention would be doable in your clinic? Probe: What would make this intervention easier for your clinic to use?

That concludes the interview. Thank you so much for your time.

10/31/2022 

#### Appendix J Physician Research Study Information Sheet for Structured Interviews

Please keep a copy of this form for your reference.

I am (fill in name/role), with the Division of Prevention & Population Sciences at Roswell Park Comprehensive Cancer Center. I am working with a team at Roswell Park to learn about the barriers and facilitators of intervention implementation within clinical practice. The goal is to gain feedback and develop the intervention for "real-world' implementation.

To accomplish this, we would like to conduct a semi-structured interview with a total of 20 physicians or health care providers within the area in Western New York. This study is funded by the National Cancer Institute.

I would like to tell you more about it before you decide whether or not to participate in this onetime interview study. Please stop me at any time if you have any questions. Your participation is completely voluntary; you do not have to participate.

During the interview, I will provide you with a brief overview of our dietary intervention for bladder cancer patients. I will then ask questions regarding facilitators and barriers of intervention adoption within clinical practice. I will ask your opinion on the needed implementation strategies to sustain the intervention, in addition to intervention modifications to maximize sustained clinic adoption. The interview should last approximately 15 minutes. I may ask your permission to electronically record the discussion so we can capture information accurately. If you object to electronically recording the conversation, please let me know now.

This information will be collected anonymously (without linking it to your name or identity, or identifying any patients; all data will be aggregated). We will not be using your name on any of the forms or any information that is gathered.

Your involvement in this study does not involve any physical risk to you. The possible risks include feeling uncomfortable answering questions, embarrassment, or someone identifying you as a participant in the project, although this would be rare. You will not receive any direct health benefit from participating in this study.

Participants that complete the interview will receive a \$100 gift card to a local retail store.

You do not have to take part in this one-time contact research study. If you decide to participate, you can stop your participation at any time. You may refuse to answer any questions and you may leave at any time.

Results of this study will yield important information on the feasibility of a dietary behavioral intervention to improve bladder cancer outcomes among bladder cancer patients. These results have the potential to improve the survivorship outcomes of a group at elevated risk of cancer recurrence, as well as for teaching, for research, for scientific publications and/or for presentations at scientific meetings. You will not be identified in any way. Your participation is completely anonymous because I am not collecting your name (or taking photographs of you).

10/31/2022 

If you have any questions, you are free to ask them now. If you have questions or concerns about the study at any time, you can call the Roswell Park Office of Research Subject Protection at (716) 845-3455. You may contact me at the telephone number I will provide in a few minutes. This study has been reviewed and approved by the Roswell Park Institutional Review Board.

#### **CONTACT INFORMATION:**

#### If you have any questions about this study, you may contact me:

Cassy Dauphin Roswell Park Comprehensive Cancer Center Elm & Carlton Streets Buffalo, NY 14263 716-845-8319

#### Or you may contact the Principal Investigator, who is the Director of this study:

Karen Yeary, PhD Roswell Park Comprehensive Cancer Center Elm & Carlton Streets Buffalo, NY 14263 716-845-1300 Ext 6231

Li Tang, PhD Roswell Park Comprehensive Cancer Center Elm & Carlton Streets Buffalo, NY 14263 716-845-8247

10/31/2022 

#### Appendix K Community Advisory Board (CAB) Research Study Information Sheet

Please keep a copy of this form for your reference.

I am (fill in name/role), with the Division of Cancer Prevention and Control at Roswell Park Comprehensive Cancer Center. I am working with a team at Roswell Park to adapt materials and methods from current evidence-based fruit and vegetable interventions in order to develop a dietary intervention for bladder cancer survivors. The goal is to gain feedback and develop the intervention for "real-world" implementation. This study is funded by the National Cancer Institute.

I would like to tell you more about it before you decide whether or not to participate. Please stop me at any time if you have any questions. Your participation is completely voluntary; you do not have to participate.

In this study, you will be asked to attend three meetings (in person or virtual) as a Community Advisory Board (CAB) member to help develop a dietary intervention that will be relevant for bladder cancer survivors. You will be asked to review intervention materials and messages and provide feedback for improvements. We will also ask you some demographic questions. Each meeting will last approximately 90 minutes. We may ask your permission to electronically record the discussion so we can capture information accurately. If you object to electronically recording the conversation, please let us know.

This information will be collected anonymously (without linking it to your name or identity or identifying any patients; all data will be aggregated). We will not be using your name on any of the forms or any information that is gathered.

Your involvement in this study does not involve any physical risk to you. The possible risks include feeling uncomfortable answering questions, embarrassment, or someone identifying you as a participant in the project, although this would be rare. You will not receive any direct health benefit from participating in this study.

CAB members will be asked to complete a structured 60 minute interview, will receive \$50 for interview, compensated \$100 per meeting attended, up to three meetings, and interviews will be conducted over the phone.

You do not have to take part in this one-time contact research study. If you decide to participate, you can stop your participation at any time. You may refuse to answer any questions and you may leave at any time

Results of this study will yield important information on the feasibility of a dietary behavioral intervention to improve bladder cancer outcomes among bladder cancer patients. These results have the potential to improve the survivorship outcomes of a group at elevated risk of cancer recurrence, as well as for teaching, for research, for scientific publications and/or for presentations at scientific meetings. You will not be identified in any way. Your participation is completely anonymous because I am not collecting your name (or taking photographs of you).

If you have questions or concerns about the study at any time, you can call the Roswell Park Office of Research Subject Protection at (716) 845-3455. You may contact me at the telephone number I will provide in a few minutes. This study has been reviewed and approved by the Roswell Park Institutional Review Board.

10/31/2022 

#### **CONTACT INFORMATION:**

#### If you have any questions about this study, you may contact me:

Nikia Clark Roswell Park Comprehensive Cancer Center Elm & Carlton Streets Buffalo, NY 14263 716-845-4888

#### Or you may contact the Principal Investigators, who are the Directors of this study:

Karen Yeary, PhD Roswell Park Comprehensive Cancer Center Elm & Carlton Streets Buffalo, NY 14263 716-845-1300 Ext 6231

Li Tang, PhD Roswell Park Comprehensive Cancer Center Elm & Carlton Streets Buffalo, NY 14263 716-845-8247

10/31/2022 

#### Appendix L Bladder Community Advisory Board (CAB) Interview Guide

Thank you for being willing to be a part of helping us make a healthy eating program for bladder cancer survivors to improve their health. We're going to start by asking some questions about you.

- 1. (Administer demographic survey, page 2)
- 2. When were you first diagnosed with bladder cancer?
  - o What type of treatment did you receive after your bladder cancer diagnosis?
  - O How long did the treatment last?
- 3. Have you had any recurrence since your initial bladder cancer diagnosis?
  - o If yes, when did it happen and what treatment did you receive?
- 4. What is the biggest concern you have regarding your bladder cancer diagnosis?
- 5. Since your bladder cancer diagnosis, did you change your eating habits?
  - o If yes, how did you change your eating habits?
- 6. Do you think what you eat can make a difference in terms of bladder cancer prevention or recurrence?
  - o If yes, how?
- 7. Recent research has shown that eating more cruciferous vegetables can reduce the chances of bladder cancer coming back in bladder cancer survivors. Cruciferous vegetables include broccoli, arugula, brussels sprouts, green or white cabbage, and turnips.
  - What do you think about this information? Is this helpful? Have you heard this before?
- 8. In your day-to-day life, what might make it easier for you to eat more cruciferous vegetables?
  - Probes: Help from your family, help from the healthcare system, help from friends, any particular information
- 9. Who does most of the shopping for food in your family?
  - o If self: What affects the kinds or amount of vegetables you buy?
  - o If not self: What role do you play in what they shop for?
- 10. Who does most of the planning or preparing of meals in your family?
  - o If not self: What role do you play in how meals are planned or prepared?
- 11. How do other people in your life impact the kinds and amounts of vegetables you eat?

10/31/2022 

#### **Demographic Survey**

| • | Are you | male or female? | |
|---|---|---|---|
| | 1 | Male | |
| | 2 | Female | |
| • | • | Hispanic or Latino/a or S | panish in origin? |
| | 1 | Yes | |
| | | Are you: | 1 Mexican, Mexican American, Chicano/a |
| | | (circle all that apply) | |
| | | | 3 Cuban |
| | • | N | 4 Another Hispanic, Latino/a, or Spanish origin |
| | 2 | No | |
| • | Which o | one or more of the followir | ng would you say is your race? (Circle all that |
| | apply) | | |
| | 1 | White | |
| | | Black or African American | |
| | | American Indian or Alaska | n Native |
| | | Asian | |
| | 5 | Other (please specify) | |
| • | How old | are you? | |
| | _ | years | |
| • | What is | your marital status? | |
| | | Married | |
| | 2 | Living as married | |
| | | Divorced | |
| | 4 | Widowed | |
| | 5 | Separated | |
| | 6 | Single, never been married | d |
| • | What is | the highest grade or level | of schooling you completed? |
| | | Less than 8 years | , I |
| | | 8-11 years | |
| | | 12 years or completed high | school |
| | | | ther than college (vocational or technical) |
| | | Some college | , |
| | | College graduate | |
| | | Postgraduate | |

10/31/2022 

• What is your occupational status?

1 Employed

- 2 Unemployed
- 3 Homemaker
- 4 Retired
- 5 Disabled
- 6 Other (Specify)
- How many people currently live in your home (include yourself)?
- In the past 12 months, have you received food stamps, also called SNAP, the Supplemental Nutrition Assistance Program on an EBT card?
  - 1 Yes
  - 2 No
  - 3 Don't know
- Do you have any kind of health care coverage, including health insurance, prepaid plans such as HMOs or government plans such as Medicare, or Indian Health Service?
  - 1 Yes (if yes, go to 11a)
  - 2 No

#### 11a. What is the primary source of your health care coverage?

- 35. A plan purchased through an employer or union (including plans purchased through another person's employer)
- 36. A plan that you or another family member buys on your own
- 37. Medicaid (primarily for people over age 65) or other state program
- 38. Medicare
- 39. TRICARE (formerly CHAMPUS), VA, or Military
- 40. Alaska Native, Indian Health Service, Tribal Health Service
- 41. Some other source

I'm going to read you several statements that people have made about their food situation. For these statements, please tell me whether the statement was often true, sometimes true, or never true for (you) in the last 12 months—that is, since last (name of current month). The first statement is:

- "The food that I bought just didn't last, and I didn't have money to get more." Was that often, sometimes, or never true for you in the last 12 months?
  - 1 Often true
  - 2 Sometimes true
  - 3 Never true
  - 4 DK or Refused
- "I couldn't afford to eat balanced meals." Was that often, sometimes, or never true for you in the last 12 months?

1 Often true

10/31/2022 

2 Sometimes true

3 Never true

4 DK or Refused

10/31/2022 

#### **Appendix M Participant 24-hour Dietary Recall Instructions**

#### 24-Hour Recalls

#### What's a 24-Hour Recall?



24-hour recalls are a way of figuring out what you usually eat and drink. We will get this

information through talking to you on the telephone, where we will ask you to remember what you ate and drank during the previous day.

The telephone recalls will occur on 3 separate days at the start of the study, and 3 separate days at the end of the study. The days will be selected at random so that weekdays (Monday through Thursday) and one weekend day (Friday through Sunday) is included. This will help us figure out your *average* diet.

#### **Scheduling the Calls**

A person from Roswell Park Cancer Institute, Buffalo, NY will be calling you to do the recalls. They will call you during the times you said would work best with your schedule when you signed up to be a part of the study. At this time, they will call and ask you for details of **everything** -- all foods and liquids (including water) -- that you ate or drank during the past 24 hours from midnight to midnight of the previous day.

The person will ask you the amount you actually ate or drank, not how much was put into the dish, cup, or bowl. Please use the "Food Amounts Booklet" that we sent you with this sheet. The following tips will also help you estimate how much you eat and drink.

#### **Measuring Tips**



Use measuring cups and spoons to help you tell the Roswell person the exact amount you ate or drank.

Instead of telling the Roswell person you had breakfast cereal, give more details like: 1 cup of wheat flakes with 1/2 cup of lowfat milk, and 1/2 of a large (8-inch) banana.

- Measure the volume of dishes, bowls, cups, and glasses that you use a lot. This will help you to figure out and report the correct volume of food/drink each time you use that container.
- For pieces of food that do not fit into a cup or spoon, describe the size using the "Food Amounts Booklet".

For example, 1 corn tortilla (6 inches across), and 1 cube of cheese (2" long x 1" wide x 1/2" high). You can use weight or dimensions for reporting meat, fish, poultry, cheese, pizza, and baked goods. Include thickness, length, and width of food using a ruler. Indicate if the weight was obtained before or after cooking.

**Be Specific.** When naming the food or drink that you ate/drank, give the Roswell person details. For example, if you ate meat, details such as the part eaten are important. If you ate chicken, tell the person whether it was from the thigh or breast, or if it was white or dark meat.

**Brand Names & Labels.** Brand names of prepared foods are very useful for the Roswell person, as are labels from the prepared foods you have eaten.

10/31/2022 

Mixed Foods. Be prepared to tell the Roswell person what is in a mixed food. For example, rather than just saying 1 cup of stew, do your best to give the amount of each major item in the stew, such as 1/4 cup stewed beef, 1/4 cup potato, 1/4 cup carrot, 1/4 cup gravy. If you made a dish at home, report the recipe used including all ingredients, and the number of servings from the recipe or what portion of the total you actually ate.

Preparation Method. It is also important for you to describe how the foo was cooked, such as baked, boiled, broiled, fried, breaded and fried. For example, one chicken drumstick (fried in shortening, no flour or batter).

Add-Ons. Remember to tell your Roswell person the little things added to foods like butter, margarine, mustard, jelly, sugar, gravy, or salad dressing.

**Nonfat Items.** Don't forget to report nonfat items. Just because they are nonfat does not mean they are not important to include.

Time & Place. The Roswell person will ask you to say about what time the food or drink was eaten or drank, and whether it was eaten at a meal or a snack. It is also very helpful if you can say where the food or drink was eaten/drank, for example at home, work, school, restaurant, store, etc. For example, at 2:00 PM, I ate a snack at home. The snack was 2 tablespoons of raisins and 8 whole-grain crackers (2-inch diameter).

also ask you what vitamin and/or mineral or herbal supplements you took during the prior day. It is important that you have these supplements handy, as the Roswell person will ask you for specific information about the supplement ingredients.

For those supplements with more than one ingredient, the Roswell person will ask you for the brand name, the manufacturer, and the manufacturer's contact information (address, phone number, and/or website).

We have information on the contents of many of these. However, we may need to ask you to read off all the ingredients for some supplements, along with the amount per tablet or capsule, and how many you ate during the previous day.

Thank you for being a part of this very important study. We look forward to talking with you.



Supplements. The Roswell person will

10/31/2022 

Appendix N. Participant Food Amounts Booklet (FAB)

# **Food**

# **Amounts**

# **Booklet**

You will use this booklet during the phone interview.

10/31/2022 

### **Squares and Rectangles**



10/31/2022 

### **Circles**




10/31/2022 




10/31/2022 

### **Thickness**




10/31/2022 
# **Measuring Spoons**




10/31/2022 

### **Eating and Serving Spoons**




10/31/2022 

# **Measuring Cups**




10/31/2022 

## Glasses




10/31/2022 

### Glasses




10/31/2022 



10/31/2022 



10/31/2022 

### Wine Glass




10/31/2022 

# Mug




10/31/2022 

## Mounds






10/31/2022 

### Mounds




10/31/2022 

### Meats




10/31/2022 

## Chicken




10/31/2022 

### Fish




10/31/2022 

Roswell Park Protocol No.: I 661820

Adapted from: Van Horn LV, Stumbo P, Moag-Stahlberg A, Obarzanek E, Hartmuller VW, Farris RP, Kimm SY, Frederick M, Snetselaar L, Liu K. The Dietary Intervention Study in Children (DISC): dietary assessment methods for 8- to 10-year-olds. J Am Diet Assoc. 1993 Dec;93(12):1396-403. Modified by Alejandra Valencia, Mary Stevens, Nutrition Coordinating Center, University of Minnesota for the Hispanic Community Health Study, Study of Latinos, 2007.

10/31/2022 

Roswell Park Protocol No.: I 661820

### Appendix O. Participant Welcome Letter

Dear POW-R Health Participant,

Welcome to the POW-R Health Program! A group of doctors and bladder cancer survivors have made this program to help you live a long and healthy life.

This mailing should include:

- 2 consent forms (1 for you to sign and mail back to us; 1 for you to keep)
- 1 Gender, Race, and Ethnicity Form (please mail back to us)
- 1 envelope (to place the signed consent form and the Gender, Race, and Ethnicity Form)
- 1 Food Amounts Booklet (Keep this for later)
- 1 Urine collection kit with one pre-paid FedEx urine shipping box

If you did not receive ALL of these things, please call us right away at: 716-845-1300, Ext 7221.

Please complete all of the forms that are white in color and mail them back to us. Place the signed consent form and the Gender, Race, and Ethnicity Form in the envelope. Place the envelop in the urine shipping box with your urine sample and mail together.

In about a week, someone will call you to ask you what you are and drank for the past day. These are called dietary recalls. You will be asked to do 3 dietary recalls.

After you complete your dietary recalls, and mail in the white forms (signed consent form; the gender, race, and ethnicity form) and the urine collection kit, you will receive the program.

Thank you again for being a part of this important study. If you have any questions, please don't hesitate to contact us at: 716-845-1300, Ext 7221.

Sincerely,

Karen Yeary, PhD

Haven yeary

Li Tang, PhD

10/31/2022 

### Appendix P. Participant Health Magazine for Intervention and Control Arm

### Intervention Magazine



10/31/2022 



# Welcome to the POW-R Health Program As a bladder cancer survivor, you know that taking care of your health is important.

As a bladder cancer survivor, you know that taking care of your health is important. You probably go and get your bladder checked often or get other treatments to keep your bladder healthy. But did you know that among bladder cancer survivors like you, there is still a 50%-80% chance that the bladder cancer could come back within 5 years? Compared to all types of cancers, bladder cancer has the highest chance of coming back.

Most bladder cancer survivors like you are doing well and don't think about the cancer coming back. Most survivors weren't even aware that they had bladder cancer to begin. When bladder cancer is in the body, most can't tell because there are no symptoms. Most survivors didn't go through intense treatment (like chemotherapy) as other cancer survivors. Many bladder cancers are caught at early stages so intense treatment is not needed.

It is good that for many survivors, the bladder cancer didn't affect their life that much. But not having a lot of symptoms and not going through a lot of treatments may make some survivors think of bladder cancer as a lesser cancer.

2 POW-R HEALTH: Power to Redefine Your Health

#### RECIPES

### Spicy Skillet Turnip Greens Recipe

A quick recipe for spicy skillet turnip greens for a comforting, home-cooked meal.

Yield: 6 servings Prep Time: 5 mins Cook Time: 20 mins Total Time: 25 mins

### INGREDIENTS

- 1 tablespoon olive oil
- 1 medium onion, cut into wedges
- 1 pound turnip greens, cleaned and chopped

1/4 cup water

Pinch brown sugar

1/4 teaspoon red pepper flakes, adjust to preference

#### INSTRUCTIONS

- 1. Drizzle olive oil into skillet over medium heat.
- 2. Add onion and cook until just tender, about 3 minutes. Then add half of turnip greens. Allow to cook down and add the remainder of the greens.
- Add water, brown sugar and red pepper flakes. Adjust the amount of red pepper to your personal taste.

Source: addapinch.com



POW-R HEALTH: Power to Redefine Your Health

### RECIPES

### Simple Arugula Salad

Yield: 4 to 6 servings

### INGREDIENTS

- 2 tablespoons olive oil
- 2 tablespoons freshly squeezed lemon juice
- 1/4 teaspoon kosher salt

Freshly ground black pepper

- 5 ounces arugula (about 5 packed cups)
- 2 ounces shaved Parmesan cheese (about 2/3 cup)

### INSTRUCTIONS

Whisk the olive oil, lemon juice, salt, and a few grinds of black pepper together in a large bowl. Add the arugula and toss to combine. Top with the shaved Parmesan and serve immediately.

### RECIPE NOTES

Make ahead: The dressing can be made up to 5 days ahead of time and stored in an airtight container in the refrigerator. Rewhisk again before using.

ource: thekitchn.co

The truth is that bladder cancer is a dangerous disease. It may come back even if you know your own body very well. Bladder cancer has a high chance of coming back. If the cancer comes back and is not caught at early stages, there is a risk of losing the bladder.

The main thing bladder cancer survivors need to do is to stop or delay the cancer from coming back. Going to your routine check-ups with doctors is good to catch bladder cancer coming back at early stages. But they are not enough. That's why a group of medical professionals, including doctors, nurses, scientists, and nutritionists, have made the POW-R Health Program. We want to make sure you live the longest, healthlest life possible so you can stay young and strong. We are here to support you. Share these materials with your spouse, partner, or others to support you too.

You most likely know that eating vegetables is a key part of eating healthy and staying healthy. Eating vegetables may be easy for you because you grew up with fresh vegetables at the dinner table. You may now eat a lot of vegetables to stay young and strong, mainly after you got cancer. But did you know that there are certain vegetables that can help stop bladder cancer from coming back? These vegetables are called power vegetables. Power vegetables are cruciferous (knoro-sifr-ub) vegetables that can help reduce death from bladder cancer by 57%, maybe by stopping or slowing down cancer growth and return. Doctors found that if made the right way, eating 1 serving of power vegetables each day can stop the growth or kill at least 50% of bladder cancer cells.

That's why doctors have made the POW-R Health Program, a program that will help you choose the vegetables (power vegetables) that are good at fighting bladder cancer.



POW-R HEALTH: Power to Redefine Your Health

POW-R HEALTH: Power to Redefine Your Health

0

10/31/2022 



### What are power vegetables?

Power vegetables are **cruciferous vegetables**: a group of vegetables where the flowers on the vegetables form the shape of a cross (in Latin, **Cruciferae** means "cross bearing"). Power vegetables include:

- Broccoli
- Turnips
- Green or white cabbage
- Brussels sprouts
- Radishes
- Arugula
- Mustard greens, and
- Other vegetables listed below

Humans have eaten power vegetables for many years. But the anti-cancer parts of power vegetables were not known until lately. Power vegetables are rich in many vitamins and minerals, such as folate, vitamins C, E, and K, and are a good source of fiber. Best for cancer survivors, power vegetables have a group of unique things called glucosinolates. Glucosinolates give power vegetables their strong smell and bitter taste. When power vegetables are cooked and eaten, glucosinolates are broken down into some active things. One of these active things is isothiocyanates. Doctors have found that isothiocvanates have strong anti-cancer actions against many types of cancer, including bladder cancer.

### Why are power vegetables good at fighting bladder cancer?

When we eat power vegetables, isothiocyanates go to the bladder through the urine and build-up in the urine. Bladder cancer cells mostly form on the inside surface of the bladder and are exposed to the urine. When the isothiocyanates builds up in the urine, bladder cancer cells get soaked in isothiocyanates that are in the urine.

Being exposed to isothiocyanates in the urine help kill bladder cancer cells and stop them from growing.

POW-R HEALTH: Power to Redefine Your Health

#### RECIPES

### Healthy No Mayo Coleslaw

This Healthy No Mayo Colesiaw recipe is the perfect middle ground between creamy, deli-style coleslaws and tangy vinegar slaws. It features a lightened-up Greek yogurt coleslaw dressing that needs just a few simple ingredients. Even better? It only takes about 5 minutes to toos together!

Yield: 9 servings, 1/2 cup each

Total Time: 30 Minutes or Less

#### INGREDIENTS

1/2 cup nonfat plain Greek yogurt

- 31/2 tablespoons cider vinega
- 3 tablespoons sugar
- 1 teaspoon kosher salt
- 1/8 teaspoon black pepper

16 ounces (about 61/4 cups) bagged colesiaw blend or shredded cabbage

### INSTRUCTIONS

- In a small bowl, combine Greek yogurt, vinegar, sugar, salt, and pepper, whisking until smooth and thoroughly combined.
- 2. Place slaw blend/cabbage in a large bowl and pour Greek yogurt dressing mixture over top. Stir to coat cabbage thoroughly.
- 3. Cover and refrigerate until using (preferably at least 30 minutes).

Make-ahead tips: This colesiaw keeps well, covered in the refrigerator, and can easily be made several hours in advance. In fact, we prefer to let it sit for at least half an hour before serving, so that the cabbage softens a bit and the whole salad melds together. We find that it's at its best, though, if eaten within a day

POW-R HEALTH: Power to Redefine Your Health

#### RECIPES

### Lemon Arugula Rigatoni Pasta Recipe

Prep Time: 15 minutes Cook Time: 10 minutes

### INGREDIENTS

- 34 pound whole wheat or gluten-free rigaton
- 4 cups baby arugula
- 15-ounce can cannellini beans 1 lemon (zest and juice)
- 2 tablespoons extra-virgin olive oil, divided
- 1 teaspoon kosher salt

% cup grated Pecorino (or Parmesan) cheese, plus more for serving (optional) Fresh ground black pepper

### INSTRUCTIONS

- 1. Bring a large pot of salted water to a boil. Cook the pasta according to package
- 2. Meanwhile, drain and rinse the cannellini beans and place them in a large bowl with 4 cups arugula. Add the lemon zest and juice of the lemon to the bowl, then add 1 tablespoon olive oil, the kosher salt, and a few grinds of black pepper. Toss gently to combine all flavors.
- 3. When pasta is done, drain it and add immediately to the large bowl with beans and arugula. Add another 1 tablespoon olive oil and ¾ cup Pecorino cheese and stir to combine (the warm pasta will wilt the arugula and warm the beans).
- 4. Serve immediately, topped with additional cheese, salt, pepper, olive oil and/or

POW-R HEALTH: Power to Redefine Your Health





- 1 Fresh or lightly cooked power vegetable eaten
- 2 Isothiocyanates released from power vegetable through digestion
- 3 Isothiocyanates are delivered to the bladder in urine
- 4 Isothiocyanates in urine soak bladder wall and directly affect abnormal bladder cells to stop any cancer from coming back

Science studies have shown that isothlocyanates from power vegetables have stopped bladder cancer from growing in animals. Isothiocyanates may fight bladder cancer through stopping chemicals that fuel cancer, guarding cells from DNA damage, killing cancer cells, stopping cancer from growing, boosting the immune system, stopping the tumor from making blood vessels, and stopping the tumor cells from moving.

Recent studies in bladder cancer survivors like you have shown that eating a lot of power vegetables, especially raw or fresh power vegetables, could help reduce death from bladder cancer by 57%, maybe by stopping or slowing down cancer growth and return. Other studies have found that if made right, eating 1 serving of power vegetables each day would make enough isothiocyanates in the urine to stop the growth or kill at least 50% of bladder cancer cells. So, there is proof that eating pow vegetables can help stop bladder cancer from coming back.

Power vegetables are not only good at fighting bladder cancer. They have lots of fiber or roughage to keep you regular. They can help you have a healthy weight. Power vegetables can also be a part of a healthy diet, which can help keep you young and

POW-R HEALTH: Power to Redefine Your Health

10/31/2022



### How can you get the most anti-cancer power from power vegetables?

The key to getting the most anti-cancer power from power vegetables is to have enough isothicoyanates in the urine and to have the inner surface of the bladder fully soaked in the isothicoyanates as long as it can. The chart on the next page lists power vegetables that are easy to find in the grocery store along with their isothiocyanates amounts when they are fresh or raw.

### What types of power vegetables should I choose?

Choose power vegetables with medium to high isothiocyanates, such as arugula, broccoli, broccoli sprouts, cabbage, mustard greens, water cress, daikon, or turnip.

### How many power vegetables should I eat?

Eat at least one serving of power vegetables per day. One serving size is 1 cup at the time you eat it. So if you have a salad with arugula, it would be 1 cup raw. If you cook the arugula, it would 1 cup cooked. 1 cup is about the size of your fist.



POW-R HEALTH: Power to Redefine Your Health

#### RECIPES

### Sautéed Greens

These sauteed greens are a breeze to make on your stove top. A little chopping and a few ingredients like garlic and tamari or soy sauce are all it takes. It's a great way to eat more greens!

Servings: 2 people Prep Time: 10 minutes Cook Time: 10 minutes

#### INGREDIENTS

- 2 bunches Swiss chard or other greens, roughly chopped
- 3 cloves garlic, chopped
- 1 tsp. low-sodium tamari or soy sauce (or to your liking)

#### INSTRUCTIONS

- 1. Water sauté the chopped garlic for a few minutes. Then add the chopped stems and a little water and sauté a few minutes. Then add the chopped stems and a little water and sauté a few minutes. Then add the rest of the greens.
- 2. Continue sautéeing the greens, turning frequently. Add more water if it dries
- 3. Add the tamari or soy sauce to your taste and continue to sauté until softened,
- 4. Serve with whole grains such as brown rice or quinoa, adding more soy sauce

Source: plantbasedcooking.com

POW-R HEALTH: Power to Redefine Your Health

### Salatet Malfouf (Lebanese Cabbage Salad)

A simple cabbage salad made with lemon juice, olive oil, garlic, and mint.

Total Time: 15 minutes

### INGREDIENTS

- 1/2 medium head of cabbage, thinly sliced
- 1 medium clove garlic, minced
- 2 Tbsp. fresh lemon juice 2 Tbsp. olive oil
- 1/4 tsp. salt
- 2 Thsp, chopped fresh dried mint leaves

### INSTRUCTIONS

- 1. In a large bowl mix the garlic, lemon juice, olive oil, salt, and mint until thoroughly combined.
- 2. Add the shredded cabbage to the bowl and toss to coat.
- 3. Let the salad sit at room temperature for 10 minutes to allow flavors to meld or cover and refrigerate to allow the flavors to meld a little more and serve at later time. Served room temperature or cold, it's a tasty salad either way.

### **NOTES & TIPS**

Drying out fresh mint leaves:

- 1. Separate the leaves from the stems and lay on a microwave safe plate in a single layer. Cook for 10 second intervals until mint begins to curl. Should only take about 30 seconds to dry.
- 2. Alternatively you can dry them out in your oven at the lowest possible temperature, place the leaves in the oven on a baking sheet for about 5 to 10
- 3. Either way you want the mint to be dry but still green

POW-R HEALTH: Power to Redefine Your Health

### Which power vegetables are high in ITCs?



POW-R HEALTH: Power to Redefine Your Health

10/31/2022




It is okay to freeze and eat power vegetables that have been frozen, but fresh is best. Just as you may have eaten fresh (not canned) vegetables when you were growing up, it is best to eat power vegetables fresh. Fresh is best because the amount of isothiocyanates may decrease from the freezing process. Fresh vegetables also have more nutrients that are good for your health. So, eating frozen power vegetables are okay, but fresh is

### What is the best way to eat power vegetables?

It is best to eat power vegetables fresh, or raw. Just like the good old days, when most vegetables were eaten fresh, it is best to eat power vegetables fresh. They can be lightly cooked too. How you cook and how long you cook will affect how much isothiocyanates a power vegetable will give you. Cooking power vegetables too much can reduce isothiocyanates. Don't use canned power vegetables. Just like in the old days when vegetables were homegrown and not canned, stay away from canned power vegetables.

DO eat power vegetables fresh or raw, or cooked a little bit (less than 10 minutes), such as:

- · stir frying
- sautéing
- microwaving
- steaming

DON'T overcook (more than 10 minutes):

- stewing
- baking



POW-R HEALTH: Power to Redefine Your Health

→ Raw

→ Microwave

POW-R HEALTH: Power to Redefine Your Health

| oday's Date: | | |
|---|---|---|
| | ting to eat more power vegetables | |
| vegetables are: | t reasons I,, want to eat more pov | wer |
| ly power vegetable | e eating goals | |
| | ge to eat serving(s) of power vegetables ea | |
| | is to eat serving(s) this week, between (dat | les) |
| and | | |
| /ho can help me | | |
| This person can he | lp me eat more power vegetables: | |
| This person can he | Ip me eat more power vegetables: | |
| - | | |
| bstacles and strat | | the |
| bstacles and strat | egles | the |
| bstacles and strat | egles<br>may make it harder for me to reach my goals and | the |
| bstacles and strat<br>The obstacles that<br>strategies I can use | egles<br>may make it harder for me to reach my goals and<br>b to overcome them are: | the |
| bstacles and strat<br>The obstacles that<br>strategies I can use | egles may make it harder for me to reach my goals and a to overcome them are: Strategles | the |
| bstacles and strat The obstacles that strategies I can use Obstacles | egles may make it harder for me to reach my goals and a to overcome them are: Strategles Strategy 1 | the |
| bstacles and strat The obstacles that strategies I can use Obstacles | egles may make it harder for me to reach my goals and to overcome them are: Strategles Strategy 1 Strategy 2 | the |
| bstacles and strat The obstacles that strategies I can use Obstacles | egles may make it harder for me to reach my goals and a to overcome them are: Strategles Strategy 1 Strategy 2 Strategy 3 | the |
| bstacles and strat The obstacles that strategies I can use Obstacles Obstacle 1 | egies may make it harder for me to reach my goals and a to overcome them are: Strategies Strategy 1 Strategy 2 Strategy 3 Strategy 1 | the |
| bstacles and strat The obstacles that strategies I can use Obstacles Obstacle 1 | egies may make it harder for me to reach my goals and a to overcome them are: Strategies Strategy 1 Strategy 2 Strategy 3 Strategy 1 Strategy 2 Strategy 2 | the |
| bstacles and strat The obstacles that strategies I can use Obstacles Obstacle 1 Obstacle 2 | egies may make it harder for me to reach my goals and a to overcome them are: Strategies Strategy 1 Strategy 2 Strategy 3 Strategy 1 Strategy 2 Strategy 2 | the |

☐ Sauté

☐ Stir-fry

→ Steam



### When is the best time of day to eat power vegetables?

Eat power vegetables at dinner time or as a late-night snack before bed. When you eat power vegetables, the isothicoyanates from the power vegetables can get in the urine within 1 hour and slowly build up in the urine over 8 hours. If you eat power vegetables during the day, the isothicoyanates could be quickly peed out of the body from peeing a lot throughout the day. If you eat power vegetables at dinner time or as a late-night snack, your body will be able to build up the isothicoyanates in our hadder Although you may pee a few times before your bladder. Although you may pee a few times before you go to the bed, a fair amount of the isothiocyanates can still build up in the urine and increase the time the inside of the bladder is soaked in isothiocyanates.



10/31/2022 

69

### Tips on how to eat more power vegetables

To get the most out of power vegetables' anti-cancer effects, it's best to eat power vegetables every day. Eating power vegetables every day can be hard, above all if you don't like vegetables. You may not like the taste, texture, or how power vegetables look. don't like vegetables. You may not like the taste, texture, or now power vegetables look. But it is vital to try. It is okey to slowly start adding more power vegetables to your diet. Eating better can also be hard because of the food ads of less healthy foods on TV. These ads are made by those who don't care about your health. You can work towards making your diet better by having more power vegetables without giving up the foods you love. If some of the foods you love are less healthy, you can still eat them a little bit AND eat more power vegetables at the same time. Ask your spouse, partner, or other possible to have. people to help you.

- · Make power vegetables in different ways. Cut them up in small pieces and put them in soup or pasta.
- · Blend power vegetables up with fruit to make a smoothie.
- · Keep power vegetables in your fridge where you can easily see them.
- Try out the recipes in this POW-R Health magazine (see page 13). These are recipes were chosen by doctors because they include power vegetables with high isothiocyanates and are easy to make.
- · Ask your spouse, partner, or someone else to make meals with power vegetables for you. Ask them to help you eat more power vegetables.



POW-R HEALTH: Power to Redefine Your Health

- $\cdot$   $\,$  Add a little sauce and/or seasonings to power vegetables to make them taste
- Store power vegetables in the crisper section of your fridge to make them last longer.
- Get power vegetables from the frozen foods section in the grocery store and store at home for easy access (for example, frozen broccoli)
- Buy already washed and cut power vegetables to eat as a snack (for example, broccolini or cauliflower)
- Make healthy eating a family and friends affairl The more support and help that you get from loved ones can make eating better simpler and more fun. Let people close to you know about your power vegetable eating goals and why you are making the change. Ask them to join you and show support. They can bring power vegetables over to you.

### Do you have questions?

In about a week, someone from the POW-R Health Team will call you to go over this magazine, answer any questions you have, and work with you to fill out your action plan (please see action plan on next page). They will also show you how to use the POW-R Health Book. Please have your copy of the magazine handy for when we call!

After talking with one of our POW-R Health Team members, you will then receive automated phone calls from the POW-R Health program. POW-R Health phone calls will show up on your phone with the phone number 716-333-7697 (POWR), so please accept phone calls from this number. This phone number is on

the POW-R Health fridge magnet, and on the POW-R Health Book



If you have any questions, please call 716-845-1300, Ext 7221.

If you need to access the POW-R automated phone system call 716-333-7697 (POWR).

POW-R HEALTH: Power to Redefine Your Health 11

Please answer

calls from 716-333-7697 (POWR)

10/31/2022

Roswell Park Protocol No.: I 661820

### Control Magazine





If you have any questions, please call 716-845-1300, Ext 7221.

If you need to access the POW-R automated phone system, call 716-333-7697 (POWR).



### Power to Redefine Your Health

INSIDE: Learn about the Health Powers of Fruits and Vegetables - Easy, Delicious Recipes



### Welcome to the

### POW-R Health Program

You probably already know that eating fruits and vegetables is an important part of eating healthy and staying healthy. Eating fruits and vegetables may have come easier to you because you grew up with fresh fruit and vegetables at the kitchen table. You may already be eating a lot of fruits and vegetables to stay young and strong, especially since your diagnosis.

Most bladder cancer survivors like you are doing well. Most survivors weren't even aware that they had bladder cancer to begin. When bladder cancer is in the body, most can't tell because there are no symptoms. Most survivors didn't go through intense treatment (like chemotherapy) as other cancer survivors. Many bladder cancers are caught at early stages so intense treatment is not needed. Not having a lot of symptoms and not going through a lot of treatments may make some survivors think of bladder cancer as a lesser cancer. The truth is that bladder cancer is a dangerous disease. No matter what your personal experience with bladder cancer is, living a healthy lifestyle is very important to all cancer survivors.

2 POW-R HEALTH: Power to Redefine Your Health

### Apples and Peanut Butter (Apple Slices)

Yield: 1 serving

### INGREDIENTS

- 1 firm eating apple (I like Gala the best)
- 2-4 tablespoons peanut butter (crunchy or creamy)

### INSTRUCTIONS

- 1. Core and slice apple into wedges.
- 2. Divide the peanut butter evenly among the slices. I usually spread mine along

Source: food.com

POW-R HEALTH: Power to Redefine Your Health

h 15

10/31/2022 

# Avocado Fruit Salad Yield: 6 servings Total Time: 20 minutes

### INGREDIENTS

1/2 cup plain yogurt

2 tablespoons honey

- 1 teaspoon grated lemon zest
- 1 teaspoon plus 2 tablespoons lemon juice, divided
- 3 medium ripe avocados, peeled and cubed
- 1 medium apple, chopped
- 1 cup halved seedless grapes
- 1 can (11 ounces) mandarin oranges, drained
- 1 medium firm banana, cut into 1/4-inch slices

#### INSTRUCTIONS

For dressing, mix yogurt, honey, lemon zest and 1 teaspoon lemon juice. Toss avocados with remaining lemon juice.

In a large bowl, combine remaining ingredients; gently stir in avocados. Serve with dressing,  $% \left( 1\right) =\left( 1\right) \left( 1\right) \left$ 

ource: tasteofhome.con

That's why a group of medical professionals, including doctors, nurses, scientists, and nutritionists, have made the POW-R Health Program. We want to make sure you live the longest, healthiest life possible. We are here to support you. Share these materials with your spouse, partner, friends, family and others to support you too.

#### What are fruits and vegetables?

Fruit and vegetables are plants that have lots of minerals, vitamins, and other healthy things that are good for the human body. A fruit develops from the flower of a plant, while the other parts of the plant are known as vegetables. Fruits have seeds, while vegetables can have roots, stems and leaves.

Some common fruits are:

- · Apples and pears
- · Citrus oranges, grapefruits, mandarins and limes
- Stone fruit nectarines, apricots, peaches and plums
  - Tropical and exotic bananas and mangoes
- Berries strawberries, raspberries, blueberries, kiwi, and passionfruit
- · Melons watermelons and honeydev
- · Tomatoes and avocados

Some common vegetable types are:

- · Leafy green lettuce and spinach
- Cruciferous cabbage, cauliflower, Brussels sprouts and broccoli
- · Marrow pumpkin, cucumber, and zucchini
- Root potato, sweet potato and yam
- Edible plant stem celery and asparagus
- · Allium onion, garlic, and shallot



POW-R HEALTH: Power to Redefine Your Health

POW-R HEALTH: Power to Redefine Your Health

### How are fruits and vegetables good for you?



Having a healthy diet full of fruits and vegetables is very important. Research has shown that eating fruits and vegetables can help you live longer. Eating fruits and vegetables reduces the risk of getting some cancers, highe blood pressure (hypertension), heart disease, and diabetes. A recent study said that eating about 2 cups (200 g) of fruits and vegetables each day can reduce the risk of heart disease by up to 16%, stroke by 18%, and cancer by 4%. Cancer survivors who eat at least 5 servings of fruits and vegetables report better overall wiel-being.

Fruits and vegetables have all of these great health benefits because they have a lot of vitamins C and A, electrolytes, and antioxidants. Vitamin C protects the immune system and protects the body from harmful effects of pollutants and toxins. Vitamin C protects cells and molecules from damage that causes many diseases, including cancer. Fruits and vegetables are also a great source of fiber. The fiber in fruits and vegetables obvers cholesterol, which reduces heart disease risk. The fiber in fruits and vegetables can also help control the body's blood sugar, which reduces risk of diabetes fruits and vegetables can also help you have a healthy weight by giving you lots of fiber and water, which can fill you up without giving too many calories.

# How can you get the best health benefits from eating fruits and vegetables?

What kinds of fruits and vegetables should I eat?

### VEGETABLES

- · Fresh, frozen, and canned vegetables can all be a part of healthy eating.
- Fresh vegetables are best! Fresh vegetables usually give your body the most nutrients. Try to eat as many different types of vegetables as you can.
- Prozen vegetables have the same amount of nutrients as fresh vegetables and can be cheaper to buy. If you buy frozen vegetables, look for types that don't have added butter, sauces, or cheese. These will have added calories and fat that can make it harder to have a healthy diet.
- Canned vegetables can be high in salt, so if you buy canned vegetables make sure you look for the 'no salt' ones.
- 4 POW-R HEALTH: Power to Redefine Your Health

### Baked Parmesan Zucchini

Crisp, tender Parmesan zucchini sticks oven-roasted to absolute perfection. It's healthy, nutritious and completely addictive!

Yield: 4 servings Prep Time: 10 Minutes Cook Time: 20 Minutes

### INGREDIENTS

- 4 zucchini, quartered lengthwise
- 1/2 cup freshly grated Parmesan
- ½ teaspoon dried thyme ½ teaspoon dried oregano
- √2 teaspoon dried oregand
  √2 teaspoon dried basil
- 1/4 teaspoon garlic powder
- Kosher salt and freshly ground black pepper, to taste
- 2 tablespoons olive oil
- 2 tablespoons chopped fresh parsley leaves

### INSTRUCTIONS

- Preheat oven to 350 degrees F. Coat a cooling rack with nonstick spray and place on a baking sheet; set aside.
- In a small bowl, combine Parmesan, thyme, oregano, basil, garlic powder, salt and pepper, to taste.
- Place zucchini onto prepared baking sheet. Drizzle with olive oil and sprinkle with Parmesan mixture. Place into oven and bake until tender, about 15 minutes. Then broil for 2-3 minutes, or until crisp and golden brown.
- 4. Serve immediately, garnished with parsley, if desired.

Source: damndelicious.net

POW-R HEALTH: Power to Redefine Your Health

13

10/31/2022 

### Butter Parmesan Corn

Total Time: Under 30 minutes

#### INGREDIENTS

6 half ears corn, cleaned, husked

2 tablespoons butter, softened ½ cup Parmesan cheese, grated

Salt, to taste

### Pepper, to taste

- 1. Preheat oven to 375°F (190°C).
- Coat each ear of corn in a thin layer of butter and roll in the parmesan cheese to coat.
- 3. Place corn in a square baking dish and sprinkle with salt and pepper.
- 4. Bake for 25 minutes.
- 5. Enjoy!

Source: tastv.co

#### FRUIT

- Fresh, frozen, and canned fruit can all be a part of healthy eating.
- Fresh fruit is best! Fresh fruit usually gives your body the most nutrients. Try to eat as many different types of fruit as you can.
- Frozen fruit can last longer than fresh fruit and can be cheaper to buy.
- Canned fruit can be high in sugar and calories, so buy canned fruit in 100% fruit juice with no sugar added.

### How many fruits and vegetables are you supposed to eat?

Eat 2<sup>1</sup>/<sub>2</sub> to 3 cups of vegetables and 1<sup>1</sup>/<sub>2</sub> to 2 cups of fruit each day. ½ cup is about the size of the front part of your fist. 1 cup is about the size of a baseball.

### SERVING SIZES





POW-R HEALTH: Power to Redefine Your Health

12 POW-R HEALTH: Power to Redefine Your Health

### How to prepare fruits and vegetables

You can eat a lot of fruits and vegetables raw. You can also cook them in many different ways:

- sautéeing
- · microwaving
- steaming
- · baking
- stir-frying
   stewing
- · boiling

### Tips on how to eat more fruits and vegetables

You can buy fruits and vegetables from many different places. You can buy them from your local grocery store, farmer's market, and online. Here are some tips on how to eat more fruits and vegetables:

- Have a healthy morning. Add sliced fruit, like a sliced banana, to your cereal for breakfast.
- 6 POW-R HEALTH: Power to Redefine Your Health

### Cucumber Salad with Grapes and Almonds

Cucumber salad with grapes, toasted almonds and a little garlic—essentially a deconstructed white gazpacho! Perfectly balanced, cool and refreshing summer salar!

Servings: 4 people Prep Time: 30 minutes Cook Time: 5 minutes

### INGREDIENTS

1/4 cup slivered and blanched almonds

- 1 pound cucumbers, peeled if the peel is bitter, unpeeled if not Kosher salt
- 1 teaspoon minced garlic
- About 20 green grapes, sliced in half
- 2 tablespoons extra-virgin olive oil
- 1 teaspoon sherry or white wine vinegar
- 2 teaspoons minced chives, for garnish

### INSTRUCTIONS

 Prep the cucumbers: Slice the cucumbers in half lengthwise. Use a spoon to scoop out the seeds in the middle, discard the seeds. If using rather large cucumbers, slice them again lengthwise. Then cut them crosswise into ¼-inch to ¼-inch slices.

Place in a large bowl and sprinkle with a teaspoon of kosher salt. Toss to distribute the salt evenly around the cucumber pieces.

Let sit for 20 to 25 minutes while the salt helps pull excess moisture out of the cucumbers.

- Toast the slivered almonds in a small pan over medium-high heat, tossing them often, until they start to brown and smell good. Move to a bowl to cool.
- Combine: Mix the cucumbers, almonds, garlic, grapes, olive oil, and vinegar together in a large bowl and add more salt to taste. Garnish with chives and serve.

Source: simplyrecipes.co

POW-R HEALTH: Power to Redefine Your Health

11

10/31/2022

### Tangy Carrot Slaw

Servings: 6 as a side dish

#### INGREDIENTS

1/4 cup Dijon mustard

1/4 cup olive oil

3 tablespoons red wine vinegar or freshly squeezed lemon juice

1 teaspoon kosher salt

Freshly ground black pepper

2 pounds carrots, peeled and shredded (about 6 cups)

1/4 cup thinly sliced scallion

#### INSTRUCTIONS

- Place the mustard, oil, vinegar or lemon juice, salt, and a few generous grinds of pepper in a large bowl and whisk to combine. Add the carrots and scallions and toss well to evenly coat.
- 2. Cover and refrigerate for at least 30 minutes or overnight to allow the flavors to meld. Taste and season with more salt and pepper as needed before serving.

Leftovers can be stored in an airtight container in the refrigerator for up to 3 days. Source: thekitchn.com

- Bag it! Toss an apple, banana or other fruit in your
- Put pizzazz in your soup. Add some grated carrots or canned or frozen vegetables in a soup, casserole, or other main dish.
- Save time cooking! Buy canned or frozen vegetables to have easy access to vegetables for meals.
- Toss it! Have more tossed salads with a lot of different vegetables and low-fat dressing.
- Don't have time? Drink 100% vegetable juices.
- Make them last. Store fruits and vegetables in the crisper in your refrigerator to make them last longer. Freeze fruits and vegetables to keep them from spoiling.
- Save money! Buy in-season fruits and vegetables, or buy less expensive fruits and vegetables like apples, oranges, bananas, carrots, and greens.
- Add chopped up vegetables to your eggs or potatoes. Try onions, celery, green or red bell peppers, or spinach.
- Put vegetables in your sandwich, like cucumber, sprouts, tomato, lettuce or avocado
- Have a piece of fruit or raw vegetables handy, such as green or red bell peppers, green beans, celery or carrots.
- Carry dried fruit, such as raisins, dates or dried apricots, in your pocket or purse.
- On hot days, munch on a bowl of frozen fruits or vegetables, such as grapes, peas or banan
- Add a side of steamed or microwaved vegetables frozen veggies are fine!
- When making rice, add some frozen peas for the last three minutes of cooking.
- If you don't like how some fruits or vegetables taste, look, or feel, try cooking or seasoning them in different ways. You will most likely find a new way to enjoy them! Be creative!



POW-R HEALTH: Power to Redefine Your Health

- Don't give up your favorite foods. You can still eat your favorite foods in moderation, while still eating more fruits and vegetables.
- TV and media advertise a lot of less healthy food choices. If you find yourself being tempted to eat foods that are less healthy, think of ways to make those foods healthier by adding vegetables or enjoying a smaller portion size.

### Do you have questions?

In about a week, someone from the POW-R Health Team will call you to go over this magazine, answer any questions you have, and work with you to fill out your action plan (please see action plan on next page). They will also show you how to use the POW-R Health Book. Please have your copy of the magazine handy for when we call!

POW-R HEALTH: Power to Redefine Your Health

Please answer After talking with one of our POW-R Health Team calls from 716-333-7697 (POWR) members, you will then receive automated phone calls from the POW-R Health program. POW-R Health phone calls will show up on your phone with the phone number 716-333-7697 (POWR), so please accept phone calls from this number. This phone number is on the POW-R Health fridge magnet, and on the POW-R Health Book.

If you have any questions, please call 716-845-1300, Ext 7221

If you need to access the POW-R automated phone system. call 716-333-7697 (POWR)

| My personal action plan to eat more fruits and v | egetables |
|---|---|
| Today's Date: | |
| My reasons for wanting to eat more fruits and vegetables The most important reasons I,, want to eat more fruits are: | iits and |
| My fruit eating goals | <u></u> |
| In 6 months, I pledge to eat cups of fruit each day. | |
| My short-term goal is to eat cups of fruit this week, between (dates) and | |

My vegetable eating goals In 6 months, I pledge to eat \_

\_ cups of vegetables each day.

My short-term goal is to eat \_\_\_\_\_ (dates) \_\_\_\_\_ and \_\_\_\_\_ \_ cups of vegetables this week, between

This person can help me eat more fruits and vegetables:

Obstacles and strategies

The obstacles that may make it harder for me to reach my goals and the strategies I can use to overcome them are:

| Obstacles | Strategles |
|------------|------------|
| | Strategy 1 |
| Obstacle 1 | Strategy 2 |
| | Strategy 3 |
| Obstacle 2 | Strategy 1 |
| | Strategy 2 |
| | Strategy 3 |

My plan this week to eat more fruits and vegetables

The next time I go to the grocery store, I will buy these fruits and vegetables

POW-R HEALTH: Power to Redefine Your Health

POW-R HEALTH: Power to Redefine Your Health

10/31/2022  Roswell Park Protocol No.: I 661820

### Appendix Q. Live Call Scripts (Intervention and Control)

| Intervention | | | | |
|-----------------|-----------------|-------|-------------|-----------|
| Participant ID: | Staff Initials: | Date: | | |
| Start Time: | End Time: | | ☐ Treatment | ☐ Control |

### Materials that should have been sent to participant

Cover Letter/Welcome Letter

POW-R Health Magazine

POW-R Track Book (24 copies)

Refrigerator Magnet

| PART A: | Getting participant on the phone, call intro, packet receipt |
|---|---|
| Note: Only make three attempts to reach the participant | |
| ☐ Phone Answ | ered |
| | ame] from the POW-R Health program calling for [participant name], she/he is expecting my call. Is nome/available right now? |
| Yes | Hi [participant name] I'm calling to review the POW-R Health program materials with you. It should take about 60 minutes; do you have time to complete it right now? |

Time to call back No That's okay, can we schedule a time that would work

better for you? Thanks, I will give you a call then.

| ☐ Leaving Message |
|-------------------|
|-------------------|

1st Attempt This is [staff name] from the POW-R Health program calling for [participant name]. I'm calling to review the POW-R Health program materials with you, which should take about 60 minutes. I'll try calling you again, but if you would like to call me back and let me know a good time for us to chat, I can be reached at 716-697-4615/716-720-2308. Thanks, and I hope I catch up with you soon!

2<sup>nd</sup> Attempt Hello again, this is [staff name] from the POW-R Health program calling for [participant name]. I left a message with you on [date] and I am calling you back to review the POW-R Health program materials with you, which should take about 60 minutes. I'll try calling you one more time, but if you would like to call me back and let me know a good time for us to chat, I can be reached at 716-697-4615/716-720-2308. Thanks, and I hope I catch up with you soon!

3<sup>rd</sup> Attempt Hello again, this is [staff name] from the POW-R Health program calling for [participant name]. I left a message with you on\_\_\_\_\_[date], and I am calling you back to review the POW-R

Health program materials with you, which should take about 60 minutes. If you would like to call me back and let me know a good time for us to chat, I can be reached at 716-697-4615/716-720-

2308. Thanks, and I hope I catch up with you soon!

10/31/2022 

### ☐ Confirm Intervention Packet Receipt

We are glad you are a part of the program. We put a program packet in the mail for you about the POW-R Health Program. The packet should have included a magazine, booklets, and a magnet.

A1. Did you receive the program packet in the mail?

If YES: (Go to Question A2)

*If NO:* It's really important that you have your packet before we go over it. Let me make a note to send you the packet again. What is your mailing address? I'll call you again after your packet is sent. Thank you for taking the time to talk with me. I'll talk to you again soon.

END CALL.

A2. If so, did you have time to review the information in this packet?



If YES: Okay great, I'm glad you got a chance to review the material. Just to make sure that the magazine clearly conveyed the information, I will now ask you some questions to go over the main points of the magazine. We will then work together to create your personal action plan to eat more power vegetables. Before we begin, please pull out the packet we sent. It would really help to have them with you for the later part of the call. Please have a pen handy too (Go to PART D).

*If NO*: That is okay. We can still go over what is in the packet right now. Before we begin, please pull out the packet we sent. It would really help to have them with you for the later part of the call Please have a pen handy too. (Go to PART B)

### ☐ PART B: OVERVIEW

I'm going to begin by going over the POW-R Magazine. After I go over the magazine's contents, we'll complete your personal action plan (page 12). I'll then go over the POW-R Books and the magnet. So, let's start with the POW-R Magazine. Please have your POW-R Magazine next to you so you can follow along what I'm going to review.

### ☐ PART C: MAGAZINE CONTENT

### **■ Welcome to the POW-R Health Program (page 2)**

- Among bladder cancer survivors like you, there is still a 50%-80% chance that the bladder cancer could come back within 5 years
- Compared to all types of cancers, bladder cancer has the highest chance of coming back
- If the cancer comes back and is not caught at early stages, there is a risk of losing the bladder
- Going to your routine check-ups with doctors is good to catch bladder cancer coming back at early stages. But they are not enough.
- Doctors made the **POW-R Health Program** to make sure you live the longest, healthiest life possible
- Certain vegetables that can help stop bladder cancer from coming back. These vegetables are called power vegetables
- Power vegetables help reduce death from bladder cancer by 57%

Interesting convo points

10/31/2022 

### ☐ What are Power Vegetables? (page 4)

- Power vegetables are cruciferous vegetables
- Examples of power vegetables are Broccoli, Turnip, Cabbage, and Arugula
- When power vegetables are eaten, they break down into active things. One of these active things is isothiocyanates (eye-so-thye-oh-sigh-nates) or ITCs.
- ITCs have strong anti-cancer actions against many types of cancer, including bladder cancer.
- Do you have any questions about what I've covered so far?

Interesting convo points

### $\square$ How are Power Vegetables Good at Fighting Bladder Cancer? (pages 4 and 5)

- (Refer participant to picture in magazine on page 5)
- (Go through Steps 1-4 of the picture)
- There is proof that eating power vegetables can help stop bladder cancer from coming back

### How Can You Get the Most Anti-Cancer Power From Power Vegetables

- The key to getting the most anti-cancer power from power vegetables is to have enough ITCs in the urine and to have the bladder inner surface fully soaked in the isothiocyanates as long as it can.
- Choose power vegetables that are high or medium in ITCs (look at page 7 in magazine for medium and high ITC power vegetables)
- Eat at least one serving of power vegetables per day. One serving size is 1 cup of power vegetables at the time you eat it. So if you eat one cup of arugula raw, that would be 1 cup raw. If you eat arugula cooked, that would be 1 cup of cooked arugula. One cup is about the size of your fist.
- It is best to eat power vegetables fresh, or raw. They can be lightly cooked too, for no more than 10 minutes. If you cook power vegetables too much it will reduce their anti-cancer power. Don't use canned power vegetables.
- Eat power vegetables at dinner time or as a late-night snack before bed. When you eat power vegetables, the ITCs from the power vegetables can get in the urine within 1 hour and slowly build up in the urine over 8 hours. If you eat power vegetables during the day, you could lose a lot of ITCs in your urine from going to the bathroom throughout the day. If you eat power vegetables at dinner time or as a late-night snack, your body will be able to build up the ITCs in your bladder. Although you may go to the bathroom a few times before you go to the bed, a fair amount of the ITCs can still build up in the urine and increase the time the bladder is soaked in ITCs.

### ☐ Tips to Eat More Power Vegetables (page 10)

• Look at pages 10 and 11 in your magazine for tips on how to eat more power vegetables

10/31/2022 

### ☐ Part D: Going over Magazine Components: Teach Back Opportunity #1

Just to make sure that the magazine clearly conveyed the information, I am now going to ask you a few questions to review some of the main points of the magazine. You may feel like I'm testing you, but the purpose of this is to make sure that the magazine communicated the information to you clearly. Are you ready? Let's go!

Note: For a question to be answered correctly, all parts of the question must be answered correctly.

TB1 What is a power vegetable?

Correct: A cruciferous vegetable

Correct: A cruciferous vegetable

**CORRECT:** Yes, that's right! A power vegetable is a certain type of vegetable called cruciferous vegetables.

**INCORRECT:** Power vegetables are cruciferous vegetables.

**CORRECT:** Yes, that's right- good job! There are a lot of vegetables that are considered cruciferous vegetables. More cruciferous vegetables are listed in your POW-R Health Magazine.

**INCORRECT**: Ok, no problem, you missed [state answers that are incorrect and correct]. Your POW-R Health Magazine lists some power vegetables on page 7.

How many power vegetable servings do you need to eat each day.

\*\*Correct Answer: 1 serving/day\*

\*\*Correct

**CORRECT:** Excellent, you're right. You only need to eat one power vegetable serving a day to help stop bladder cancer from coming back.

**INCORRECT:** Okay, no problem, the correct answer is 1 serving or cup a day. You only need to eat one power vegetable serving a day to help stop bladder cancer from coming back.

10/31/2022 

TB4 What is the amount of 1 serving of a power vegetable?

\*\*Correct Answer: 1 cup at time of eating/consumption\*

\*\*No Yes\*\*

**CORRECT:** Excellent, you're right. 1 serving of a power vegetable is 1 cup at the time you eat it. 1 cup is about the size of your fist.

**INCORRECT:** Okay, no problem, the correct answer is 1 serving of a power vegetable is 1 cup at the time you eat it. 1 cup is about the size of your fist.

TB5 QUESTION: What is an isothiocyanate or ITC?

No Yes

Correct Answer: An active compound in power vegetables that has strong anti-cancer properties

**CORRECT:** Ok great, you really seem to understand what an isothiocyanate/ITC is.

**INCORRECT:** Isothiocyanates/ITCs are an active compound in power vegetables that has strong anti-cancer properties.

TB6 What is the best way to prepare power vegetables so they give you most isothiocyanates/ITCs?

\*\*Correct Answer: It is best to eat power vegetables fresh or raw. You can also lightly cook them too (cook for less than 10 minutes).

\*\*Correct No Yes\*\*

\*\*Correct No Yes\*\*

\*\*Correct Answer: It is best to eat power vegetables fresh or raw. You can also lightly cook them too (cook for less than 10 minutes).

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** It's best to eat power vegetables fresh or raw. If you want to cook them, it's best to eat them lightly cooked, where you cook them for less than 10 minutes.

TB7 Why is it important to eat power vegetables at dinner or as a late-night snack before bedtime?

\*\*Correct Answer: Isothiocyanates from power vegetables go to the urine. The isothiocyanates in the urine soak the inside of the bladder; the longer the isothiocyanates in the urine are in the bladder, the longer the bladder will be exposed to the anti-cancer activities. Many people urinate several times throughout the day, and less often at night. If you eat power vegetables later at night, there is a greater chance that the isothiocyanates from the power vegetables will stay in your bladder longer.

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** Isothiocyanates/ITCs from power vegetables goes to your urine. The urine then goes to your bladder. The isothiocyanates in your urine will work to kill any cancer cells in your bladder. The longer the bladder is exposed to the isothiocyanates in your urine, the longer it will be exposed to anti-cancer activities. Many people urinate several times a day a less often at night. So, there is a greater chance that the isothiocyanates from the power vegetables will say in your bladder longer if you eat power vegetables at night.

10/31/2022 

| Scoring | Circle all questions that were answered <u>incorrectly</u> . | none | TB1 | TB2 | # Incorrect |
|---|---|---|---|---|---|
| | | TB3 | TB4 | TB5 | |
| | | ТВ6 | ТВ7 | | |

**ALL CORRECT:** Excellent job! You understand the main points of the POW-R Magazine and you got all of those questions correct. Now let's move on and put together an Action Plan! [Go to Part F]

ANY INCORRECT: [GO TO PART E]

### □ Part E: Going over Magazine Components: Teach Back Opportunity #2

Only ask questions that were answered incorrectly in Part D. SKIP if all questions were answered correctly in Part D.

Is this part applicable?

No Yes

You did a good job remembering information that I just covered. I know there was a lot of information covered. So, let's just briefly recap the ones you missed.

**TB1.2** What is a power vegetable?

Correct: A cruciferous vegetable

Correct **No Yes** 

**CORRECT**: Yes, that's right! A power vegetable is a certain type of vegetable called cruciferous vegetables.

**INCORRECT:** Power vegetables are cruciferous vegetables.

**TB2.2** Please give me three examples of power vegetables.

Correct Answer: Anything listed in the POW-R Health magazine.

| 1) | | Correct |
|----|------|---------|
| 1) | — No | Yes |
| 2) | _ | |
| 3) | | |

**CORRECT:** Yes, that's right- good job! There are a lot of vegetables that are power vegetables.

**INCORRECT:** Ok, no problem, you missed [state answers that are incorrect and correct]. There is a list of power vegetables in your POW-R Magazine on page 7.

**TB3.2** How many power vegetable servings do you need to eat each day.

Correct

No Yes

Correct Answer: 1 serving/day

**CORRECT:** Excellent, you're right. You only need to eat one power vegetable serving a day to help stop bladder cancer from coming back.

**INCORRECT:** Okay, no problem, the correct answer is 1 serving a day. You only need to eat one power vegetable serving a day to help stop bladder cancer from coming back.

10/31/2022 

**TB4.2** What is the amount of 1 serving of a power vegetable? No Yes Correct Answer: 1 cup at time to eating/consumption

**CORRECT:** Excellent, you're right. 1 serving of a power vegetable is 1 cup at the time you eat it. 1 cup is about the size of your fist.

**INCORRECT:** Okay, no problem, the correct answer is 1 serving of a power vegetable is 1 cup at the time you eat it. 1 cup is about the size of your fist.

Correct **TB5.2 QUESTION:** What is an isothiocyanate/ITC? No Yes Correct Answer: An active compound in power vegetables that has strong anti-cancer properties

**CORRECT:** Ok great, you really seem to understand what an isothiocyanate is.

**INCORRECT:** Isothiocyanates/ITCs is an active compound in power vegetables that has strong anti-cancer properties.

Correct **TB6.2** What is the best way to prepare power vegetables so they give you most isothiocyanates/ITCs? No Yes Correct Answer: It is best to eat power vegetables fresh or raw. You can also lightly cook them too (cook for less than 10 minutes).

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** It's best to eat power vegetables fresh or raw. If you want to cook them, it's best to eat them lightly cooked, where you cook them for less than 10 minutes.

**TB7.2** Why is it important to eat power vegetables at dinner or as a late night snack before bedtime?

> Correct Answer: Isothiocyanates from power vegetables go to the urine. The isothiocyanates in the urine soak the inside of the bladder; the longer the isothiocyanates in the urine are in the bladder, the longer the bladder will be exposed to the anti-cancer activities. Many people urinate several times throughout the day, and less often at night. If you eat power vegetables later at night, there is a greater chance that the isothiocyanates from the power vegetables will stay in your bladder longer.

Correct No Yes

Correct

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** Isothiocyanates/ITCs from power vegetables goes to your urine. The urine then goes to your bladder. The isothiocyanates in your urine will work to kill any cancer cells in your bladder. The longer the bladder is exposed to the isothiocyanates in your urine, the longer it will be exposed to anti-cancer activities. Many people urinate several times a day a less often at night. So there is a greater chance that the isothiocyanates from the power vegetables will say in your bladder longer if you eat power vegetables at night.

10/31/2022  Roswell Park Protocol No.: I 661820

| Scoring | Circle all questions that were answered <u>incorrectly</u> . | none<br>TB3 | TB1<br>TB4 | TB2 | # Incorrect |
|---|---|---|---|---|---|
| | | тв6 | TB7 | 150 | |

**ALL** *CORRECT*: Excellent job! You're an expert now on the POW-R Health Magazine and you got all of those questions correct. Now let's move on and put together an Action Plan! *[Go to Part F]]* 

**ANY INCORRECT:** We'll go over these questions one more time before we end our call today. [GO TO PART F]

10/31/2022 

### □ Part F: Complete Action Plan with Participant

Now let's go to the Action plan, which is on page 12 of the POW-R Health Magazine. Please fill out this page with me.

| ☐ Reasons for joining POW-R Health | |
|---|---|
| What are the most important reasons you have for oining the POW-R Health Program. Write this/these down in your action plan. | Participant reason(s): |
| ☐ Power vegetable eating goals | |
| Let's set some short- and long-term goals. Let's start with a long-term goal. In 6 months, which is by the end of this program, how many power vegetable cups do you pledge to eat each day. | Long term goal |
| Now let's set your short-term goal. For this week, how many cups of power vegetables will you try to eat this week? | Short-term goal |
| ☐ Who can help me | |
| Who can help you eat more power vegetables? Who can support you? | Support person |
| ☐ Power vegetable obstacles and strategies | |
| Let's now talk about some obstacles that could<br>make it harder for you to complete your plan. What<br>are one or two obstacles that could make it harder | Obstacle 1 |
| for you to eat your power vegetables every day? | Obstacle 2 |
| What are some strategies you could use to help overcome the obstacles you listed? | Obstacle 1, Strategies (2-4) |
| | Obstacle 2, Strategies (2-4) |

10/31/2022 

| $\square$ My plan this week to eat more power vegetables | |
|---|---|
| Now let's make a plan to eat more power vegetables this week. The next time you or someone else goes to the grocery store, which power vegetables will you buy with medium to high isothiocyanates (page 7)? | Power vegetables to buy |
| The next time you eat power vegetables, how will you make them? Remember that when you cook the power vegetable, to cook it for less than 10 minutes. | Raw, microwave, sauté/stir-fry, steam |

### ☐ Part G: Go over POW-R Track Book

One of the things you received in the packet we mailed to you is a POW-R Book. Please have your POW-R Book ready to review. In this book, I am asking that you keep track of how many power vegetables you eat every day, and each week. Science shows that keeping track of what you eat is a powerful way to change your habits. Keeping track of how many power vegetables you eat will help you eat more power vegetables. Let's go over all of the parts of the POW-R Book.

| DOOK. | | | |
|---|---|---|---|
| Check box when section is covere | ed | | |
| 1. 1 POW-R book for each week; 24 sent to you—1 is for practice to use now. We are asking you to keep track of how many power vegetables you eat every week for the entire | 3. 7 days in one POW-R book | 5. Each day you say whether you ate at least 1 power vegetable cup where you prepared it in a POW-R Health Preferred way (explain what this is) | 7. On the back is<br>the phone number<br>of the person from<br>our team that you<br>can call if you<br>have any |
| program. 2. Cover page—write down | 4. Each day you write down | 6. On the first page, is where | questions. 8. Any questions? |
| dates of the week you are keeping track | how many cups of power vegetables you had at dinner or after dinner. Only write down those power vegetables you ate at dinner or after dinner (have them open book) | you will write down the total<br>number of power vegetables<br>you at dinner or after dinner<br>for that week. After our phone<br>call, you will receive<br>automated messages and will<br>be asked to enter the number<br>of cups of power vegetables<br>you ate for the week. | 6. Party questions: |

Let's practice using the POW-R Track Book.

| ☐ Practice using POW-R Track Book | | | | | |
|---|---|---|---|---|---|
| Take a POW-R Track Book. Can you think back this past week of any power vegetables you ate at | Monday | Tuesday | | Wed | |
| dinner or after dinner? If you did not eat any power vegetables, how about any type of vegetable? Let's go through each day. | Thursday | Friday | Sat | Sunday | |
| Not let's add how many cups you ate that week | Total | Correct | | | |
| | | | ٨ | lo | Yes |

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** Ok, so the correct total is X. Let's try that again to make sure you can use the POW-R Book correctly.

Feel free to use a calculator if that would make things easier.

10/31/2022 
## ☐ Part H: Going over magazine components: Teach Back Opportunity #3

Only ask questions that were answered incorrectly in Part E. SKIP if all questions were answered correctly in Part D or E.

| Is this Part applicable? | No | Yes |
|--------------------------|----|-----|
|--------------------------|----|-----|

Before we end the call, I just want to re-ask you the questions about the key points from the magazine that you were not able to recall last time

TB1.3 What is a power vegetable?

\*\*Correct: A cruciferous vegetable\*

\*\*Correct: A c

**CORRECT:** Yes, that's right! A power vegetable is a certain type of vegetable called cruciferous vegetables.

**INCORRECT:** Power vegetables are cruciferous vegetables.

**CORRECT:** Yes, that's right- good job! There are a lot of vegetables that are considered cruciferous vegetables.

**INCORRECT:** Ok, no problem, you missed [state answers that are incorrect and correct]. If you look at on page X of your POW-R Health Magazine, there is a list of cruciferous vegetables.

TB3.3 How many power vegetable servings do you need to eat each day.

\*\*Correct Answer: 1 serving/day\*\*

\*\*Correct Answer

**CORRECT:** Excellent, you're right. You only need to eat one power vegetable serving a day to help stop bladder cancer from coming back.

**INCORRECT:** Okay, no problem, the correct answer is 1 serving a day. You only need to eat one power vegetable serving a day to help stop bladder cancer from coming back.

TB4.3 What is the amount of 1 serving of a power vegetable?

\*\*Correct Answer: 1 cup at time of eating/consumption.\*\*

Correct Answer: 1 cup at time of eating/consumption.

Correct Answer: 1 cup at time of eating/consumption.

**CORRECT:** Excellent, you're right. 1 serving of a power vegetable is 1 cup at the time you eat it. 1 cup is about the size of your fist.

**INCORRECT:** Okay, no problem, the correct answer is 1 serving of a power vegetable is 1 cup at the time you eat it. 1 cup is about the size of your fist.

10/31/2022 

| TB5.3 | QUESTION: What is an isothiocyanate? | No | Correct<br><b>Yes</b> |
|---|---|---|---|
| | Correct Answer: An active compound in power vegetables that has strong anti-cancer properties | | |

**CORRECT:** Ok great, you really seem to understand what an isothiocyanate is.

**INCORRECT:** Isothiocyanates are an active compound in power vegetables that has strong anti-cancer properties.

TB6.3 What is the best way to prepare power vegetables so they give you most isothiocyanates?

\*\*Correct Answer: It is best to eat power vegetables fresh or raw. You can also lightly cook them too (cook for less than 10 minutes).

\*\*Correct No. Yes\*\*

\*\*Correct Answer: It is best to eat power vegetables fresh or raw. You can also lightly cook them too (cook for less than 10 minutes).

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** It's best to eat power vegetables fresh or raw. If you want to cook them, it's best to eat them lightly cooked, where you cook them for less than 10 minutes.

| TB7.2 | Why is it important to eat power vegetables at dinner or as a late night snack before bedtime? | Correct<br>No Yes |
|---|---|---|
| | Correct Answer: Isothiocyanates from power vegetables go to the urine. The isothiocyanates in the urine soak the inside of the bladder; the longer the isothiocyanates in the urine are in the bladder, the longer the bladder will be exposed to the anti-cancer activities. Many people urinate several times throughout the day, and less often at night. If you eat power vegetables later at night, there is a greater chance that the isothiocyanates from the power vegetables will stay in your bladder longer. | |

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** Isothiocyanates from power vegetables goes to your urine. The urine then goes to your bladder. The isothiocyanates in your urine will work to kill any cancer cells in your bladder. The longer the bladder is exposed to the isothiocyanates in your urine, the longer it will be exposed to anti-cancer activities. Many people urinate several times a day a less often at night. So, there is a greater chance that the isothiocyanates from the power vegetables will say in your bladder longer if you eat power vegetables at night.

| Scoring | Circle all questions that were answered <u>incorrectly</u> . | none | TB1 | TB2 | # Incorrect |
|---|---|---|---|---|---|
| | | ТВ3 | TB4 | TB5 | |
| | | ТВ6 | ТВ7 | | |

**ALL** *CORRECT*: Excellent job! You know all the important parts of the POW-R Health Magazine and you got all of those questions correct.

**ANY INCORRECT:** You did a good job remembering information from the magazine. I know there was a lot of information covered. So, let's just briefly recap the ones you missed before ending the call.

10/31/2022 

# □ PART I: Closing

Thanks for taking the time to complete this call. Next week you will start receiving automated phone calls from our POW-R Health Program. The purpose of the calls will be to support you to eat more power vegetables. The calls will be tailored personally to you. Each call will ask you how many cups of power vegetables you ate for the week, figure out whether you are meeting your action plan goals, and then give you tailored support based on the obstacles and strategies you wrote down in your action plan. So, it will really be important for you to complete your POW-R Book every day, calculate your total power vegetables eaten at dinner or after dinner at the end of every week, and have that available when you receive the phone call.

The system will call you from this number: 716-333-POWR (7697). You can also call this number if you miss the call. This number is on the magnet we mailed to you to remind you that this is not a spam number. Can you please get the magnet we sent you out? Please place this magnet in a place that you'll be able to see it. If you miss a call, you can also call this number too to complete your automated phone call. There will be 11 automated phone call and we ask you to complete all 11 calls.

Each call will start by asking you what your date of birth is, so the system will know it is you. For example, if you were born January 3, 1953, you would enter 01-03-1953. The system will call you from this number: 716-333-POWR. You can also call this number if you miss the call.

Can you tell me how you will enter your date of birth? [Confirm that the participant can provide their DOB correctly]

DOB Correctly read
No Yes

Each automated phone call will last about 10-15 minutes. Please stay on the phone until the call is complete, otherwise the system will think that you did not complete the call and it will call you again.

(Go over any magazine content questions they missed: Let's go over one last time the question(s) you missed)

What questions do you have for me before we hang up?

Okay, just remember, if you ever have any questions or concerns, you can always get a hold of us by calling one of our team members at 716-845-1300, Ext 7221. This number is on the back of the Track Book and the last page of the magazine.

Record questions

Thank you for completing the call!

Control

10/31/2022 

| Participant ID: | Staff Initials: Date: _ | | |
|---|---|---|---|
| Start Time: | End Time: | ☐ Treatment | ☐ Control |
| Materials that sho | ould have been sent to participant | | |
| Cover Letter/Welcome | e Letter | | |
| POW-R Health Magaz | zine | | |
| POW-R Track Book (2 | 24 copies) | | |
| Refrigerator Magnet | | | |
| PART A: G | etting participant on the phone, call i | ntro, packet recei | pt |
| Note: Only make three attempts | to reach the participant | | |
| ☐ Phone Answered | | | |
| Hello, this is [staff name] [participant name] home/a | from the POW-R Health program calling for [participa available right now? | nt name], she/he is expect | ing my call. Is |
| Yes | Hi [participant name] I'm calling to review the POW should take about 60 minutes; do you have time to co | | als with you. It |
| No | That's okay, can we schedule a time that would work better for you? Thanks, I will give you a call then. | | Time to call back |
| ☐ Leaving Message | | | |
| 1 <sup>st</sup> Attempt | This is [ <i>staff name</i> ] from the POW-R Health program to review the POW-R Health program materials with try calling you again, but if you would like to call me chat, I can be reached at 716-697-4615/716-720-2308 soon! | you, which should take ab<br>back and let me know a g | oout 1 hour. I'll ood time for us to |
| 2 <sup>nd</sup> Attempt | Hello again, this is [staff name] from the POW-R Heat I left a message with you on[date] and I am Health program materials with you, which should tak time, but if you would like to call me back and let me reached at 716-697-4615/716-720-2308. Thanks, and | calling you back to review<br>e about 1 hour. I'll try call<br>know a good time for us t | the POW-R ing you one more to chat, I can be |
| 3 <sup>rd</sup> Attempt | Hello again, this is [staff name] from the POW-R Heal I left a message with you on[date], and I am Health program materials with you, which should tak | calling you back to review | the POW-R |

back and let me know a good time for us to chat, I can be reached at 716-697-4615/716-720-

10/31/2022 

2308. Thanks, and I hope I catch up with you soon!

#### ☐ Confirm Intervention Packet Receipt

We are glad you are a part of the program. We put a program packet in the mail for you about the POW-R Health Program. The packet should have included a magazine, booklets, and a magnet.

A1. Did you receive the program packet in the mail?

If YES: (Go to Question A2)

If NO: It's really important that you have your packet before we go over it. Let me make a note to send you the packet again. What is your mailing address? I'll call you again after your packet is sent. Thank you for taking the time to talk with me. I'll talk to you again soon.

END CALL.

A2. If so, did you have time to review the information in this packet?

| | Mailing<br>Address |
|----|--------------------|
| No | Yes |

# ☐ PART B: OVERVIEW

#### $\square$ How can you get the best health benefits from fruits and vegetables?

- Vegetables: Fresh, frozen, and canned vegetables can all be a part of healthy eating.
  - o Fresh vegetables are best
  - o Canned vegetables can be high in salt, so if you buy canned vegetables make sure you look for the 'no salt' ones.
- Fruit: Fresh, frozen, and canned fruit can all be a part of healthy eating
  - Fresh fruit is best
  - Canned fruit can be high in sugar and calories, so buy canned fruit in 100% fruit juice with no sugar added.
  - o Be careful of fruit juices! They're high in sugar and calories, and you can miss out on a lot of other vitamins and minerals that <u>eating fruits</u> will give you.
- Eat 2½ to 3 cups of vegetables and 1½ to 2 cups of fruit each day; or a total of 4-5 cups of both fruits and vegetables a day. 1/2 cup is about the size of the **front** of a closed fist. 1 cup is about the size of your entire fist or a baseball.

10/31/2022 

#### ☐ How to prepare fruits and vegetables?

 You can eat a lot of fruits and vegetables raw. You can also cook them in many different ways too

#### $\square$ Tips to Eat More Fruits and Vegetables

O Tips on how to eat more fruits and vegetables are on pages 6-7 of your POW-R Health Magazine.

I'm going to begin by going over the POW-R Magazine. After I go over the magazine's contents, we'll complete your personal action plan. I'll then go over the POW-R Books and the magnet. So let's start with the POW-R Magazine. Please have your POW-R Magazine next to you so you can follow along what I'm going to review.

#### ☐ PART C: MAGAZINE CONTENT

#### $\square$ Welcome to the POW-R Health Program (page 2)

- Living a healthy lifestyle is important for bladder cancer survivors
- Eating fruits and vegetables is an important part of health
- Doctors made the **POW-R Health Program** to make sure you live the longest, healthiest life possible

Interesting convo points

#### ■ What are fruits and vegetables?

- Fruit and vegetables are plants that have lots of minerals, vitamins, and other healthy things that are good for the human body.
- Common fruits and vegetables are listed in the POW-R magazine on page 3.

10/31/2022 

#### ☐ How are fruits and vegetables good for you? (page 4)

- Research has shown that eating fruits and vegetables can help you live longer. Eating fruits and vegetables reduces the risk of getting some cancers, high blood pressure (hypertension), heart disease, and diabetes.
- Fruits and vegetables have all of these great health benefits because they have a lot of vitamins C and A, electrolytes, and antioxidants. Vitamin C protects cells and molecules from damage that causes many diseases, including cancer.
- Fruits and vegetables are also a great source of fiber. The fiber in fruits and vegetables lowers cholesterol, which reduces heart disease risk. The fiber in fruits and vegetables can also help control the body's blood sugar, which reduces risk of diabetes. Fruits and vegetables can also help you have a healthy weight by giving you lots of fiber and water, which can fill you up without giving too many calories.

If YES: Okay great, I'm glad you got a chance to review the material. Just to make sure that the magazine clearly conveyed the information, I will now ask you some questions to go over the main points of the magazine. We will then work together to create your personal action plan to eat more power vegetables. Before we begin, please pull out the packet we sent. It would really help to have them with you for the later part of the call. Please have a pen handy too (Go to PART D).

*If NO:* That is okay. We can still go over what is in the packet right now. Before we begin, please pull out the packet we sent. It would really help to have them with you for the later part of the call Please have a pen handy too. (Go to PART B)

# ☐ Part D: Going over Magazine Components: Teach Back

Just to make sure that the magazine clearly conveyed the information, I am now going to ask you a few questions to review some of the main points of the magazine. You may feel like I'm testing you, but the purpose of this is to make sure that the magazine communicated the information to you clearly. Are you ready? Let's go!

Note: For a question to be answered correctly, all parts of the question must be answered correctly.

**CTB1** How are fruits and vegetables good for you?

Correct: 1) have lots of vitamins that 2) reduces the risk of getting some cancers, high blood pressure (hypertension), heart disease, and diabetes, 3) fiber in fruits and vegetables can also help you have a healthy weight

Correct No Yes

10/31/2022 

**CORRECT**: Yes, that's right!

**INCORRECT:** Let's go to page X in the POW-R Health magazine. On this page, there is a description of fruits and vegetables are good for you. Fruits and vegetables are good for you because they 1) have lots of vitamins that 2) reduces the risk of getting some cancers, high blood pressure (hypertension), heart disease, and diabetes, 3) fiber in fruits and vegetables can also help you have a healthy weight.

How many cups of fruit do you need to eat each day?

\*\*Correct Answer: 1 ½ to 2 cups/day\*

\*\*Correct Answer:

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is the recommendation on how many cups of fruit to each day for best health. For best health, you need to eat 1 ½ to 2 cups of fruit a day. 1 cup of fruit is about the size of your fist.

How cups of vegetables do you need to eat each day?

\*\*Correct Answer: 2 ½ to 3 cups/day\*\*

\*\*Co

**CORRECT:** Excellent, you're right.

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is the recommendation on how many cups of vegetables to each day for best health. For best health, you need to eat 2 ½ to 3 cups of vegetables a day. 1 cup of vegetables is about the size of your fist.

CTB4 What does 1 cup of fruit or vegetable look like?

\*\*Correct Answer: 1 cup is about the size of your fist.\*\*

Correct Answer: 1 cup is about the size of your fist.\*\*

No Yes

**CORRECT:** Excellent, you're right. 1 cup of vegetables or fruit is about the size of your fist.

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there are pictures of what 1 cup looks like. The size of your fist is about 1 cup.

Fresh, frozen, and canned fruits can all be a part of healthy eating. Can you please tell me what you need to watch out for when you buy canned fruit?

\*\*Correct Answer: Added sugars in canned fruit (buy no added sugar, 100% fruit juice kind)\*\*

\*\*Correct Answer: Added sugars in canned fruit (buy no added sugar, 100% fruit juice kind)\*\*

**CORRECT:** Ok great, you're right.

10/31/2022 

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is describes what types of fruit are best to eat. Fresh, frozen, and canned fruits can all be a part of healthy eating. When it comes to canned fruits, you just need to watch out for too much sugar. Buy the no added sugar type.

Fresh, frozen, and canned vegetables can all be a part of healthy eating. Can you please tell me what you need to watch out for when you buy canned vegetables

\*\*Correct Answer: Too much salt in canned vegetables\*\*

(buy no salt added kind)

\*\*Correct Answer: Too much salt in canned vegetables\*\*

Correct Answer: Too much salt in canned vegetables\*\*

**CORRECT:** Ok great, you're right.

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is describes what types of vegetables are best to eat. Fresh, frozen, and canned vegetables can all be a part of healthy eating. When it comes to canned vegetables, you just need to watch out for too much salt. Buy the no salt added.

| СТВ7 | Can fruit juices be a part of a healthy diet? | Correct |
|---|---|---|
| | Correct Answer: It's best to choose fruits you can eat instead of drink. Many fruit juices are high in sugar and calories and don't have a lot of minerals that fruit has when you eat them instead. | No Yes |

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there it talks about fruit juices. It's best to choose fruits you can eat instead of drink. Many fruit juices are high in sugar and calories and don't have a lot of minerals that fruit has when you eat them instead.

| <b>Scoring</b> Circle all questions that were answered <u>incorrectly</u> . | none | TB1 | TB2 | # Incorrect |
|---|---|---|---|---|
| | ТВ3 | TB4 | TB5 | |
| | TB6 | TB7 | | |

**ALL** *CORRECT*: Excellent job! You really read through the POW-R Health Magazine and you got all of those questions correct. Now let's move on and put together an Action Plan! *[Go to Part F]* 

**ANY INCORRECT**: [GO TO PART E]

10/31/2022 

# ☐ Part E: Going over Magazine Components: Teach Back Opportunity

Only ask questions that were answered incorrectly in Part D. SKIP if all questions were answered correctly in Part D.

Is this part applicable?

No Yes

You did a good job remembering information that I just covered. I know there was a lot of information covered. So, let's just briefly recap the ones you missed.

**CTB1.2** How are fruits and vegetables good for you?

Correct: 1) have lots of vitamins that 2) reduces the risk of getting some cancers, high blood pressure (hypertension), heart disease, and diabetes, 3) fiber in fruits and vegetables can also help you have a healthy weight

Correct No Yes

CORRECT: Yes, that's right!

**INCORRECT:** Let's go to page X in the POW-R Health magazine. On this page, there is a description of fruits and vegetables are good for you. Fruits and vegetables are good for you because they 1) have lots of vitamins that 2) reduces the risk of getting some cancers, high blood pressure (hypertension), heart disease, and diabetes, 3) fiber in fruits and vegetables can also help you have a healthy weight.

CTB2.2 How many cups of fruit do you need to eat each day?

Correct Answer: 1 ½ to 2 cups/day

Correct No Yes

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is the recommendation on how many cups of fruit to each day for best health. For best health, you need to eat 1 ½ to 2 cups of fruit a day. 1 cup of fruit is about the size of your fist.

**CTB3.2** How cups of vegetables do you need to eat each day?

Correct Answer: 2 1/2 to 3 cups/day

Correct
No Yes

**CORRECT:** Excellent, you're right.

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is the recommendation on how many cups of vegetables to each day for best health. For best health, you need to eat 2 ½ to 3 cups of vegetables a day. 1 cup of vegetables is about the size of your fist.

10/31/2022 

# CTB4.2 What does 1 cup of fruit or vegetable look like? \*\*Correct Answer: 1 cup is about the size of your fist.\*\* Correct Answer: 1 cup is about the size of your fist.\*\* No Yes

**CORRECT:** Excellent, you're right. 1 cup of vegetables or fruit is about the size of your fist.

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there are pictures of what 1 cup looks like. The size of your fist is about 1 cup.

CTB5.2 Fresh, frozen, and canned fruits can all be a part of healthy eating. Can you please tell me what you need to watch out for when you buy canned fruit?

\*\*Correct Answer: Added sugars in canned fruit (buy no added sugar, 100% fruit juice kind)\*\*

\*\*Correct Answer: Added sugars in canned fruit (buy no added sugar, 100% fruit juice kind)\*\*

CORRECT: Ok great, you're right.

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is describes what types of fruit are best to eat. Fresh, frozen, and canned fruits can all be a part of healthy eating. When it comes to canned fruits, you just need to watch out for too much sugar. Buy the no added sugar type.

CTB6.2 Fresh, frozen, and canned vegetables can all be a part of healthy eating. Can you please tell me what you need to watch out for when you buy canned vegetables

Correct Answer: Too much salt in canned vegetables (buy no salt added kind)

**CORRECT:** Ok great, you're right.

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is describes what types of vegetables are best to eat. Fresh, frozen, and canned vegetables can all be a part of healthy eating. When it comes to canned vegetables, you just need to watch out for too much salt. Buy the no salt added.

| CTB7.2 | Can fruit juices be a part of a healthy diet? | Correct |
|---|---|---|
| | Correct Answer: It's best to choose fruits you can eat instead of drink. Many fruit juices are high in sugar and calories and don't have a lot of minerals that fruit has when you eat them instead. | No Yes |

**CORRECT:** Yes, that's right- good job!

10/31/2022 

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there it talks about fruit juices. It's best to choose fruits you can eat instead of drink. Many fruit juices are high in sugar and calories and don't have a lot of minerals that fruit has when you eat them instead.

| Scorin<br>g | Circle all questions that were answered <u>incorrectly</u> . | non<br>e | TB1<br>TB4 | TB2<br>TB5 | # Incorrect |
|---|---|---|---|---|---|
| | | ТВ3 | ТВ7 | | |
| | | ТВ6 | | | |
| ALL CORRECT: Excellent job! You really read through the POW-R Health Magazine and you got all | | | | | |

**ALL CORRECT:** Excellent job! You really read through the POW-R Health Magazine and you got all of those questions correct. Now let's move on and put together an Action Plan! [Go to Part F]

**ANY INCORRECT:** We'll go over these questions one more time before we end our call today. [GO TO PART F]

# ☐ Part F: Complete Action Plan with Participant

☐ Reasons for joining the POW-R Health Program

Now let's go to the Action plan, which is on page 9 of the POW-R Health Magazine. Write your answers down in the plan.

| The asons for joining the Fow-K fleath Frogra | ani |
|---|---|
| What are the most important reasons you have for joining the POW-R Health Program? Write this/these down in your action plan. | Participant reason(s): |
| ☐ Power vegetable eating goals | |
| Let's set some short- and long-term goals. Let's start with a long-term goal. In 6 months, which is by the end of this program, how many cups of fruit and vegetables do you pledge to eat <u>each</u> <u>day</u> . | Long term goal |
| Now let's set your short-term goal. For this week, how many cups of fruit and vegetables will you try to eat <u>this week</u> ? | Short-term goal |
| ☐ Who can help me | |
| Who can help you eat more fruit and vegetables? Who can support you? | Support person |

10/31/2022 

| ☐ Fruit and vegetable obstacles and strategies | |
|---|---|
| Let's now talk about some obstacles that could make it harder for you to complete your plan. What are one or two obstacles that could make it harder for you to eat more fruit and vegetables every day? | Obstacle 1 Obstacle 2 |
| What are some strategies you could use to help overcome the obstacles you listed? | Obstacle 1, Strategies (2-4) |
| | Obstacle 2, Strategies (2-4) |
| $\square$ My plan this week to eat more fruit and vege | tables |
| Now let's make a plan to eat more fruit and vegetables this week. The next time you or someone else goes to the grocery store, which fruit and vegetables will you buy? | Fruit and vegetables to buy |

#### ☐ Part G: Go over POW-R Track Book

One of the things you received in the packet we mailed to you is a POW-R Book. Please have your POW-R Book ready to review. In this book, I am asking that you keep track of how many fruit and vegetables you eat every day, and each week. Science shows that keeping track of what you eat is a powerful way to change your habits. Keeping track of how many fruit and vegetables you eat will help you eat more fruit and vegetables. Let's go over all of the parts of the POW-R Book.

#### Check box when section is covered

- 1. 1 POW-R book for each week; 24 sent to you—1 is for practice to use now; we are asking you to complete a track book each week for the entire program
- 3. 7 days in one POW-R book
- 5. Each day write down how many cups of fruit you had that day. (have them go through pages of book)
- 7. On the back is the phone number of the person from our team that you can call

10/31/2022 

Cover page—write down dates of the week you are keeping track 4. Each day write down how many cups of vegetables you had that day. (have them open up book)

6. On the front page, is where you will write down: 1) the total cups of fruit, 2) total cups of vegetables, and 3) total number of fruits AND vegetables you ate that week. Place a check-mark by whether you ate at least 1.5 cups of fruit that week (yes/no). Same with vegetables. After our phone call, you will receive automated messages and will be asked to enter the total number of cups of fruit AND vegetables you ate for the week (refer them to last line). It will also ask you whether you ate at least 1.5 cups of fruit, and 2.5 cups of vegetables and you will use the information here to tell them 'yes' or 'no'

if you have any questions. 8. Any questions?

Let's practice using the POW-R Track Book.

| ☐ Practice using POW-R Track Book | | | | | |
|---|---|---|---|---|---|
| Take a POW-R Track Book. Can you think back this past week of any fruit you ate? Let's go | Monday | Tuesday | | Wed | |
| through each day. | Thursday | Friday | Sat | Sunday | |
| Now let's add how many cups you ate that week | Total | | | Correct | |
| | | | | No | Yes |

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** Ok, so the correct total is X. Let's try that again to make sure you can use the POW-R Book correctly. Feel free to use a calculator if that would make things easier.

# ☐ Part H: Going over magazine components: Teach Back Opportunity #3

Only ask questions that were answered incorrectly in Part E. SKIP if all questions were answered correctly in Part D or E.

Is this Part applicable?

No Yes

Before we end the call, I just want to re-ask you the questions about the key points from the magazine that you were not able to recall last time

**CTB1.3** How are fruits and vegetables good for you?

Correct: 1) have lots of vitamins that 2) reduces the risk of getting some cancers, high blood pressure (hypertension), heart disease, and Correct **No Yes** 

10/31/2022 

diabetes, 3) fiber in fruits and vegetables can also help you have a healthy weight

**CORRECT**: Yes, that's right!

**INCORRECT:** Let's go to page X in the POW-R Health magazine. On this page, there is a description of fruits and vegetables are good for you. Fruits and vegetables are good for you because they 1) have lots of vitamins that 2) reduces the risk of getting some cancers, high blood pressure (hypertension), heart disease, and diabetes, 3) fiber in fruits and vegetables can also help you have a healthy weight.

| CTB2.3 | How many cups of fruit do you need to eat each day? | | Correc | et |
|---|---|---|---|---|
| | Correct Answer: 1 ½ to 2 cups/day | No | | Yes |

**CORRECT:** Yes, that's right- good job!

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is the recommendation on how many cups of fruit to each day for best health. For best health, you need to eat 1 ½ to 2 cups of fruit a day. 1 cup of fruit is about the size of your fist.

| CTB3.3 | How cups of vegetables do you need to eat each day? | | Correct | • |
|---|---|---|---|---|
| | Correct Answer: 2 ½ to 3 cups/day | No | ` | Yes |

**CORRECT:** Excellent, you're right.

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is the recommendation on how many cups of vegetables to each day for best health. For best health, you need to eat 2 ½ to 3 cups of vegetables a day. 1 cup of vegetables is about the size of your fist.

| CTB4.3 | What does 1 cup of fruit or vegetable look like? | | Correct | |
|---|---|---|---|---|
| | Correct Answer: 1 cup is about the size of your fist. | No | Ye | s |

**CORRECT:** Excellent, you're right. 1 cup of vegetables or fruit is about the size of your fist.

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there are pictures of what 1 cup looks like. The size of your fist is about 1 cup.

10/31/2022 

**CTB5.3** Fresh, frozen, and canned fruits can all be a part of healthy eating. Can you please tell me what you need to watch out for when you buy canned fruit?

Correct No Yes

Correct Answer: Added sugars in canned fruit (buy no added sugar, 100% fruit juice kind)

**CORRECT:** Ok great, you're right.

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is describes what types of fruit are best to eat. Fresh, frozen, and canned fruits can all be a part of healthy eating. When it comes to canned fruits, you just need to watch out for too much sugar. Buy the no added sugar type.

**CTB6.3** Fresh, frozen, and canned vegetables can all be a part of healthy eating. Can you please tell me what you need to watch out for when you buy canned vegetables

Correct
No Yes

Correct Answer: Too much salt in canned vegetables (buy no salt added kind)

**CORRECT:** Ok great, you're right.

**INCORRECT:** If you look at on page X of your POW-R Health Magazine, there is describes what types of vegetables are best to eat. Fresh, frozen, and canned vegetables can all be a part of healthy eating. When it comes to canned vegetables, you just need to watch out for too much salt. Buy the no salt added.

**CTB7.3** Can fruit juices be a part of a healthy diet?

Correct

Yes

No

Correct Answer: It's best to choose fruits you can eat instead of drink. Many fruit juices are high in sugar and calories and don't have a lot of minerals that fruit has when you eat them instead

**CORRECT:** Yes, that's right- good job!

**INCORRECT**: If you look at on page X of your POW-R Health Magazine, there it talks about fruit juices. It's best to choose fruits you can eat instead of drink. Many fruit juices are high in sugar and calories and don't have a lot of minerals that fruit has when you eat them instead.

Scoring Circle all questions that were answered incorrectly.

TB1

TB2

# Incorrect

TB3

TB4

TB5

TB6

TB7

10/31/2022 

**ALL CORRECT:** Excellent job! You know all the important parts of the POW-R Health Magazine and you got all of those questions correct.

**ANY INCORRECT:** You did a good job remembering information from the magazine. I know there was a lot of information covered. So, let's just briefly recap the ones you missed before ending the call.

# ☐ PART I: Closing

Thanks for taking the time to complete this call. Next week you will start receiving automated phone calls from our POW-R Health Program. The purpose of the calls will be to support you to eat more fruit and vegetables. The calls will be tailored personally to you. Each call will ask you how many fruit and vegetables you ate for the week, figure out whether you are meeting your action plan goals, and then give you tailored support based on the obstacles and strategies you wrote down in your action plan. So, it will really be important for you to complete your POW-R Book every day, calculate your total cups of fruit and vegetables eaten at the end of every week, and have that available when you receive the phone call.

The system will call you from this number: 716-333-POWR (7697). You can also call this number if you miss the call. This number is on the magnet we mailed to you to remind you that this is not a spam number. Can you please get the magnet we sent you out? Please place this magnet in a place that you'll be able to see it. If you miss a call, you can also call this number too to complete your automated phone call. There will be 11 automated phone call and we ask you to complete all 11 calls.

Each call will start by asking you what your date of birth is, so the system will know it is you. For example, if you were born January 3, 1953, you would enter 01-03-1953. The system will call you from this number: 716-333-POWR. You can also call this number if you miss the call.

Can you tell me how you will enter your date of birth? [Confirm that the participant can provide their DOB correctly]

DOB Correctly read
No Yes

Each automated phone call will last about 10-15 minutes. Please stay on the phone until the call is complete, otherwise the system will think that you did not complete the call and it will call you again.

(Go over any magazine content questions they missed: Let's go over one last time the question(s) you missed)

What questions do you have for me before we hang up?

Okay, just remember, if you ever have any questions or concerns, you can always get ahold of us by calling one of our team members at 716-845-1300, Ext 7221. This number is on the back of the Track Book and the last page of the magazine.

Thank you for completing the call!

10/31/2022 

call 716-333-POWR (7697).

# Appendix R. Participant Track Books

#### Intervention

| Su | INDAY | |
|---|---|---|
| Hov | w many cups of vegetables did you eat? | Dates This Week:/ to/ |
| O | 0 | |
| 0 | ½ cup | |
| O | 1 cup | |
| 0 | 1 ½ cups | |
| O | 2 cups | |
| O | 2 ½ cups | |
| O | 3 cups | HEALTH |
| O | OTHER: | HEALIH |
| Hov | w many cups of fruit did you eat? | |
| 0 | 0 | TRACK BOOK |
| O | ½ cup | IRACK DOOK |
| 0 | 1 cup | How many fruits and vegetables did you eat |
| O | 1 ½ cups | this week? |
| O | 2 cups | 200 COM |
| O | OTHER: | Total cups of vegetables eaten this week: |
| | | Did you eat at least 2.5 cups of vegetables this week? ○YES ○NO |
| | | tills week: OTES ONO |
| | If you have any questions, | Total cups of fruit eaten this week: |
| | please call 716-845-1300, Ext 7221. | Did you eat at least 1.5 cups of FRUIT |
| | If you need to access the | this week? OYES ONO |
| | POW-R automated phone system, | |

10/31/2022 

| MU | INDAY | 5A | IURDAY |
|---|---|---|---|
| How | v many cups of vegetables did you eat? | Hov | v many cups of vegetables did you eat? |
| 0 | 0 | O | 0 |
| 0 | ½ cup | O | ½ cup |
| 0 | 1 cup | 0 | 1 cup |
| 0 | 1 ½ cups | 0 | 1 ½ cups |
| 0 | 2 cups | O | 2 cups |
| 0 | 2 ½ cups | O | 2 ½ cups |
| 0 | 3 cups | O | 3 cups |
| 0 | OTHER: | O | OTHER: |
| How | v many cups of fruit did you eat? | Hov | v many cups of fruit did you eat? |
| 0 | 0 | O | 0 |
| 0 | ½ cup | O | ½ cup |
| 0 | 1 cup | O | 1 cup |
| 0 | 1 ½ cups | O | 1 ½ cups |
| O | 2 cups | O | 2 cups |
| 0 | OTHER: | 0 | OTHER: |

10/31/2022 

| ŀ | R | IDAY | L | U | ESDAY |
|---|---|---|---|---|---|
| Н | lov | many cups of vegetables did you eat? | Н | οw | many cups of vegetables did you eat? |
| ( | C | 0 | | ) | 0 |
| ( | C | ½ cup | | ) | ½ cup |
| ( | C | 1 cup | | ) | 1 cup |
| ( | C | 1 ½ cups | | ) | 1 ½ cups |
| ( | C | 2 cups | | ) | 2 cups |
| ( | C | 2 ½ cups | | ) | 2 ½ cups |
| ( | C | 3 cups | | ) | 3 cups |
| ( | C | OTHER: | | ) | OTHER: |
| Н | lov | many cups of fruit did you eat? | Н | οw | many cups of fruit did you eat? |
| ( | C | 0 | | ) | 0 |
| ( | C | ½ cup | | ) | ½ cup |
| ( | C | 1 cup | | ) | 1 cup |
| ( | C | 1 ½ cups | | ) | 1 ½ cups |
| ( | C | 2 cups | | ) | 2 cups |
| ( | C | OTHER: | | ) | OTHER: |

10/31/2022 

| WE | DNESDAY | TH | URSDAY |
|---|---|---|---|
| How | many cups of vegetables did you eat? | Hov | v many cups of vegetables did you eat? |
| O | 0 | 0 | 0 |
| O | ½ cup | 0 | ½ cup |
| 0 | 1 cup | 0 | 1 cup |
| 0 | 1 ½ cups | 0 | 1 ½ cups |
| 0 | 2 cups | 0 | 2 cups |
| 0 | 2 ½ cups | 0 | 2 ½ cups |
| O | 3 cups | 0 | 3 cups |
| O | OTHER: | 0 | OTHER: |
| How | many cups of fruit did you eat? | Hov | v many cups of fruit did you eat? |
| 0 | 0 | 0 | 0 |
| O | ½ cup | O | ½ cup |
| O | 1 cup | $\circ$ | 1 cup |
| 0 | 1 ½ cups | 0 | 1 ½ cups |
| 0 | 2 cups | 0 | 2 cups |
| 0 | OTHER: | O | OTHER: |

10/31/2022 

call 716-333-POWR (7697).

### Control

# **SUNDAY**

| Hov | many cups of vegetables did you eat? | Dates This Week:/ to/ |
|---|---|---|
| 0 | 0 | |
| 0 | ½ cup | |
| O | 1 cup | |
| 0 | 1 ½ cups | |
| O | 2 cups | |
| 0 | 2 ½ cups | |
| O | 3 cups | HEALTH |
| O | OTHER: | |
| Hov | v many cups of fruit did you eat? | |
| 0 | 0 | TRACK BOOK |
| O | ½ cup | I KACK DUUK |
| 0 | 1 cup | How many fruits and vegetables did you eat |
| O | 1 ½ cups | this week? |
| 0 | 2 cups | |
| 0 | OTHER: | Total cups of vegetables eaten this week: |
| | | Did you eat at least 2.5 cups of vegetables |
| | | this week? OYES ONO |
| | If you have any questions, | Total cups of fruit eaten this week: |
| | please call 716-845-1300, Ext 7221. | Did you eat at least 1.5 cups of FRUIT |
| | If you need to access the | this week? OYES ONO |
| | POW-R automated phone system, | |
| | row-k automateu phone system, | |

10/31/2022 

| MU | INDAY | SA | TURDAY |
|---|---|---|---|
| How | many cups of vegetables did you eat? | Hov | v many cups of vegetables did you eat? |
| O | 0 | O | 0 |
| O | 1/2 cup | O | ½ cup |
| 0 | 1 cup | O | 1 cup |
| 0 | 1 ½ cups | 0 | 1 ½ cups |
| 0 | 2 cups | 0 | 2 cups |
| 0 | 2 ½ cups | 0 | 2 ½ cups |
| O | 3 cups | O | 3 cups |
| 0 | OTHER: | 0 | OTHER: |
| How | many cups of fruit did you eat? | Hov | v many cups of fruit did you eat? |
| 0 | 0 | O | 0 |
| O | 1/2 cup | O | ½ cup |
| O | 1 cup | O | 1 cup |
| 0 | 1 ½ cups | O | 1 ½ cups |
| 0 | 2 cups | 0 | 2 cups |
| O | OTHER: | O | OTHER: |

10/31/2022 

| FR | IDAY | IU | ESDAY |
|---|---|---|---|
| How | v many cups of vegetables did you eat? | Hov | v many cups of vegetables did you eat? |
| O | 0 | O | 0 |
| O | ½ cup | O | ½ cup |
| 0 | 1 cup | O | 1 cup |
| 0 | 1 ½ cups | 0 | 1 ½ cups |
| 0 | 2 cups | 0 | 2 cups |
| 0 | 2 ½ cups | 0 | 2 ½ cups |
| O | 3 cups | O | 3 cups |
| O | OTHER: | O | OTHER: |
| How | v many cups of fruit did you eat? | Hov | v many cups of fruit did you eat? |
| 0 | 0 | O | 0 |
| O | ½ cup | O | ½ cup |
| O | 1 cup | O | 1 cup |
| 0 | 1 ½ cups | O | 1 ½ cups |
| O | 2 cups | 0 | 2 cups |
| 0 | OTHER: | 0 | OTHER: |

10/31/2022 

| WE | DNESDAY | TH | URSDAY |
|---|---|---|---|
| How | many cups of vegetables did you eat? | How | many cups of vegetables did you eat? |
| O | 0 | O | 0 |
| O | ½ cup | O | ½ cup |
| 0 | 1 cup | 0 | 1 cup |
| 0 | 1 ½ cups | 0 | 1 ½ cups |
| O | 2 cups | 0 | 2 cups |
| O | 2 ½ cups | 0 | 2 ½ cups |
| O | 3 cups | O | 3 cups |
| 0 | OTHER: | O | OTHER: |
| How | many cups of fruit did you eat? | How | many cups of fruit did you eat? |
| O | 0 | O | 0 |
| O | ½ cup | 0 | ½ cup |
| O | 1 cup | 0 | 1 cup |
| 0 | 1 ½ cups | 0 | 1 ½ cups |
| O | 2 cups | 0 | 2 cups |
| 0 | OTHER: | 0 | OTHER: |

10/31/2022 

#### Appendix S. Participant Thank You Letter

[DATE] [FIRST AND LAST NAME OF PARTICIPANT] [STREET ADDRESS] [CITY, STATE ZIP CODE]

Dear [FIRST NAME OF PARTICIPANT],

I am writing to thank you personally for completing the [baseline/follow-up] assessment of the POW-R Health Program. To show our appreciation for your time and effort, we have enclosed Tops gift card for \$X. In 6 months, we will ask you to complete these surveys again and if you do, you will earn another \$X.

On behalf of the POW-R Health team, thank you so much for supporting our research! Please don't hesitate to contact us at: 716-845-1300, Ext 7221.

Sincerely,

Karen Yeary, PhD

Haven yeary

Principal Investigator

Li Tang, PhD

Principal Investigator

10/31/2022 

#### Appendix T. Recruitment Letter for Roswell Park Cancer Registry

Date

Dear Participant,

We recently received funding from the National Institutes of Health to learn more about how diet may reduce the risk of recurrence in individuals with early-stage bladder cancer. Men and women who were recently diagnosed with early-stage bladder cancer and who live in the counties of Niagara, Orleans, Genesee, Erie, Wyoming, Chautauqua, Cattaraugus, and Allegany may be eligible for the study.

We are asking you to take part in this study because you have been diagnosed and treated for bladder cancer. The goal of this study is to make a healthy eating program to improve cancer outcomes. The purpose of this study is to compare two types of healthy eating programs. This study will allow the researchers to know whether different types of healthy eating programs can improve the bladder cancer outcomes of the patients. The intervention that you will receive as part of this study will be given to you at no cost.

If you agree to take part in this research study, you will receive a \$100 gift card for completion of the baseline surveys and you will receive another \$100 gift card for completion of the 6-month survey.

This study has been reviewed and approved by the Roswell Park Institutional Review Board to assure that the study plans will not put any participants at risk. Your involvement in this study does not involve any physical risk to you. The possible risks might be feeling uncomfortable answering questions, embarrassment, or someone identifying you as a participant in the group, although this would be rare. You will not receive any direct health benefit from participating in this study.

Someone from our office will call you to make sure you received this letter and to discuss the study with you. If you have any questions, please call us at 716-845-XXXX. We hope that you will be able to help us by completing the survey.

We hope to hear from you soon!

10/31/2022 

#### Appendix U. Invitation Letter for Physician Interview and Opt-In/Out Card

Date

Dear Dr. X,

Your patient or colleague recently participated in the POW-R Health research study, a National Cancer Institute (NCI)-funded study that is testing different dietary strategies to lower the risk of bladder cancer recurrence. We are excited about this study because it may produce a dietary intervention that helps reduce the risk of bladder cancer recurrence and improve bladder cancer survivorship. To be noted, the funded study is a behavior intervention program that has no relevance to clinical treatment regardless of whether clinical care is provided.

We are contacting you because either your patient or colleague nominated you to be a part of this study. To be part of the study, all we need is to conduct a 15-minute phone interview with you to gain a physician's insight on how our dietary intervention—if proven to be successful—could be incorporated into routine care. Physicians who participate will receive a \$100 gift card from a local store as a small token of our appreciation.

If you can participate in a 15-minute phone interview, please let us know by filling out the card included in this mailing. If you do not want to participate, please let us know on the card so we do not contact you in the future.

For more detailed information about the study, please review the included information sheet.

Thanks so much for our consideration. We hope to hear from you soon.

Sincerely,

Karen Yeary, PhD

Haven youry

**Professor** 

Cancer Prevention and Control

Roswell Park Comprehensive Cancer Center

Li Tang, PhD Associate Professor

Cancer Prevention and Control

Roswell Park Comprehensive Cancer Center

10/31/2022 



| ☐ Yes, I'm intere | ested in participating in the phone interview. Please call |
|---|---|
| me at: | during the following days and times: |
| □ No, I'm not in | terested in participating. Please do not contact me again |
| about this study. | |

10/31/2022 

#### Appendix V. POW-R Sympathy Card



Study Number and title: I 661820; POW-R Health: Power to Redefine your Health (Internal Title: A Pragmatic Dietary Intervention to Improve Bladder Cancer Survivorship)

Dear [...],

We wanted to write to extend our deepest sympathy for the loss of your [partner/wife/husband/loved one], [Participant's name].

No one should ever have to experience such pain and loss - we are sorry that you are.

Please know that we are thinking of you and your loved ones. We send our heartfelt condolences and strength your way.

Sincerely,
[Names of research staff]
The POW-R Study Research Team
Roswell Park Comprehensive Cancer Center

10/31/2022 

# Appendix W. Participant Information Sheet for Cruciferous Arm Feedback Questions (For Participants that Completed the 6-Month Follow-up Assessment)



[DATE]

Dear POW-R Health Participant,

Thank you for participating in the POW-R Health Program! Your participation will make a difference in understanding how to improve the health of bladder cancer survivors like you. To make the program better, a Roswell Park team member will call you to ask a few questions about what you liked and didn't like about the program. The phone call will take about 10-15 minutes.

Your participation is voluntary. All responses will remain confidential and anonymous and will be shared with only the Roswell Park POW-R Health Program team. If you don't want to talk with us, please tell us when we call you.

We believe that your valuable feedback will help make the POW-R Health program better, so it can be more useful to more bladder cancer survivors like you. Please be on the lookout for a phone call from our POW-R Health team. If you have any questions regarding the upcoming phone call please don't hesitate to contact us at: 716-845-1300, Ext 4236.

Sincerely,

Karen Yeary, PhD Principal Investigator

Haven yeary

Li Tang, PhD Principal Investigator

10/31/2022 